

## **Clinical Trial Protocol**

| | | Doc. No.: c01618200-19 |
|---|---|---|
| EudraCT No.: | 2009-013157-15 | |
| BI Trial No.: | 1218.74 | |
| BI Investigational Product(s): | Linagliptin | |
| Title: | blind study to evaluate C | nal, randomised, parallel group, double ardiovascular safety of linagliptin ents with type 2 diabetes mellitus at |
| | The <b>CAROLINA</b> Trial. | |
| Clinical Phase: | III | |
| Trial Clinical Monitor | : | |
| | Phone: | Fax: |
| Co-ordinating Investigators: | | |
| | phone: | phone: |
| | fax: | fax: |
| Status: | Final Protocol | |
| Version and Date: | Version 7, 20 April 2016 | |
| | Proprietary confidentia | Linformation |

© 2019 Boehringer Ingelheim International GmbH or one or more of its affiliated companies. All rights reserved. This document may not - in full or in part - be passed on, reproduced, published or otherwise used without prior written permission.

## **CLINICAL TRIAL PROTOCOL SYNOPSIS**

| Name of company: | | Tabulated<br>Trial Protocol | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished produ | uct | | |
| Not applicable | | | 4 |
| Name of active ingredi | ent: | | |
| Linagliptin | | | 10' |
| Protocol date:<br>17 August 2010 | <b>Trial number:</b> 1218.74 | | Revision date:<br>20 April 2016 |
| Title of trial: | evaluate Cardiovascular | nal, randomised, parallel group, dou<br>safety of <b>lina</b> gliptin versus glimepi<br>th cardiovascular risk. The <b>CAROL</b> | ride in patients with type |
| Co-ordinating<br>Investigators: | | ~O? 50° | |
| | and: | RIFE | |
| | \(\sigma\) | 1 | |
| Trial sites: | Approximately 700 study | y centres, on average 8 to 10 patient | s per site |
| Clinical phase: | III | | |
| Objectives: | upper limit of a two-side inferiority margin of 1.3 (as monotherapy or as aco of the adjudicated comportion [CV] death, non-fatal str MI) in patients with type hypothesis with margin 1 primary composite endposuperiority test has reveal endpoint will be tested his first key secondary hypothesis secondary endpoint will Other objectives are to composite the composite of the compos | ompare HbA1c change from baselir | terval with the non- imparison to glimepiride to first occurrence of any dpoint (i.e. cardiovascular ion [MI] (excluding silent e non-inferiority then secondly, the hypothesis. If the the first key secondary othesis. If the test of the alt, then fourthly the If the test of the second men fifthly the third key he, the incidence of |
| | patients that are on study | change, treatment sustainability [defortreatment at study end without need in glycaemic control (HbA <sub>1c</sub> $\leq$ 7.0%) | d for rescue medication, |

| Name of company: | | Tabulated | |
|---|---|---|---|
| | | Trial Protocol | |
| Boehringer Ingelheim | | | |
| Name of finished produ | ıct | | |
| Not applicable | | | |
| Name of active ingredic | ent: | | |
| Linagliptin | | | |
| Protocol date: | Trial number: | | Revision date: |
| 17 August 2010 | 1218.74 | | 20 April 2016 |
| Methodology: | | altinational, randomised, double blin<br>ady of linagliptin versus glimepirid | |
| No. of patients: | | 0 | |
| total entered: | An estimated number of primary endpoints. | 6000 randomised patients to obtain | a minimum of 631 |
| each treatment | : An estimated number of | 3000 randomised patients per treatr | nent group. |
| Diagnosis : | T2DM | | |
| Inclusion criteria: | | f T2DM and concurrently insufficie prior to informed consent: | ent glycaemic control and |
| | <ul> <li>Insufficient glyc</li> </ul> | caemic control (at Visit 1a) defined | as: |
| | | 8.5% (48 - 69 mmol/mol) while patientra-indicated to first line anti-diabe | |
| | | lase inhibitor monotherapy (e.g. aca | rhose voglihose) or |
| | | lpha-glucosidase inhibitor, or | 10050, 105110050), 01 |
| | 1 | 8-11-11-11-11-11-11-11-11-11-11-11-11-11 | |
| | b) HbA <sub>1c</sub> <u>6.5 - 7</u> | 7.5% (48 - 58 mmol/mol) while patie | ent is treated with |
| | - sulphonylurea | (SU) monotherapy, or | |
| | - glinide monotl | herapy (e.g. repaglinide, nateglinide | ), or |
| | - metformin + S | SU (combination maximal up to 5 years) | ears), or |
| A . | - metformin + g | clinide (combination maximal up to | 5 years), or |
| | - alpha-glucosid<br>or | lase inhibitor + SU (combination ma | aximal up to 5 years), |
| | - alpha-glucosid | lase inhibitor + glinide (combination | n maximal up to 5 years) |

Doc No.: c01618200-19 Protocol Revision 6 

| Name of company: | | Tabulated<br>Trial Protocol | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished production | ct | | |
| Not applicable | | | |
| Name of active ingredie | nt: | | |
| Linagliptin | | | |
| Protocol date:<br>17 August 2010 | Trial number: 1218.74 | | Revision date:<br>20 April 2016 |
| Inclusion criteria: | | Vevents defined as any one (or more | - |
| | A) Previous Va | • | |
| | * | infarction (> 6 weeks prior to infor | med concent) |
| | • | d coronary artery disease (≥ 50% lu | |
| | | coronary artery or ≥50% in at leas | |
| | | us Coronary Intervention (PCI) > 6 | weeks prior informed |
| | - Coronary A | artery By-pass Grafting (CABG) > 4 | |
| | | with recurrent angina pectoris follow<br>hemorrhagic stroke (> 3 months pr | • • • |
| | | occlusive arterial disease (previous l | * |
| | stenting or<br>amputation<br>detected sig<br>(common il<br>artery), hist | percutaneous transluminal angioplas due to circulatory insufficiency, angunificant vessel stenosis ( $\geq$ 50%) of diac-, internal iliac-, external iliac-, fory of intermittent claudication with pressure ratio $<$ 0.90). | sty; previous limb or foot<br>giographic or ultrasound<br>major limb arteries<br>emoral- and/or popliteal |
| | B) Evidence of | vascular related end-organ damage: | |
| | - Moderately | impaired renal function (as defined | by modified diet of |
| | | e (MDRD) formula) with estimated | glomerular filtration |
| ٨ ( | | ) 30-59 mL/min/1.73 m <sup>2</sup> | |
| | | ot urinary albumin creatinine ratio ≥ | |
| | • , | n two of three unrelated specimens i | n previous 12 |
| | months prio | | |
| | | e retinopathy defined as retinal neov | ascularisation of |
| | • | inal laser coagulation therapy. | |
| | C) Age $\geq 70$ year. | of the following CV risk factors: | |
| $\bigcup'$ | | etes mellitus duration > 10 years at | Visit 1a |
| | | stolic blood pressure (SBP) > 140 m | |
| | | ressure lowering treatment at Visit 1 | = : |
| | <del>-</del> | y cigarette smoking | <del>"</del> ) |

treatment for this lipid abnormality at Visit 1a)

Current\* LDL cholesterol ≥ 135 mg/dL (3.5 mmol/l) (or specific current

Doc No.: c01618200-19 Protocol Revision 6 

| Name of company: | Tabulated<br>Trial Protocol | |
|---|---|---|
| Boehringer Ingelheim | | |
| Name of finished product | | |
| Not applicable | | |
| Name of active ingredient: | | |
| Linagliptin | | |
| Protocol date: Trial number: 17 August 2010 1218.74 | | Revision date:<br>20 April 2016 |
| <ul> <li>Age ≥ 40 ar</li> <li>Signed and 1a, in according to the stable antileast 8 weel medication randomisati</li> <li>Treatment compliance eligible for randomis</li> <li>Note: To ensure approximate approximate to the stable patients being recruit country). In consultation particular category in This process will be worldwide.</li> </ul> | Index (BMI) ≤ 45 kg/m2 at Visit 1b and ≤ 85 years at Visit 1a dated written informed consent at the lardance with GCP and local legislation diabetic background medication (unchange prior V1a and without short term use should be stable during screening/run-inton at the placebo run-in should be between the | nged daily dose) for at of insulin. Background in phase to allow the different attor the proportion of by region and/or and/or country level). Ition of CV risk categories |

| | | T | |
|---|---|---|---|
| Name of company: | | Tabulated | |
| Boehringer Ingelheim | | Trial Protocol | |
| Name of finished produc | et | | |
| Not applicable | | | |
| Name of active ingredien | nt: | | |
| Linagliptin | | | |
| Protocol date: | Trial number: | | Revision date: |
| 17 August 2010 | 1218.74 | | 20 April 2016 |
| Criteria for exclusion: | Type 1 diabetes Any history and rosiglitazone, prosiglitazone, prosiglitazione, prosigliare, prosiglitazione, | A/or current treatment with other anticoglitazone, GLP-1 analogue/agonis for to informed consent. Note 1: This is antidiabetic drugs have been proved term use of insulin (up to two contring hospitalisation) if taken at least anti-obesity drugs within 3 months appropriate with a glucose level of an overnight fast during placebo rundement (not on the same day) or planned within next 12 months) by intervention (gastric sleeve) and with systemic corticosteroids at the initiation of such therapy. Note: inhabitation of such therapy. Note: inhabitation of thyroid hormones within 6 week the ease or impaired hepatic function, depth. AST (SGOT), or alkaline phose (ULN) as determined at visit 1a gronary artery re-vascularisation (PC) and or any previous PCI and/or CABC. | idiabetic drugs (e.g. its, DPP-IV inhibitors or also includes clinical rided to the patient. Note secutive weeks) is t 8 weeks prior informed prior to informed consent >240 mg/dl (>13.3 - in and confirmed by a ariatric surgery (open or ime of informed consent aled use of steroids (e.g. does not cause systemic sprior informed consent efined by serum levels of sphatase above 3 x upper I, CABG) within next 6 $G \le 6$ weeks prior information in patient history) informed consent that |

Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19 20 April 2016

**Protocol Revision 6** 


| Name of company: | | Tabulated<br>Trial Protocol | |
|---|---|---|---|
| Boehringer Ingelheim | | | |
| Name of finished produ | ıct | | |
| Not applicable | | | |
| Name of active ingredic | ent: | | |
| Linagliptin | | | |
| Protocol date: | Trial number: | | Revision date: |
| 17 August 2010 | 1218.74 | | 20 April 2016 |
| Test product: | of birth control devices/systems sexual abstinent vasectomised probirth control thricontrol thricontro | and an acceptable method of birth continctude tubal ligation, transdermal per (IUDs/IUSs), oral, implantable or ce (if allowed by local authorities), cartner) or do not plan to continue us roughout the study and do not agreeing during participation in the trial. ered unreliable by the investigator continue, has a life expectancy less than ancer other than non-melanoma skingy other condition than mentioned would not allow safe participation in the syndrome ≤ 6 weeks prior to inform ≤ 3 months prior to informed consen | patch, intra uterine injectable contraceptives, double barrier method and ing acceptable method of to submit to periodic oncerning the compliance with study 5 years for non-CV in cancer within last 3 hich in the opinion of the he study ned consent |
| | Linagliptin | | |
| dose: | 5 mg once daily | | |
| mode of admin. : | Tablets per os | | |
| Comparator product: | Glimepiríde | | |
| dose: | 1-4 mg once daily | | |
| mode of admin. : | Tablets (overencapsulate | ed) per os | |
| Duration of treatment: | | run-in phase followed by up to an e<br>days follow-up after study drug tern | |

| Name of company: | | Tabulated | |
|---|---|---|---|
| Boehringer Ingelheim | | Trial Protocol | |
| Name of finished produ | uct | | |
| Not applicable | | | |
| Name of active ingredie | ent: | _ | |
| , and the second | | | 4 |
| Linagliptin | T | | |
| Protocol date: | Trial number: | | Revision date: |
| 17 August 2010 | 1218.74 | | 20 April 2016 |
| Criteria for efficacy: | components of the p | ime to first occurrence of any of the<br>orimary composite endpoint: CV dea<br>atal stroke or non-fatal MI (excluding) | oth (including fatal stroke |
| | adjudicated compon<br>stroke and fatal MI) | endpoint: time to first occurrence of<br>nents of the composite endpoint: CV<br>of non-fatal stroke, non-fatal MI (excurstable angina pectoris. | death (including fatal |
| | defined as the propo<br>at Final Visit mainta<br>rescue medication (I<br>without any modera | Second key secondary endpoint: composite endpoint of (treatment sustainability defined as the proportion of patients that are on study treatment at study end, that at Final Visit maintain glycaemic control (HbA1c $\leq$ 7.0%) without need for rescue medication (between end of titration [Visit 6] and Final Visit) and patients without any moderate/severe hypoglycaemic episodes (between Visit 6 and Final Visit) and without $>$ 2% weight gain at Final Visit (between Visit 6 and Final | |
| | defined as the propo<br>at Final Visit mainta<br>rescue medication (l | y endpoint: composite endpoint of (to ortion of patients that are on study train glycaemic control (HbA1c $\leq$ 7.00 between Visit 6 and Final Visit) and Visit (between Visit 6 and Final Vi | eatment at study end, that %) without need for patients without > 2% |
| Criteria for safety: | (including fatal stro<br>hospitalisation for u<br>heart failure, hospita | nd time to each of the following adj<br>ke and fatal MI), (non)- fatal MI, (n | on)- fatal stroke,<br>alisation for congestive<br>ion procedures (CABG, |
| | | sity of adverse events, physical exame in laboratory parameters | nination, vital signs, ECG, |
| | | its with serious and non-serious hype | |
| | | ne in weight and proportion of patier without rescue medication during r | |
| | Refer to section 5.2 for a | a comprehensive list of safety criteri | a |
| Statistical methods: | first event with factor tree<br>performed on the full an<br>hypotheses will be one-s<br>The first key secondary or<br>regression model of time | a cox proportional hazards regressive atment will be conducted. The primalysis set. The non-inferiority margisided with an overall significance levendpoint will be analysed with a coxe to the first event with factor treatmes will be analysed with Chi-Square to | nary analysis will be n will be 1.3 and the wel of alpha=0.025. The proportional hazards nent. The second and third |

## **FLOW CHART**

| Trial Period | Screening | Placebo<br>run-in | Т | Treatment phase (titration) | | |
|---|---|---|---|---|---|---|
| Visit | 1a | 1b <sup>A</sup> | 2 | 3 | 4 | 5 |
| Study week | | -4 / -2 | 0 | 4 | 8 | 12 |
| Days from randomisation | -35/ -15 | -28 / -14 | 0 | 28 | 56 | 84 |
| Time window (days) <sup>J</sup> | | | | ±7 | ±7 | ±7 |
| Informed Consent | X | | | | | |
| In-/exclusion criteria | X | X | Xc | | | |
| Medical History/<br>Concomitant diagnoses | X | | | | | |
| Demographics <sup>o</sup> | X | X | | | | |
| Physical examination | | $X^{\mathrm{M}}$ | | | | |
| Vital signs | | $X^{\mathrm{M}}$ | X | X | X | X |
| Height | | X <sup>I</sup> | | | | |
| Weight | | X <sup>I</sup> | X | | | |
| Waist circumference | | X | X | | | |
| 12-lead-ECG | | | X <sup>M</sup> | | | |
| Diet and exercise counselling | X | | X | X | X | X |
| Pregnancy Test <sup>F</sup> | X | | X | | | |
| Fasted Home Blood<br>Glucose Monitoring<br>(HBGM) <sup>G</sup> | | X | $X^{L}$ | X | X | X |
| Safety lab Tests (Urine and Blood) <sup>H</sup> | X | | X | | | |
| Glomerular filtration rate <sup>K</sup> | X | | X | | | |

| Trial Period | Screening | Placebo<br>run-in | Treatment phase (titration) | | | |
|---|---|---|---|---|---|---|
| Visit | 1a | 1b <sup>A</sup> | 2 | 3 | 4 | 5 |
| Study week | | -4 / -2 | 0 | 4 | 8 | 12 |
| Days from randomisation | -35/ -15 | -28 / -14 | 0 | 28 | 56 | 84 |
| Time window (days) <sup>J</sup> | | | | ±7 | ±7 | ±7 |
| Fasting Plasma Glucose <sup>B</sup> | | X | X | X | X | X |
| HbA <sub>1c</sub> | X | | X <sup>C</sup> | | | |
| PG sampling <sup>E</sup> | | | X | | | |
| Lipid profile | | | X | | | |
| Adverse events | | X | X | X | X | X |
| Concomitant Therapy | X | X | X | X | X | X |
| Dispense placebo run-in medication (via IXRS) | | X | | | | |
| Randomisation (via IXRS) | | | X | | | |
| Dispense double-blind medication | | | X | X | X | X |
| Medication compliance check | | | X | X | X | X |

BI Trial No.: 1218.74 Doc No.: c01618200-19

| Trial Period | | Treatment phase (maintenance) | | | | | | | | | | | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 6 | 7 | 8 | 9 | 10 | 11 | 12 | 13 | 14 | 15 | 16 | 17 | 18 |
| Study week | 16 | 32 | 48 | 64 | 80 | 96 | 112 | 128 | 144 | 160 | 176 | 192 | 208 |
| Days from randomisation | 112 | 224 | 336 | 448 | 560 | 672 | 784 | 896 | 1008 | 1120 | 1232 | 1344 | 1456 |
| Time window (days) | ±7 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 |
| Physical examination | X | | | X | | | X | | | X | | | X |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Waist circumference | X | | | X | | | X | | | X | | | X |
| 12-lead-ECG | X | | | X | | | X | | | X | | | X |
| Diet and exercise counselling | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Pregnancy Test <sup>F</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Fasted Home<br>Blood Glucose<br>Monitoring<br>(HBGM) <sup>G</sup> | | | | | | | | | | $X^{L}$ | | | |
| Safety lab Tests<br>(Urine and<br>Blood) | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Glomerular filtration rate <sup>K</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Fasting Plasma<br>Glucose <sup>B</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| HbA <sub>1c</sub> | X | X | X | X | X | X | X | X | X | X | X | X | X |
| 1 | | | | | | | | | | | | | |

| Lipid profile | X | | | X | | | X | | | X | | | X |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Therapy | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Dispense<br>double-blind<br>medication | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Medication compliance check | X | X | X | X | X | X | X | X | X | X | X | X | X |

20 April 2016

| Trial Period | | | Treatment phase (maintenance) | | | | | | | | | | | F'<br>up | |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | 27 | 28 | 29 | 30 | 31 | 32<br>EOT <sup>N</sup> | 33 |
| Study week | 224 | 240 | 256 | 272 | 288 | 304 | 320 | 336 | 352 | 368 | 384 | 400 | 416 | 432 | 436 |
| Days from randomisation | 1568 | 1680 | 1792 | 1904 | 2016 | 2128 | 2240 | 2352 | 2464 | 2576 | 2688 | 2800 | 2912 | 3024 | 3054 |
| Time window (days) | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | +7 |
| Physical examination | | | X | | | X | | | X | | | X | | X | |
| Vital signs | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Weight | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Waist circumference | | | X | | | X | | | X | | | X | | X | |
| 12-lead-ECG | | | X | | | X | | | X | | | X | | X | |
| Diet and exercise counselling | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Pregnancy<br>Test <sup>F</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |
| Fasted Home<br>Blood Glucose<br>Monitoring<br>(HBGM) <sup>G</sup> | | | | | | | | | | | | | | $X^{L}$ | |
| Safety lab<br>Tests (Urine<br>and Blood) | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Glomerular<br>filtration rate <sup>K</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Fasting Plasma<br>Glucose <sup>B</sup> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| HbA <sub>1c</sub> | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |

| Trial Period | | | | | | Tı | eatme | nt phas | se (mai | ntenan | ce) | | | | F'<br>up |
|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|---|
| Visit | 19 | 20 | 21 | 22 | 23 | 24 | 25 | 26 | 27 | 28 | 29 | 30 | 31 | 32<br>EOT <sup>N</sup> | 33 |
| Study week | 224 | 240 | 256 | 272 | 288 | 304 | 320 | 336 | 352 | 368 | 384 | 400 | 416 | 432 | 436 |
| Days from randomisation | 1568 | 1680 | 1792 | 1904 | 2016 | 2128 | 2240 | 2352 | 2464 | 2576 | 2688 | 2800 | 2912 | 3024 | 3054 |
| Time window (days) | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | ±14 | +7 |
| Lipid profile | | | X | | | X | | | X | | | X | | X | |
| Adverse events | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Concomitant<br>Therapy | X | X | X | X | X | X | X | X | X | X | X | X | X | X | X |
| Dispense<br>double-blind<br>medication | X | X | X | X | X | X | X | X | X | X | X | X | X | | |
| Medication compliance check | X | X | X | X | X | X | X | X | X | X | X | X | X | X | |

Boehringer Ingelheim 20 April 2016 BI Trial No.: 1218.74

| A | Visit 1b to be performed within 1 week from Visit 1a |
|---|------------------------------------------------------|
| В | Overnight fasting (10 hours no food and only water) |

C HbA<sub>1c</sub> measured at Visit 1a will be used for inclusion

- F For female patients (local urine pregnancy test in women of child bearing potential). More frequent testing can be done if required by local regulations/authorities.
- G Home blood glucose monitoring (HBGM) device provided at Visit 1b. The patient should be instructed to bring their HBGM device to the clinic at least at the specified visits for an additional measurement of fasted glucose.
- H Visit 1a safety laboratory only includes ALT (SGPT), AST (SGOT), alkaline phosphatase, serum creatinine, urine analysis and urine albumin and creatinine, in addition to HbA1c and does not need to be collected in fasted state.
- I Body Mass Index will be calculated automatically.
- J Maximal time window between two visits during titration phase is 5 weeks and during maintenance phase 18 weeks.
- K Calculated based on MDRD formula (see Section <u>5.2.3.4</u>). This formula considers the race as an adjustment factor, therefore, the race must be known (and will be collected) for accurate estimation.

- M Clinically relevant abnormalities found at physical examination, vital signs or ECG that are not pre-existing prior to signing of informed consent (study inclusion) should be reported as adverse event. If such abnormalities already pre-exist prior study inclusion they should be considered as baseline conditions.
- N The End of Treatment Visit (EOT) activities will be performed when a patient discontinues study medication treatment permanently. A follow-up visit will take place 30 days after the EOT visit. Patients who discontinue study drug prematurely should be observed until study end as if they were still receiving blinded study treatment, but no (safety) laboratory sampling (including pregnancy test), ECG or vital signs will be required. If a patient who prematurely discontinued study drug is not willing to return at the pre-defined regular visit schedule at minimum a yearly telephone call and a telephone call at study end (through the patient or alternative person designated by the patient) will be asked for, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit should be recorded.

In some situations, it might be necessary to interrupt study medication temporarily. Patients are encouraged to restart study treatment after an interruption if appropriate in the opinion of the investigator and if not contraindicated. In case the patient is re-instituted on study treatment, the preferred dosage for glimepiride/glimepiride placebo is the dose used before stopping treatment (unless hypoglycaemia was the reason to temporarily stop treatment, see section 4.1.4). In case there is a need for further adjustments after this reinstitution the guidance for treatment initiation should be followed.

O Race of patients will be collected because T2DM treatment results maybe race sensitive. Furthermore, the renal function will be assessed using the MDRD formula. This formula considers the race as an adjustment factor, therefore, the race must be known for accurate estimation.

## **TABLE OF CONTENTS**

| TIT | LE P | AGE | 1 |
|---|---|---|---|
| CLI | NICA | L TRIAL PROTOCOL SYNOPSIS | 2 |
| | | HART | |
| | | OF CONTENTS | |
| | | IATIONS | |
| | | TRODUCTION | |
| 1.<br>1.1 | | MEDICAL BACKGROUND | |
| | | DRUG PROFILE | |
| 2. | | ATIONALE, OBJECTIVES, AND BENEFIT - RISI | |
| 4. | | | |
| 2.1 | | SESSMENT | |
| 2.1<br>2.2 | | RATIONALE FOR PERFORMING THE TRIAL | |
| 2.2 | <u>.</u><br>R | TRIAL OBJECTIVESBENEFIT - RISK ASSESSMENT | ∠∂<br>29 |
| 3. | | SCRIPTION OF DESIGN AND TRIAL | 40 |
| <b>J.</b> | | | 21 |
| 2.1 | | OVERALL TRIAL DESIGN AND BLAN | |
| 3.1 | | OVERALL TRIAL DESIGN AND PLAN | |
| 3.2 | 3.1.1 | | 32 |
| 3.2 | | DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP | 22 |
| 3.3 | | SELECTION OF TRIAL POPULATION | |
| 3.5 | 3.3.1 | | |
| | 3.3.2 | | |
| | 3.3.3 | | |
| | 3.3.4 | Removal of patients from therapy or assessments | |
| | | 3.4.1 Removal of individual patients | |
| | | 3.4.2 Discontinuation of the trial by the sponsor | |
| 4. | TR | EATMENTS | |
| 4.1 | | TREATMENTS TO BE ADMINISTERED | |
| | 4.1.1 | Identity of investigational product(s) | |
| | 4.1.2 | • | |
| | 4.1.3 | Selection of doses in the trial | |
| | 4.1.4 | Drug assignment and administration of doses for each | |
| | | patient | |
| | 4.1.5 | Blinding and procedures for unblinding | |
| | | .5.1 Blinding | |
| | | .5.2 Procedures for emergency unblinding | |
| | 4.1.6 | Packaging, labelling, and re-supply | |
| | 4.1.7 | Storage conditions | |
| 4.3 | 4.1.8 | Drug accountability | 47 |
| 4.2 | 2 | CONCOMITANT THERAPY, RESTRICTIONS, AND RESCUE TREATMENT | 40 |
| | 4.2.1 | Rescue medication, emergency procedures, and addition | |
| | 7.4.1 | treatment(s) | |
| | 4.2.2 | | |


| | 4.2.2.2 Restrictions on diet and life style | |
|---|---|---|
| | 4.2.2.2 Restrictions on diet and me style | 50 |
| 4.3 | TREATMENT COMPLIANCE | 50 |
| <b>5.</b> | VARIABLES AND THEIR ASSESSMENT | 52 |
| 5.1 | | |
| | 5.1.1 Endpoint(s) of efficacy | |
| | 5.1.2 Assessment of efficacy | |
| 5.2 | <b>y</b> | |
| J.2 | 5.2.1 Endpoint(s) of safety | |
| | 5.2.1.1 Reporting waiver for cardiovascular outcome events | |
| | 5.2.2 Assessment of adverse events | |
| | 5.2.2.1 Definitions of adverse events | |
| | 5.2.2.2 Adverse event and serious adverse event reporting | |
| | 5.2.2.3 Oncological adverse events | |
| | 5.2.3 Assessment of safety laboratory parameters | |
| | 5.2.3.1 Haematology | |
| | 5.2.3.2 Clinical chemistry | |
| | 5.2.3.3 Urinalysis | |
| | 5.2.3.4 Renal function impairment | |
| | 5.2.4 Electrocardiogram (ECG) | |
| | 5.2.5 Assessment of other safety parameters | |
| 5.4 | | |
| | APPROPRIATENESS OF MEASUREMENTS | 65 |
| 6. | INVESTIGATIONAL PLAN | 67 |
| 6.1 | INVESTIGATIONAL PLANVISIT SCHEDULE | 67 |
| | INVESTIGATIONAL PLANVISIT SCHEDULE | 67<br>67 |
| 6.1 | INVESTIGATIONAL PLAN<br>VISIT SCHEDULE<br>DETAILS OF TRIAL PROCEDURES AT SELECTED<br>VISITS | 67<br>67 |
| 6.1 | INVESTIGATIONAL PLAN | 67<br>67<br>67 |
| 6.1 | INVESTIGATIONAL PLAN | 67<br>67<br>67<br>68 |
| 6.1<br>6.2 | INVESTIGATIONAL PLAN | 67<br>67<br>67<br>68<br>68 |
| 6.1 | INVESTIGATIONAL PLAN | 67<br>67<br>67<br>68<br>68 |
| 6.1<br>6.2 | INVESTIGATIONAL PLAN | 67<br>67<br>67<br>68<br>68 |
| 6.1<br>6.2 | INVESTIGATIONAL PLAN | 67<br>67<br>67<br>68<br>68<br>DN<br>70 |
| 6.1<br>6.2<br>7. | INVESTIGATIONAL PLAN | 67 67 67 68 68 DN 70 |
| 6.1<br>6.2<br>7.<br>7.1<br>7.2 | INVESTIGATIONAL PLAN | 67<br>67<br>67<br>68<br>68<br>DN<br>70<br>70 |
| 6.1<br>6.2<br>7. | INVESTIGATIONAL PLAN VISIT SCHEDULE | 67 67 67 68 68 DN 70 74 75 |
| 6.1<br>6.2<br>7.<br>7.1<br>7.2 | INVESTIGATIONAL PLAN | 67 67 68 68 70 70 75 77 |

| | 7.3.3 | Safety analyses | 78 |
|---|---|---|---|
| | 7.3.4 | v v | |
| | 7.4 | HANDLING OF MISSING DATA | 80 |
| | 7.5 | RANDOMISATION | |
| | 7.6 | DETERMINATION OF SAMPLE SIZE | |
| 8. | IN | FORMED CONSENT, DATA PROTECTION, | |
| | | RIAL RECORDS | 82 |
| | 8.1 | STUDY APPROVAL, PATIENT INFORMATION, AND | 0_ |
| | 0.1 | INFORMED CONSENT | |
| | 8.2 | DATA QUALITY ASSURANCE | 83 |
| | 8.3 | RECORDS | |
| | 8.3.1 | | |
| | 8.3.2 | | |
| | 8.3.3 | Storage of records | 84 |
| | 8.4 | LISTEDNESS AND EXPEDITED REPORTING OF | |
| | | ADVERSE EVENTS | 84 |
| | 8.4.1 | Listedness | 84 |
| | 8.4.2 | I | |
| | 8.5 | STATEMENT OF CONFIDENTIALITY | |
| | 8.6 | COMPLETION OF TRIAL | |
| | <b>8.7</b> | PROTOCOL VIOLATIONS | |
| | 8.8 | COMPENSATION AVAILABLE TO THE PATIENT IN | |
| _ | | EVENT OF TRIAL RELATED INJURY | |
| 9. | | EFERENCES | |
| | 9.1 | PUBLISHED REFERENCES | |
| | 9.2 | UNPUBLISHED REFERENCES | |
| 1( | ). AI | PPENDICES | 92 |
| | 10.1 | INCLUSION OF ILLITERATE PATIENTS | |
| | 10.1. | 8 | 92 |
| | 10.1. | 2 Patient information and informed consent | |
| | | | 92 |
| | 10.2 | DEFINITIONS OF ENDPOINT EVENTS | 93 |
| | 10.3 | BLOOD PRESSURE MEASUREMENT PROCEDURE AT | |
| | 40.4 | TREATMENT RECOMMENDATIONS | 93 |
| | 10.4 | TREATMENT RECOMMENDATIONS FOR | 0.4 |
| | 10.5 | DYSLIPIDAEMIA SILENT MYOCARDIAL INFARCTION | 94 |
| | 10.5 | | |
| | 10.6<br>10.6. | CLINICAL EVALUATION OF LIVER INJURY 1 Introduction | |
| | | 2 Procedures | |
| | | 3 Decision to Stop Drug Administration | |
| 11 | | JMMARY OF CLINICAL TRIAL PROTOCOL | · · · フ / |
| 11 | | ODIFICATIONS | 0.0 |
| | <b>™</b> /■ | 4 /\ | ~ · · |

BI Trial No.: 1218.74

#### **ABBREVIATIONS**

ACE Angiotensin Converting Enzyme ADA American Diabetes Association

AE Adverse Event

AESI Adverse Event of Special Interest

ALP Alkaline Phosphatase

ALT Alaline transaminase (SGPT) ANCOVA Analysis of covariance

AST Aspartate transaminase (SGOT)

AT-II Angiotensin II

BI Boehringer Ingelheim

BMI Body Mass Index (weight divided by height squared)

BP Blood Pressure CA Competent Authority

CABG Coronary Artery Bypass Graft CEC Clinical Event Committee

CI Confidence Interval CK Creatinine Kinase

CK-MB Creatinine Kinase isoenzyme
CML Clinical Monitor Local

COPD Chronic Obstructive Pulmonary Disease

CRA Clinical Research Associate

CRF Case Report Form

CRO Clinical Research Organisation
CT Computerized Tomography
CTMF Clinical Trial Master File
CTP Clinical Trial Protocol
CTR Clinical Trial Report
CTSU Clinical Trial Supply Unit

CV Cardiovascular

DBP Diastolic Blood Pressure
DILI Drug Induced Liver Injury
DMC Data Monitoring Committee
DPP-IV Dipeptidyl-peptidase IV
ECG Electrocardiogram

eCRF Electronic Case Report Form

EASD European Association for the Study of Diabetes

EOS End Of Study
EOT End Of Treatment

eGFR Estimated Glomerular filtration Rate EudraCT European Clinical Trials Database

EU SmPc European Summary of Product characteristics

FAS Full Analysis Set

FDA Food and Drug Administration

FPG Fasting Plasma Glucose GCP Good Clinical Practice Boehringer Ingelheim 20 April 2016 BI Trial No.: 1218.74

γ-GT Gamma-glutamyl-transferase (GGT)

GI GastroIntestinal

GIP Glucose-dependent Insulinotropic Peptide

GLP-1 Glucagon-like peptide 1
HAs Health Authorities

HbA<sub>1c</sub> Glycosylated haemoglobin HBGM Home Blood Glucose Monitoring HDL-C High Density Lipoprotein - Cholesterol

HR Hazard Ratio

ICH International Conference of Harmonisation

IEC Independent Ethics Committee
INR International Normalized Ratio
IRB Institutional Review Board
ISF Investigator Site File

ITT Intent To Treat
IUD IntraUterine Device
IUS IntraUterine System

IXRS Interactive Voice and Web-based Response System

LADA Latent autoimmune diabetes of adults
LDL-C Low Density Lipoprotein - Cholesterol
LOCF Last Observational Carried Forward

LTFU Lost To Follow Up

MACE Major Adverse Cardiovascular Event MDRD Modification of Diet in Renal Disease

MedDRA Medical Dictionary for Drug Regulatory Activities

MMRM Mixed Model Repeated Measures

MI Myocardial infarction

MRI Magnet Resonance Imaging

NGSP National Glycohemoglobin Standardization Program

NPH Neutral Protamine Hagedorn (insulin)

NYHA New York Heart Association
OAD Oral Antidiabetic Drug

OPU Operative Unit

PCI Percutaneous Coronary Intervention

PG PharmaGenetic p.o. per os (oral) PPS Per Protocol Set

PR Pulse rate

RDC Remote Data Capture

REML Restricted Maximum Likelihood

REP Residual Effect Period
SAE Serious Adverse Event
SBP Systolic Blood Pressure
SC Steering Committee

SU Sulfonylurea

SOP Standard Operating Procedure SPC Summary of Product Characteristics Boehringer Ingelheim 20 April 2016 BI Trial No.: 1218.74

SUSAR Suspected Unexpected Serious Adverse Reaction

TCM Trial Clinical Monitor T2DM Type 2 diabetes mellitus

TDMAP Trial Data Management and Analysis Plan

TG Triglyceride

TIA Transient Ischemic Attack

TMT Trail Making Test

TSAP Trial Statistical Analysis Plan UAP Unstable Angina Pectoris

UKPDS United Kingdom Prospective Diabetes Study

ULN Upper Limit of Normal

#### 1. INTRODUCTION

Linagliptin is an orally available inhibitor of the enzyme dipeptidyl-peptidase IV (DPP-IV) facilitating a decrease of blood glucose levels in type 2 diabetes mellitus (T2DM).

#### 1.1 MEDICAL BACKGROUND

T2DM is a chronic metabolic disease defined by elevated glucose levels that is associated with an increased risk for acute and/or late complications related to the micro- and macrovascular circulation. The latter is primarily related to increased athero-thrombosis that leads to increased morbidity and premature mortality from cardiovascular (CV) disease [R10-0116, P08-06509]. Studies suggest that 70-75% of all deaths in people with diabetes can be attributed to CV complications [R10-0117]. Since hyperglycaemia in itself probably plays a causal role in this, strategies aiming at improving glycaemic control, could contribute in reducing complications and thereby also societies cost.

Strategies for glycaemic management of T2DM; guidelines and limitations

Patients with T2DM are usually treated by combinations of lifestyle and pharmacological interventions and several international guidelines for the treatment of T2DM have been issued [R07-1076, P10-00533, R09-1164, R09-6397, R08-1310, R10-4077, P08-01788. Most guidelines suggest that the therapeutic goal for HbA<sub>1c</sub> should be 6.5-7.0%, which by the use of available tools seem hard to obtain after more than 5-10 years of diabetes duration. A survey in the US (National Health and Nutrition Examination Survey [NHANES] 2003-2004) found that only 57% of participants had HbA<sub>1c</sub> < 7.0% [R10-0133]. Poor control was also noted among the 7000 individuals with T2DM in the Cost of Diabetes in Europe – Type 2 study where only 31% achieved the < 6.5% HbA<sub>1c</sub> goal for HbA1c [R10-0134].

Reasons for this are, amongst other factors, related to a progressive failure of the pancreatic B-cells to compensate for an endogenous insulin resistance by an adequately increased insulin secretion, and the lack of treatment with sustainable effects. Ample evidence tells that lifestyle modification alone, or oral monotherapy, are not sufficient to maintain target levels of glycaemic control in most patients over time. In guidance for the clinician on which pharmacological compounds to use to achieve glycaemic goals amongst patients with T2DM the international guidelines differs slightly [R07-1076, P10-00533, R09-1164, R09-6397, R08-1310, R10-4077, P08-01788]. In general however, all bodies recommend that metformin should be first line treatment, despite its cautions against use in patients with impaired kidney function [P96-4362] where current product information documents include a 'boxed warning' or contraindication for metformin use if estimated glomerular filtration rate (eGFR) is below 60 mL/min/1.73 m<sup>2</sup> [R10-4375]. Besides this also acute diabetic ketoacidosis, acute conditions with the potential to alter renal function acute or chronic disease which may cause tissue hypoxia, hepatic insufficiency, acute alcohol intoxication and alcoholism, are contraindications against its use. In a UK population study (published in Diabetic Medicine 2001;18:483-488), Emslie-Smith et al found that 6.4% of all patients with T2DM had some of these contraindications against using Boehringer Ingelheim 20 April 2016 BI Trial No.: 1218.74

this drug. Further limitations of metformin is gastrointestinal (GI) side effects [R10-4375] that e.g. in the A Diabetes Outcome Prevention Trial (ADOPT) affected more than 1/3 of the participants [R09-6400]. However, despite these limitations, this compound is the most widely used and has a good safety profile and also has some degree of support for being cardio protective [R09-6405, R09-6409], or at least without associated cardiotoxicity. Most other drugs on the market lack such documentation.

As a second line treatment, because of the progressive loss of \$\beta\$-cell function in T2DM, traditional insulin secretagogues such as the sulfonylureas (SUs) that stimulate to insulin secretion in a non-glucose-dependent manner is widely used; in fact it is the most used second line therapy. However, this treatment carries an increased risk for hypoglycaemia and weight gain [R09-6400] and, as for metformin, is also associated with a lack of sustainable effect [R09-6400]. Therefore, international treatment guidelines have opened for the use of other drugs, e.g. insulins, glitazones, glinides and alpha-glucosidase inhibitors, to be used as 2nd line or 3rd line in certain settings. However, most these drugs have also some side effects that limit their use, e.g. hypoglycaemia, weight gain, GI side effects and peripheral oedema. This could even also have prognostic implications since hypoglycaemia and weight gain was recently postulated as contributors to the adverse outcomes in the "Action to Control Cardiovascular Risk in Diabetes" (ACCORD) [R09-6407] and in the Veterans Affairs Diabetes trial (VADT) serious hypoglycaemia was the 2nd strongest predictor for developing a new myocardial infarction (MI) [R09-6408].

Since CV caveats with drugs to treat T2DM, historically also have been found to arise at relatively late stage; just before, or even after, the compound reached the market, regulating authorities such as the US Food and Drugs Administration (FDA) has issued some guidance to industry in order to rule out potential excessive morbidity and mortality potentially associated with all new drugs for the treatment of T2DM [R09-2151]. Such an assessment could involve dedicated trials. Having seen the potential limitations of drugs that are associated with weight gain and hypoglycaemia it is therefore of interest to explore novel treatment options that offer glycaemic reduction without associated such side effects.

#### Emerging treatment for T2DM; DPP- IV inhibitors

The incretin effect is a phenomenon where the glucose-dependent insulin secretion is augmented by intestinally derived peptides (i.e. incretins), which are released in the presence of glucose or nutrients in the gut and thereby contribute to the maintenance of long term and post-meal glycaemic control. Glucagon like peptide 1 (GLP-1) is an important member of the incretin hormone family and accounts, together with glucose-dependent insulinotropic peptide (GIP), for more than 50% of the incretin effect in humans [R09-6409]. These hormones are almost instantaneously inactivated by the enzyme DPP-IV. DPP-IV is widely expressed in many tissues including kidney, liver, intestine, lymphocytes and vascular endothelial cells. Since postprandial GLP-1 secretion has been reported to be attenuated in T2DM [R09-6409], a prolongation of the half-life of GLP-1 by DPP-IV inhibition has been proven as a therapy. Besides its stimulatory effects on insulin secretion, that depend on the actual glucose concentration [R09-6409], resulting in a reduction of HbA<sub>1c</sub>, GLP-1 has also

been shown to inhibit glucagon secretion, to delay gastric emptying, to induce satiety, and, in animal models, to maintain long-term \(\beta\)-cell function. Especially the maintenance of \(\beta\)-cell function is of interest, that, if also would be the case in humans, would represent the first modulating therapy of the T2DM. However, no long term studies in human have actually confirmed this yet. An added interesting feature of this therapeutic option is that it seems to be associated with no weight gain and no hypoglycaemia (at least in monotherapy).

### Study proposal

In this large-scale intervention trial we will test the impact of treatment with the DPP-IV inhibitor linagliptin head-to-head versus a SU (glimepiride) on CV safety and efficacy. The study will be given the acronym **CAROLINA** (**Cardio**vascular safety of **lina**gliptin).

#### 1.2 DRUG PROFILE

The DPP-IV inhibitor compound linagliptin was discovered by Boehringer Ingelheim [BI] Pharma GmBH & Co. KG, Biberach, Germany.

Linagliptin is a potent inhibitor of DPP-4 activity and prolongs the half-life of GLP-1. This has been shown in vitro, in various animal models, and in clinical trials. Linagliptin is an orally available compound with a low risk for hypoglycaemic episodes [U04-1767].

#### Clinical Pharmacokinetics

In earlier PK trials, linagliptin showed nonlinear PK in the therapeutic dose range, with a less than dose proportional increase in plasma concentrations. Clearance, volume of distribution, and amount excreted unchanged in urine increased with increasing doses, possibly due to nonlinear protein binding. Linagliptin was predominantly excreted unchanged in faeces. Renal excretion was considered to be a minor elimination pathway. No dose adjustment of linagliptin based on hepatic impairment, renal impairment, age, body mass index (BMI), weight, gender, or race is considered necessary. Linagliptin showed no clinically relevant interaction with metformin, pioglitazone, glyburide or empagliflozin.

#### Clinical efficacy and safety

Treatment with 5 mg linagliptin once daily has resulted in clinically meaningful and statistically significant reductions in HbA<sub>1c</sub>, FPG, and postprandial glucose. There is a consistent pattern in the improvement in HbA<sub>1c</sub> levels when linagliptin was used in patients with different background therapies. These findings demonstrate efficacy for up to 18 to 24 weeks duration for different background therapies and are further supported by trials of longer duration up to 104 weeks.

Overall, in phase III studies the overall incidence of adverse events (AEs), drug related AEs, AEs of severe intensity, AEs leading to discontinuation, and serious AEs (Serious Adverse Event, SAEs) were very similar across studies, with linagliptin being mostly comparable with placebo. For description of side effects of linagliptin

refer to the current Investigator's Brochure [ $\underline{U04-1767}$ ] and the local prescribing information for linagliptin.

# 2. RATIONALE, OBJECTIVES, AND BENEFIT - RISK ASSESSMENT

#### 2.1 RATIONALE FOR PERFORMING THE TRIAL

The aim of the present study is to investigate the long–term impact on CV morbidity and mortality and relevant efficacy parameters (HbA $_{1c}$ , fasting plasma glucose, treatment sustainability) of treatment with linagliptin in a relevant population of patients with T2DM and compare outcome against one compound of the second most used OAD class, i.e., SU (glimepiride). To date this has not been tested in a long-term trial; as also is the case for other DPP-IV inhibitors. However, there are currently no safety signals that indicate that linagliptin should be inferior to glimepiride in this respect. A recent meta-analysis of the marketed DPP-IV inhibitors on the contrary indicates a potential beneficial CV effect of DPP-IV inhibitors as a class; although this meta-analysis mainly included trials of shorter duration where trial participants were not at a particular high CV risk, leaving the findings as hypothesis generating [R09-6410].

Since most guidelines state that metformin should be first line treatment, this study will in principal be conducted as add-on to metformin background. Since a relatively large proportion of patients with T2DM have some degree of contraindications or intolerance to metformin, or local guidelines may indicate other treatments as first line therapy, the study is also open for inclusion of patients being treatment naïve or on other antidiabetic treatments as specified in Section 3.3.2. In brief, the patients included might be OAD naïve (due to contraindications or intolerant to first line treatment), previously receiving monotherapy with metformin, any SU, any glinide or any alpha-glucosidase inhibitor or previously on dual therapy with metformin + SU, metformin + glinide, metformin + alpha-glucosidase inhibitor, SU + alpha-glucosidase inhibitor or glinide + alpha-glucosidase inhibitor.

Hence, the study has two study arms: linagliptin or glimepiride as monotherapy or as add-on to other allowed treatments. The study design is described in more detail in Section 3.1.

Allowing this will generate a trial population with a short to moderate diabetes duration with a high CV risk (e.g., due to renal impairment, chronic cardiac disease or a recent MI, advanced age) to participate, thereby it will assess the CV safety profile of the drug as compared to one of the most widely used oral antidiabetic drug (OAD) globally (i.e. glimepiride) in a broad and relevant population of patients with T2DM. This study design therefore also concurs with the recent FDA guidelines for target population whom to in particular address CV risk of novel OADs in T2DM [R09-2151] and will also be an integral part of the ongoing CV safety assessment for linagliptin and data will also be used to support regulatory submission.

#### 2.2 TRIAL OBJECTIVES

The primary objective is to demonstrate non-inferiority (by means of comparing the upper limit of a two-sided (1-2\*alpha)\*100% confidence interval with the noninferiority margin of 1.3) of treatment with linagliptin in comparison to glimepiride (as monotherapy or as add-on therapy) with respect to time to first occurrence of any of the adjudicated components of the primary composite endpoint (i.e. cardiovascular death, non-fatal stroke or non-fatal myocardial infarction (excluding silent MI) in patients with type 2 diabetes mellitus. If the non-inferiority hypothesis with margin 1.3 has revealed a significant result, then secondly, the primary composite endpoint will be tested with a superiority hypothesis. If the superiority test has revealed a significant result, then thirdly the first key secondary endpoint of time to first occurrence of any of the adjudicated components of cardiovascular death, non-fatal stroke, non-fatal myocardial infarction (excluding silent MI) or hospitalisation for unstable angina pectoris will be tested hierarchically with a superiority hypothesis. If the test of the first key secondary hypothesis has revealed a significant result, then fourthly the second key secondary endpoint will be tested hierarchically. If the test of the second key secondary hypothesis has revealed a significant result, then fifthly the third key secondary endpoint will be tested hierarchically.

Other objectives are to compare  $HbA_{1c}$  change from baseline, the incidence of hypoglycaemia, weight gain and treatment sustainability defined as the proportion of patients that are on study treatment at study end without need for rescue medication, that at Final Visit maintain glycaemic control ( $HbA1c \le 7.0\%$ ).

For a description of the endpoints chosen and statistical analyses to assess these objectives, please refer to Section  $\underline{5}$  and  $\underline{7}$ .

#### 2.3 BENEFIT - RISK ASSESSMENT

Potential general benefits for study participants in this trial (irrespective of investigational drug received, i.e. linagliptin or glimepiride) are 1) improvements in glycaemic control, 2) improvements of other CV risk factors and 3) general medical benefit from careful and close monitoring by medical personnel during the study. Further, the participants can contribute to generate a potential future benefit for larger groups of patients with T2DM by participating in this clinical trial if linagliptin fulfils much of its promises as a future treatment of T2DM.

General risk associated with participating is related to trial specific procedures such as blood sampling that can be associated with bruising and pain. The amount of blood taken during the whole course of the trial is not believed to be associated with any discomfort for the patients.

20 April 2016

#### Investigational drug specific risk

Glimepiride is a drug that has been on the market for a long time, is widely used and therefore is believed to be well characterized in term of risk profile. Patients randomised to glimepiride can nevertheless experience hypoglycaemia as a consequence of its mode of action. However, in a cohort of patients with T2DM of short-to-moderate duration this risk is relatively small as was seen in the UKPDS where yearly rate of severe hypoglycaemia was 1.0% for chlorpropamide (a first generation SU) and 1.4% with glibenclamide (a second generation SU) [R04-2173]. Also, there is a certain risk for patients to gain weight with this treatment; however not all trials with glimepiride has shown a weight increase [R09-6394].

Linagliptin from its clinical phase III testing has shown a "placebo-like" safety profile. It carries a low risk for inducing hypoglycaemia and weight gain. However, linagliptin has by far not the same cumulative exposure compared to glimepiride. Safety will be ensured by monitoring the patients for AEs both clinically and by laboratory testing. If any investigator should have a clinical concern, the safety of the patients will be of paramount importance. Given the large safety margin derived from the toxicology studies, the wide therapeutic window of linagliptin, the very good tolerability seen in previous trials in subjects with T2DM, and the monitoring throughout the trial the sponsor is of the opinion that the risks for the participating patients are minimal and justified when compared to the potential benefits of a successful clinical development of linagliptin for patients with T2DM.

Pioglitazone, metformin, alpha-glucosidase inhibitor or basal insulin could be used in this trial as rescue therapy (see Section 4.2.1). Pioglitazone has been extensively tested and has been associated with CV benefits [R09-6395]. However, some side effects might occur with this drug; i.e. weight gain, peripheral oedema, osteopenia and heart failure. The latter is however relatively infrequent and occurs in those susceptible to this. In combination with SU also hypoglycaemia risk is increased.

Metformin might be used as rescue therapy; however BI expects that the proportion of patients that would be eligible for this would be low due to our inclusion criteria. However, metformin is associated with side effects as gastrointestinal discomfort, nausea and increases also the risk of hypoglycaemia.

An alpha-glucosidase inhibitor may also be used as rescue therapy to maintain glycaemic control; however BI expects that the proportion of patients that would accept this treatment predominantly would be in the Asian study population due to the higher usage of this drug in this region. Side-effect of alpha-glucosidase inhibitors includes gastrointestinal discomfort, diarrea, nausea and increases also the risk of hypoglycaemia, in particular if combined with SU.

Insulin might, as per all international guidelines, be expected required to certain patients as other OADs fail to control blood glucose levels adequately. Basal insulin (i.e. intermediate or long-acting insulin) is all widely used. Side effects of these are weight gain and hypoglycaemia. Some insulins also require need for re-suspension (at least NPH insulin) and they all need to be subcutaneously injected.

Boehringer Ingelheim BI Trial No.: 1218.74

20 April 2016

#### Pregnancy

Metformin, alpha-glucosidase inhibitors, glimepiride, pioglitazone, most of the long acting insulin analogues and linagliptin are not approved for use in pregnancy. In the embryofoetal and fertility studies in rats and rabbits with linagliptin, no effects on early embryonic development, mating, male and female fertility, and bearing live young were observed up to and including the high dose group given 240 mg/kg. Therefore, women who are of child-bearing potential will be included in this study provided that they are using adequate contraceptive methods.

#### *Induced liver injury*

Based on principal considerations, there is always the possibility that so fare unknown safety issues are upcoming. One of those issues is drug induced liver injury. Albeit there was no risk identified so far, this study will follow a careful protocol to follow-up laboratory alterations of liver parameters in order to safeguard patients' safety and to stay in compliance with international regulatory requirements. Although rare, drug induced liver injury is under constant surveillance by sponsors and regulators. This study requires follow-up and expedited reporting of laboratory alterations of selected liver laboratory parameters to ensure patient safety and to remain compliant with international regulations.


## 3. DESCRIPTION OF DESIGN AND TRIAL POPULATION

#### 3.1 OVERALL TRIAL DESIGN AND PLAN

This multicentre, multinational, randomised, double-blind, parallel group, comparator -controlled study compares treatment with linagliptin (5 mg once daily) to treatment with glimepiride (1-4 mg) as monotherapy or as add-on therapy to metformin and/or other antidiabetic treatment as specified in Section 3.3.2.

The trial is event driven and will run with an estimated number of 6000 patients for an estimated treatment time of 432 weeks, beginning with the randomisation of the first patient. In the case the number of events is not or may not be reached within this period the trial duration and/or the number of patients enrolled will be increased until the defined number of adjudicated primary events is reached.

Patients will enter an open-label placebo (add-on) run-in period of 2 up to 4 weeks before randomisation. Patients who successfully complete at least two weeks of the placebo-run (should have a treatment compliance between 80% to 120%) and who still meet the inclusion/exclusion criteria will be randomised to receive either linagliptin or glimepiride. Patients who do not successfully complete at least two weeks of the placebo run-in, may continue the placebo run-in phase up to four weeks to meet the compliance criterion as specified above. Any SU or glinide will be discontinued at randomisation Visit 2 (SU/glinide should not be taken in the morning of Visit 2).

The randomised treatment will be double-blind within the dose groups of linagliptin and glimepiride (i.e. each patient will receive one active treatment and placebo matching the alternative active treatment in a double-dummy design).



Figure 3.1: 1 Treatment periods and treatment groups in the trial design

For all patients, contacts are scheduled at regular time intervals (see flow chart). The estimated treatment duration for the first randomised patient is 432 weeks. The End of Treatment Visit (EOT) activities will be performed when a patient discontinues study medication permanently. Patients who discontinue study drug prematurely should be observed until study end as if they were still receiving blinded study treatment, but no (safety) laboratory sampling (including pregnancy test), ECG or vital signs will be required. If a patient who prematurely discontinued study drug is not willing to return

at the pre-defined regular visit schedule at minimum a yearly telephone call and a telephone call at study end will be asked for (through the patient or alternative person designated by the patient), to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit should be recorded.

All patients will have a follow up visit 30 days following completion of the treatment period. The follow-up visit may be performed as a phone visit for patients who completed the planned treatment period and who do not have any abnormalities at the EOT visit (only adverse events/outcome events and changes in concomitant therapy to be obtained).

The number of confirmed adjudicated primary endpoint events will be continuously monitored during the trial. Based on the available number of events the projected number of expected future events will be calculated. As soon as the projection reliably suggests that the total number of patients with a by adjudication confirmed primary endpoint event will reach 631, the trial team will perform respective actions to stop the trial. From this time point on, all patients are expected to perform their last visit (EOT visit) within the proposed time schedule, communicated via an investigator letter. A follow-up visit will take place 30 days after the EOT visit.

In case early study termination is to be performed (e.g. based on recommendation by the DMC), a reasonable timeframe to stop the trial (perform last patient visits) will be defined and communicated to the investigators.

#### 3.1.1 Administrative structure of the trial

The study is sponsored by Boehringer Ingelheim. The following committees will participate in the conduct of the trial, their specific functions are summarised below:

#### **Steering Committee**

A Steering Committee (SC) will have a scientific and clinical advisory function in the study. The Steering Committee is composed by university and sponsor based scientists with clinical and methodological expertise.

#### **Data Monitoring Committee**

An independent Data Monitoring Committee (DMC) will review safety and efficacy data and make recommendations whether to continue the study, continue the study with modifications, or terminate the study. The DMC analyses and operations will be formally separated from the sponsor, the investigators and the steering committee.

#### **Clinical Event Committees**

The study is set up with prospective adjudication of all cardio/cerebrovascular pancreatic trigger events. The prospectively defined adjudication process will assess cardiac and neurological vascular events through an independent, blinded, external Clinical Event Committee (CEC). Details on the composition of the committee, its

procedures and interactions are provided in a separate CEC Charter. Additionally, a separate independent, blinded, external committee will be set up for adjudication of pancreatic events. The adjudication process for these events will be clarified in a separate CEC charter.

## 3.2 DISCUSSION OF TRIAL DESIGN, INCLUDING THE CHOICE OF CONTROL GROUP

According to current guidelines of the ADA/EASD, metformin should be initiated concurrently with lifestyle intervention at diagnosis in patients newly diagnosed with T2DM when  $HbA_{1c} > 7.0\%$  and be titrated to a maximum tolerated dose (up to 2x 1000 mg/day or total 2500 mg/day) [R09-1164]. Therefore, patients enrolling on metformin monotherapy represent an important proportion of patients with T2DM. However, contraindications or intolerance to metformin due to e.g. congestive heart failure or severe renal impairment also constitutes a significant amount of people with T2DM. Further, local guidelines may indicate other first line treatment. Therefore this trial also allows for patients that are treatment naïve or are on other antidiabetic treatments as specified in Section 3.3.2.

Treatment with linagliptin is compared against glimepiride, a drug from the second most widely used antidiabetic class after metformin (i.e. SUs). Treatment goal for HbA<sub>1c</sub> is in this trial, according to most international guidelines,  $\leq 7.0\%$ . During the trial additional therapy ("rescue therapy") is allowed, and encouraged, if HbA<sub>1c</sub> > 7.5% during maintenance phase. This is considered important as to ensure that an optimal level of standard of care is reached. However, the decision to initiate rescue medication remains with the investigator and the appropriate local treatment guidelines.

The protocol also encourages the investigators to treat all other CV risk factors (lipid levels, blood pressure, micro/macroalbuminuria, unhealthy lifestyle, smoking) according to an optimal level of standard of care. In a high CV risk population this usually implies liberal use (if tolerated or not contraindicated) of statins, ACE-inhibitors, AT-II receptor blockers, aspirin, beta-blockers, calcium channel blockers, etc.). This should be conducted in the context of local or regional guidance for primary or secondary CV prevention.

The treatment period is planned for up to an estimated 432 weeks. The treatment period will be followed by a follow-up period of 30 days.

#### 3.3 SELECTION OF TRIAL POPULATION

Approximately 10000 patients will be screened for the trial in about 45 countries. Approximately 700 trial centres will be participating to randomise the estimated number of 6000 patients.

Participating sites are expected to randomise a least 8 patients. Investigators who fail to randomise at least one study subject in the first 12 weeks of the trial may be excluded from further participation. If enrolment is delayed, additional centres may be recruited.

Screening of patients for this trial is competitive, i.e. screening for the trial will stop at all centres when a sufficient number of patients has been randomised to trial treatment. Investigators will be notified when the appropriate number of patients has been screened and screening is complete, and will not be allowed to recruit additional patients for this study. Patients who have completed Visit 1a procedures prior to notification of the termination of recruitment will be allowed to continue in the study, if they meet all entry criteria.

The check for subject eligibility will be based upon a complete medical history including a physical examination and clinical laboratory tests. Judgement of the clinical relevance of a concomitant disease is at the discretion of the investigator. Conditions under therapy are always clinically relevant.

A log of all patients included into the study (i.e. having given informed consent) will be maintained in the ISF at the investigational site irrespective of whether they have been treated with investigational drug or not.

Re-screening and/or re-testing (of assessments) is permitted under certain circumstances. Whilst the information provided below is not an exhaustive list, it provides some guidance as to when such re-screening and/or re-testing would be considered appropriate. If a site is in any doubt as to whether re-screening and/or re-testing is appropriate in their particular situation, then clarification should be sought with the CML.

#### Re-testing:

Re-testing is only to be performed for a lab result which is obviously received beyond stability at the central laboratory or thought to be a spurious result. It is not permitted to perform re-testing (in any time window after V1a sampling) for HbA<sub>1c</sub> when it does not meet the study criteria only.

#### Re-screening:

- Re-screening of the same patient is only allowed once.
- The patient should be declared a screening failure in the eCRF/RDC with their original patient number.
- Upon re-screening, the next available (= new) patient number should be selected from RDC.
- The patient must be re-consented using the current approved version of the information sheet and consent form.
- There is no time limit for re-screening as long as the patient fits the eligibility criteria they could be re-screened whenever the investigator feels they may become eligible.

#### 3.3.1 Main diagnosis for study entry

Patients with documented diagnosis of T2DM with insufficient glycaemic control and at high risk of CV events prior to informed consent can be enrolled in the study. Any antidiabetic background medication at Visit 1a should be on a stable (unchanged) daily dose for at least 8 weeks. There is no short term use of insulin within 8 weeks prior informed consent. Background medication should be stable during screening/run-in phase to allow randomisation.

As local guidelines for management of T2DM will be followed, treatment naive T2DM patients should be offered first line anti-diabetic treatment (e.g. metformin) before allowing them for study inclusion, unless they have specific contra-indications or intolerances to its use (see also Section 2.1).

Prior SU or glinide treatment will be discontinued at Visit 2, whereas if medications such as metformin and alpha-glucosidase inhibitor are being used, these should be continued.

#### 3.3.2 Inclusion criteria

- 1) Documented diagnosis of T2DM and concurrently 2) insufficient glycaemic control and a high risk of CV events 3) prior to informed consent.
- 2) Insufficient glycaemic control (at Visit 1a) defined as:
  - a)  $HbA_{1c}$  <u>6.5 8.5%</u> (48 69 mmol/mol) while patient is treatment naïve (if intolerant or contra-indicated to first line anti-diabetic treatment) or treated with:
  - metformin monotherapy, or
  - alpha-glucosidase inhibitor monotherapy (e.g. acarbose, voglibose), or
  - metformin + alpha-glucosidase inhibitor (e.g. acarbose, voglibose), or
  - b) HbA<sub>1c</sub> 6.5 7.5% (48 58 mmol/mol) while patient is treated with
  - sulphonylurea (SU) monotherapy, or
  - glinide monotherapy (e.g. repaglinide, nateglinide), or
  - metformin + SU (combination maximal up to 5 years), or
  - metformin + glinide (combination maximal up to 5 years), or
  - sulphonylurea + alpha-glucosidase inhibitor (combination maximal up to 5 years), or
  - glinide + alpha-glucosidase inhibitor (combination maximal up to 5 years)
- 3) High risk of CV events defined as any one (or more) of A), B), C) or D):
  - A) Previous Vascular Disease:
    - Myocardial infarction (> 6 weeks prior to informed consent)


- Documented coronary artery disease (≥ 50% luminal diameter narrowing of left main coronary artery or ≥ 50% in at least two major coronary arteries in angiogram) Note: CT or MRI detection of this will not suffice for inclusion; only invasive angiography. The left main coronary artery is often abbreviated to LCA or LCMA. As this is a very important artery that is branched to other major arteries it suffices to have a ≥ 50% stenosis in this artery (any segment) for inclusion. If there are no stenosis in this artery patient could be included if patient has a ≥ 50% stenosis in two, or more, of the other major coronary arteries (any segment): LAD (Left Anterior Descending; also called AIB = Anterior interventricular branch), CX (= art. Circumflex, also called CB=Circumflex branch) or RCA (right coronary artery).

- Percutaneous Coronary Intervention (PCI) > 6 weeks prior informed consent
- Coronary Artery By-pass Grafting (CABG) > 4 years prior to informed consent or with recurrent angina following surgery
- Ischemic or hemorrhagic stroke (> 3 months prior to informed consent)
- Peripheral occlusive arterial disease (previous limb bypass surgery, stenting or percutaneous transluminal angioplasty; previous limb or foot amputation due to circulatory insufficiency, angiographic or ultrasound detected significant vessel stenosis (> 50%) of major limb arteries (common iliac artery, internal iliac artery, external iliac artery, femoral artery, popliteal artery), history of intermittent claudication, with an ankle: arm blood pressure ratio < 0.90 on at least one side).

#### B) Evidence of vascular related end-organ damage:

- Moderately impaired renal function (as defined by modified diet of renal disease (MDRD) formula) with estimated glomerular filtration rate [eGFRF]) 30-59 mL/min/1.73 m<sup>2</sup>
- Random spot urinary albumin: creatinine ratio  $\geq$  30 µg/mg ( $\geq$  3.4 mg/mmol) in two of three unrelated specimens in previous 12 months prior Visit 1a
- Proliferative retinopathy defined as retinal neovascularisation or previous retinal laser coagulation therapy.

#### C) Age $\geq 70$ years (at Visit 1a)

#### D) At least two of the following CV risk factors:

- Type 2 diabetes mellitus duration > 10 years at Visit 1a.
- Current\* systolic blood pressure (SBP) > 140 mmHg (or on at least one blood pressure lowering treatment at Visit 1a)
- Current daily cigarette smoking
- Current\* LDL cholesterol ≥ 135 mg/dL (3.5 mmol/L) (or specific current treatment for this lipid abnormality at Visit 1a).
- \* Current = Blood pressure or LDL cholesterol measurement < 6 months prior V1a.


Note: To ensure appropriate representation of patients from the different cardiovascular risk categories (A-D), the trial team will monitor the proportion of patients being recruited into these categories (trial level, and by region and/or country). In consultation with the steering committee, limitation of recruitment of a particular category may be arranged (trial level, or per region and/or country level). This process will be implemented to ensure a proper distribution of CV risk categories worldwide.

If a patient fulfils more than one CV risk category all CV risk categories will be indicated in the CRF. For CV risk distribution the patient will be allocated to highest CV risk category. CV risk category A is relatively highest category, followed by B, C, D.

Examples: if patient is at age of 71 years and has T2DM > 10 years and is currently smoking, this patient will be allocated to category C.

A patient with vascular end-organ damage and previous stroke will be allocated to category A.

Patients may be included if any criterion A - D is fulfilled as long as it is not in conflict with any other exclusion criteria. Example: a patient at age 73 years may be included [fulfils criterion C] in case CABG was conducted two years ago.

If a patient fulfils CV risk category A, C and/or D <u>and</u> has only one albumin creatinine ratio  $\geq 30~\mu g/mg$  in previous 12 months prior Visit 1a, and an albumin creatinine ratio  $\geq 30~\mu g/mg$  at V1a, such patient will also be identified as Cat. B patient in the CRF. The patient will be allocated to highest CV risk group for (A or B).

In consultation with the Steering Committee, enrolment of patients currently at least on SU or glinide may be limited.

- 4) Body Mass Index (BMI)  $\leq$  45 kg/m<sup>2</sup> at Visit 1b.
- 5) Age  $\geq$  40 and  $\leq$  85 years at Visit 1a
- 6) Signed and dated written informed consent at the latest by the date of Visit 1a, in accordance with GCP and local legislation
- 7) Stable anti-diabetic background medication (unchanged daily dose) for at least 8 weeks prior V1a and without short term use of insulin. Background medication should be stable during screening/run-in phase to allow randomisation.

#### 3.3.3 Exclusion criteria

- 1) Type 1 diabetes mellitus
- 2) Any history and/or current treatment with other antidiabetic drugs (e.g. rosiglitazone, pioglitazone, GLP-1 analogue/agonists, DPP-IV inhibitors or any insulin) prior to informed consent.
  - Note 1: This also includes clinical trials where these antidiabetic drugs have been provided to the patient. Note 2: Previous short term use of any insulin (up to two consecutive weeks) is allowed (e.g. during hospitalisation) if taken at least 8 weeks prior informed consent
- 3) Treatment with anti-obesity drugs 3 months prior to informed consent
- 4) Uncontrolled hyperglycaemia with a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast during placebo run-in and confirmed by a second measurement (not on the same day).
- 5) Active liver disease or impaired hepatic function, defined by serum levels of either ALT (SGPT), AST (SGOT), or alkaline phosphatase above 3 x upper limit of normal (ULN) as determined at Visit 1a.
- 6) Any previous (or planned within next 12 months) bariatric surgery (open or laparascopic) or intervention (gastric sleeve)
- 7) Pre-planned coronary artery re-vascularisation (PCI, CABG) within next 6 months after V1a or any previous PCI and/or CABG  $\leq$  6 weeks prior informed consent
- 8) Known hypersensitivity or allergy to the investigational product or its excipients, or glimepiride (or the SU class).
- 9) Inappropriateness of glimepiride treatment for renal safety issues or other issues (e.g. allergy) according to local prescribing information
- 10) Congestive heart failure of NYHA class III or IV
- 11) Acute or chronic metabolic acidosis (present condition in patient history)
- 12) Hereditary galactose intolerance
- 13) Alcohol or drug abuse within the 3 months prior to informed consent that would interfere with trial participation
- 14) Current treatment with systemic corticosteroids at time of informed consent or pre-planned initiation of such therapy. Note: inhaled use of steroids (e.g. for

asthma/COPD) is no exclusion criterion, as this does not cause systemic steroid action.

- 15) Change in dose of thyroid hormones within 6 weeks prior informed consent
- 16) Participation in another trial with an investigational drug given within 2 months prior to informed consent
- 17) Pre-menopausal women (last menstruation ≤ 1 year prior to informed consent) who:
  - are nursing or pregnant,
  - or are of child-bearing potential and are not practicing an acceptable method of birth control (acceptable methods of birth control include tubal ligation, transdermal patch, intra uterine devices/systems (IUDs/IUSs), oral, implantable or injectable contraceptives, sexual abstinence (if allowed by local authorities), double barrier method and vasectomised partner) or do not plan to continue using acceptable method of birth control throughout the study and do not agree to submit to periodic pregnancy testing during participation in the trial.
- 18) Patients considered unreliable by the investigator concerning the requirements for follow-up during the study and/or compliance with study drug administration, has a life expectancy less than 5 years for non-CV causes, or has cancer other than non-melanoma skin cancer within last 3 years, or has any other condition than mentioned which in the opinion of the investigator, would not allow safe participation in the study
- 19) Acute coronary syndrome  $\leq 6$  weeks prior to informed consent
- 20) Stroke or TIA  $\leq$  3 months prior to informed consent

#### 3.3.4 Removal of patients from therapy or assessments

#### 3.3.4.1 Removal of individual patients

This is a long-term safety outcome study and every effort should be made by the site staff to encourage patients to remain in the study and on study drug if medically safe. Patients who prematurely discontinue study drug should remain in the study and should be observed until study end, preferably at the study time points as pointed out in the Flow Chart.

If a patient who prematurely discontinued study drug is not willing to return at the pre-defined regular visit schedule, at minimum a yearly telephone call (preferably every 6 months) and a telephone call at study end (through the patient or alternative person designated by the patient) will be required, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit should be recorded. Every attempt will be made by the investigator to ensure patients continue participating in the study during study drug interruptions and after discontinuation of study drug.

Patients who prematurely discontinue study medication are allowed to restart the study medication at any time if appropriate in the opinion of the investigator and if not contraindicated. In this study, patients are allowed to have multiple study drug interruptions. There is no limit on either the number of study drug interruptions or the maximum length of any study drug interruption. Investigators should routinely consider re-starting study drug at every visit following study drug discontinuation.

A patient could be instructed to stop the study drug only after discussion between sponsor representative and investigator, if eligibility criteria are being violated, or if the patient fails to comply with the protocol (e.g. non-attendance at study assessments). Early discontinuation of study medication is not a criterion for withdrawal of consent for participating in the study.

If determined by investigator as necessary for patient safety, new antidiabetic medication regimen can be started immediately after discontinuation of study treatment and must be recorded in the eCRF (see further details in Section 4.2).

If a patient becomes pregnant during the trial the study treatment will be stopped, the patient will be followed up during the study and until birth or otherwise termination of the pregnancy (see further details in Section 5.2.2.2)

If pancreatitis is suspected, the study treatment should be stopped.

Patients who drop out during the screening/run-in phase prior to randomisation (Visit 2) will be considered a screening failure. They have to be recorded as screening failure in eCRFs and no further follow-up is required.

Patients who withdraw or discontinue from the study after randomisation will not be replaced.

If a patient needs to take concomitant drugs that interfere with the investigational product (or other study medications) or in the occurrence of hypoglycaemia that may put the patient at risk with continued participation (e.g. repeated hypoglycaemic episodes) the trial medication can be discontinued temporarily, or if needed permanently. Since this is an outcome study, the primary analysis will be performed based on all randomised patients who were treated with at least one dose of study drug. Therefore investigators are encouraged to re-administer study medication to a randomised patient if there are no further safety concerns.

A patient has the right to withdraw informed consent for participation at any time for any reason. However, withdrawal of consent from study participation should be very rare and unusual. Because of this, the investigator must be involved in the discussions with the patient regarding a withdrawal of consent.

If the patient withdrew informed consent the patient should stop taking study medication and should be asked to complete the study ending tests and procedures as described in the <u>Flow Chart</u> for End of Treatment Visit and Visit 33 (Follow up visit). Completing these procedures is strongly recommended for the patient's safety. The

Doc No.: c01618200-19

20 April 2016


reason for discontinuing treatment will be recorded in the eCRF. The data will be included in the trial database and will be reported.

For patients that have withdrawn informed consent, the patient will be asked to resign an informed consent form, which will allow to enquire at least about the patient's vital status and occurred outcome events through contacts to relatives, acquaintances, family physicians, hospital records, etc.

**Protocol Revision 6** 

If patients who discontinue from treatment after randomisation could not be followed-up until the end of study (i.e. at least the vital status could not be collected) those patients will be indicated as Lost To Follow Up (LTFU). The number of LTFU patients should be limited.

The End of Treatment Visit (EOT) activities will be performed when a patient discontinues study treatment permanently.

A follow-up visit will take place 30 days after the EOT visit. Patients who discontinue study drug prematurely should be observed until study end as if they were still receiving blinded study treatment, but no (safety) laboratory sampling (including pregnancy test), ECG or vital signs will be required. If a patient who prematurely discontinued study drug is not willing to return at the pre-defined regular visit schedule at minimum a yearly telephone call and a telephone call at study end will be required, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit might be recorded.

Patients should keep their antidiabetic medication stable for the course of the trial (except prior SU or glinide treatment which should be stopped at V2. SU/glinide should not be taken in the morning of Visit 2).

## 3.3.4.2 Discontinuation of the trial by the sponsor

Boehringer Ingelheim reserves the right to discontinue the trial overall or at a particular trial site at any time for the following reasons:

- 1. Failure to meet expected enrolment goals overall or at a particular trial site,
- 2. Emergence of any efficacy/safety information that could significantly affect continuation of the trial,
- 3. Violation of GCP, the CTP, or the contract by a trial site or investigator, disturbing the appropriate conduct of the trial.

The investigator / the trial site will be reimbursed for reasonable expenses incurred in case of trial termination (except in case of the third reason).

BI Trial No.: 1218.74

Dog No.: e01618200 10

Protocol Poy

## 4. TREATMENTS

#### 4.1 TREATMENTS TO BE ADMINISTERED

The study medication will be provided by Boehringer Ingelheim Pharma GmbH & Co. KG.

## 4.1.1 Identity of investigational product(s)

The characteristics of the test product are below.

Substance: Linagliptin (BI linagliptin)

Pharmaceutical form: tablet

Source: Boehringer Ingelheim Pharma GmbH & Co. KG

Unit Strength: 5 mg

Route of administration: p.o., once daily

Substance: Placebo matching linagliptin 5 mg

Pharmaceutical form: tablet

Source: Boehringer Ingelheim Pharma GmbH & Co. KG

Unit Strength: -

Route of administration: p.o., once daily

The characteristics of the reference product are below.

Substance: glimepiride 1 mg (Amaryl® 1 mg)

Pharmaceutical form: tablet (overencapsulated)

Source: Sanofi-Aventis

Unit Strength: 1 mg

Route of administration: p.o., once daily

Substance: glimepiride 2 mg (Amaryl® 2 mg)

Pharmaceutical form: tablet (overencapsulated)

Source: Sanofi-Aventis

Unit Strength: 2 mg

Route of administration: p.o., once daily

Substance: glimepiride 3 mg (Amaryl® 3 mg)

Pharmaceutical form: tablet (overencapsulated)

Source: Sanofi-Aventis

Unit Strength: 3 mg

Route of administration: p.o., once daily

Substance: glimepiride 4 mg (Amaryl® 4 mg)

Pharmaceutical form: tablet (overencapsulated)

Source: Sanofi-Aventis

Unit Strength: 4 mg

Route of administration: p.o., once daily

Boehringer Ingelheim 20 April 2016 BI Trial No.: 1218.74

Substance: Placebo matching glimepiride (Amaryl® 1-4 mg)

Pharmaceutical form: tablet (overencapsulated)

Source: Boehringer Ingelheim Pharma GmbH & Co. KG

Unit Strength: -

Route of administration: p.o., once daily

# 4.1.2 Method of assigning patients to treatment groups

Patients who meet the trial entry criteria at the end of the 2-4 weeks placebo run-in phase will be randomly assigned to linagliptin 5 mg or glimepiride in a balanced ratio (see Section 7.5). Patient assignment to the treatment groups will be determined by a computer generated random sequence using an interactive voice and web-based response system (IXRS). To facilitate the use of IXRS, each study site will receive an information manual describing the steps to randomise a patient, to obtain a medication kit assignment and to acknowledge receipt of study medication.

The assigned medication number will be entered in the eCRF, and the corresponding medication kit should be given to the patient. Using this procedure, the investigator will not know to which treatment group the next patient will belong.

#### 4.1.3 Selection of doses in the trial

The dose of 5 mg linagliptin was selected based on the results from previous dose finding studies (please refer to the actual version of the Investigator's Brochure [U04-1767]) and represents the marketed dose for linagliptin.

## 4.1.4 Drug assignment and administration of doses for each patient

Following the screening period and the placebo run-in period, patients who qualify will be randomised (Visit 2) to one of the dosage and treatment schedules outlined in Table 4.1.4: 1 below. Medication will be dispensed in a double-blind and double-dummy manner as either 5 mg linagliptin (plus glimepiride placebo) or an initial dose of 1 mg /day of glimepiride (plus linagliptin placebo). IXRS will allocate medication kit numbers at each scheduled in-clinic visit (V2 – 31). At visits 2-5 patients will receive one treatment box, sufficient for 4 weeks treatment (plus 1 week reserve). At visits 6-31 patients will receive one treatment box, sufficient for 16 weeks (plus two weeks reserve) of treatment.

After the starting dose of 1 mg/day, glimepiride/ glimepiride placebo has to be uptitrated in 4 week intervals during the first 16 weeks of treatment to the next dose to a potential maximum dose of 4 mg/day, if the fasted HBGM values are > 110 mg/dl (6.1 mmol/l) at the day of visit 3, 4 and 5 (in-clinic HBGM measurement at the day of the visit), unless the investigator considers that it would place the patient at an increased risk for hypoglycaemia. The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value.

Boehringer Ingelheim 20 April 2016 BI Trial No.: 1218.74

Patients on previous glimepiride may continue on their previous glimepiride dose up to Visit 2 (SU/glinide should not be taken in the morning of Visit 2). These patients will start the glimepiride/glimepiride placebo at their pre-trial glimepiride dose. If prior glimepiride dose was  $\geq 4$  mg/day, the patient will start the glimepiride/glimepiride placebo in the randomisation phase at a dose of 4 mg/day combined with 5 mg/day linagliptin/ linagliptin placebo. Patients on a previous SU, that is not glimepiride, or glinide should start glimepiride /glimepiride placebo at Visit 2 at a starting dose of 1 mg/day combined with 5 mg/day linagliptin/ linagliptin placebo.

The patients will be instructed to bring their HBGM devices to a visit for an additional measurement of fasted glucose during the titration phase, and if required, during maintenance phase (see flow chart).

HBGM measurements at visits during Titration Phase are mandatory to efficaciously uptitrate dosing of the glimepiride/glimepiride placebo.

Uptitration of glimepiride/glimepiride placebo may occur at (un)scheduled visits during the maintenance phase in case of deterioration of glucose control to the next dose to a potential maximum of 4 mg/day (glimepiride or placebo) combined with 5 mg/day linagliptin/ linagliptin placebo (with at least a dose interval of 4 weeks), provided fasted and confirmed HBGM values are > 110 mg/dl (6.1 mmol/L).

At any time during the study, the glimepiride/glimepiride placebo can be down titrated to prevent recurrent hypoglycaemic events.

Glimepiride/glimepiride placebo may be uptitrated again to the next dose (in case it was down titrated due to hypoglycaemia) to the potential maximum dose of 4 mg/day with 5 mg/day linagliptin/ linagliptin placebo.

Table 4.1.4: 1 Linagliptin and glimepiride oral administration per dose group and day

| Dose group | Tablet | Capsule<br>(overencapsulated<br>tablet) |
|---|---|---|
| (For run-in phase only) Placebo | Placebo tablet matching to linagliptin | Placebo capsule matching to glimepiride |
| (For treatment phase only) linagliptin 5 mg | 5 mg tablet | Placebo capsule matching to glimepiride |
| glimepiride<br>1 mg | Placebo matching to linagliptin 5 mg tablet | 1 mg capsule |
| glimepiride<br>2 mg | Placebo matching to linagliptin 5 mg tablet | 2 mg capsule |
| glimepiride<br>3 mg | Placebo matching to linagliptin 5 mg tablet | 3 mg capsule |
| glimepiride<br>4 mg | Placebo matching to linagliptin 5 mg tablet | 4 mg capsule |

If applicable, patients will continue with their standard metformin therapy (preferably  $\geq 1500$  mg daily) throughout the entire study with an unchanged dose unless medical emergencies or other plausible reasons (e.g. renal impairment, lactacidosis, heart failure, dose intolerance, hypoglycaemia or hyperglycaemia) necessitates changes (at the discretion of the investigator). In case of contrast exposure for investigation of coronary artery pathology or other vessel assessment, metformin is allowed to be discontinued according to local guidelines (see also Section 4.2.2.1). The above principle also applies for patients being included on a background of alphaglucosidase inhibitor.

During the maintenance phase it is investigator's judgement to change the glimepiride/glimepiride placebo and/or background medication dose. Rescue medication could also be initiated provided protocol criteria are met (see section 4.2.1)

Administration of the study medication is once daily. Patients should be instructed to take their trial medication once daily with 150 mL of water.

To ensure a dose interval of about 24 hours, the medication should be taken at the same time every day. If a dose is missed by more than 12 hours, that dose should be skipped and the next dose should be taken as scheduled. No double doses should be taken. Study medication should be taken shortly before or during a meal.

In some situations, it might be necessary to interrupt study medication temporarily. Patients are encouraged to re-start study treatment after an interruption if appropriate

Doc No.: c01618200-19

20 April 2016

Protocol Revision 6 

in the opinion of the investigator and if not contraindicated. In case the patient is reinstituted on study treatment, the preferred dosage for glimepiride/glimepiride placebo is the dose used before stopping treatment (unless hypoglycaemia was the reason to temporarily stop treatment). In case there is a need for further adjustments after this re-institution the guidance for treatment initiation should be followed.

Patients should be instructed not to take their trial medication in the morning of visit days as they will be dosed whilst in the clinic. Patients who fail to do so should have the visit rescheduled as soon as possible, ideally on the following day. Background and/or rescue medication will be taken as prescribed including visit days.

Patient visits should be routinely scheduled in the morning (preferably between 7:00 AM and 11:00 AM), at approximately the same time at each visit. The actual date/time of trial drug administration at the study visit will be recorded in the eCRF.

## 4.1.5 Blinding and procedures for unblinding

#### 4.1.5.1 Blinding

After randomisation at Visit 2, neither the patients nor the investigators or sponsor will be aware of the treatment allocation.

Patients assigned to one of the double-blind treatments will take 1 tablet and 1 capsule daily, either:

- One 5 mg tablet of linagliptin plus one inactive placebo capsule (overcapsulated tablet) matching glimepiride
- One 1 mg or 2 mg or 3 mg or 4 mg glimepiride capsule (overencapsulated tablet) plus one inactive placebo tablet matching linagliptin.

The placebo tablets and capsules will be identical in appearance to the respective active treatments.

At any time during the study, glimepiride/glimepiride placebo can be down titrated to prevent recurrent hypoglycaemic events. Glimepiride/glimepiride placebo dose adjustments can be done through IXRS in a blinded manner.

# 4.1.5.2 Procedures for emergency unblinding

In the event of a medical emergency which requires identification of an individual patient's treatment, investigators will be able to access this information via IXRS. The local Clinical Monitor or the Onsite Monitor/CRA should be contacted immediately (preferably before unblinding takes place) and the reason for unblinding the patient's treatment should be documented in the medical records. A patient could continue with study medication after unblinding.


**Protocol Revision 6** 

# 4.1.6 Packaging, labelling, and re-supply

Drug supplies will be provided by the Department of Pharmaceutical Development of Boehringer Ingelheim Pharma GmbH & Co. KG, Biberach, Germany. All study medication will be contained in medication boxes identified with the trial number and medication number. Each medication box will contain an appropriate amount of BI linagliptin tablets or glimepiride capsules, plus some reserve, for dosing until the next scheduled visit.

Trial drug will be supplied on a per visit basis. Supply will be managed by an IXRS.

Examples of the labels will be available in the Investigator's Site File (ISF)

# 4.1.7 Storage conditions

All trial medication should be stored at room temperature (not above 25 °C) in the original containers. Patients should be instructed not to remove the trial medication from the blisters/wallets until immediately prior to the time of intake to protect tablets from humidity and light. Patients will be reminded to keep the study drug out of the sight and reach of children.

A temperature log must be maintained at site. If the storage conditions are found to be outside the specified range, the CML, IXRS and the BI CTSU must be contacted immediately in order to clarify whether the trial medication can still be used.

#### 4.1.8 Drug accountability

Drug supplies, which will be provided by the sponsor and/or appointed CRO, must be kept in a secure, limited access storage area under the storage conditions defined by the sponsor. Throughout the trial, drug receipt, usage, and return must be documented by the site and verified by the CRA, any discrepancies in drug supplies will be noted and explained. All unused medication including blisters/wallets and patient boxes (empty or filled) must be returned to the sponsor.

The investigator, pharmacist and/or investigational drug storage manager will receive the investigational drugs delivered by the sponsor when all country specific required approvals are in place and all required country specific essential documents are in house e.g.:

- approval of the study protocol by the IRB / ethics committee.
- availability of a signed and dated clinical trial contract between the sponsor and the trial centre.
- approval/notification of the regulatory authority, e.g. competent authority,
- availability of the curriculum vitae of the principal investigator,
- availability of a signed and dated clinical trial protocol
- if applicable availability of the proof of a medical licence for the principal investigator
- for USA only: availability of the Form 1572

The investigator, pharmacist and/or investigational drug storage manager must maintain records of the product's delivery to the trial site, the inventory at the site, the use by each patient, and the return to the sponsor or alternative disposition of unused product(s).

These records will include dates, quantities, batch/serial numbers, expiry ('use by') dates, and the unique code numbers assigned to the investigational product(s) and trial patients. The investigator, pharmacist and/or investigational drug storage manager will maintain records that document adequately that the patients were provided the doses specified by the CTP and reconcile all investigational product(s) received from the sponsor. At the time of return to the sponsor and/or appointed CRO, the investigator, pharmacist and/or investigational drug storage manager must verify that all unused or partially used drug supplies have been returned by the clinical trial patient and that no remaining supplies are in the investigator's possession.

This text is only applicable to Japan:

The Investigator / pharmacist / investigational drug storage manager should return the unused and collected investigational drugs (including the empty containers) to the Sponsor after unblinding the trial.

In case investigational drugs are returned before unblinding of the trial, the Investigator / pharmacist / investigational drug storage manager should seal the opened container (excluding empty containers) for the patient, and before returning the unused and collected investigational drugs (including the empty boxes) to the Sponsor.

When returning the investigational drugs, the Investigator / pharmacist / investigational drug storage manager should exercise utmost caution to assure that the Sponsor and other relevant trial staff members remain blinded to the patient's name on the package (container or label) of the investigational drugs.

Upon completion of the trial, the Investigator / pharmacist / investigational drug storage manager will submit to the Sponsor a copy of the investigational drug dispensing and return log. When submitting the copy, the Investigator / pharmacist / investigational drug storage manager should exercise caution to assure that the Sponsor and other relevant trial staff members remain blind to the patient's name.

# 4.2 CONCOMITANT THERAPY, RESTRICTIONS, AND RESCUE TREATMENT

#### 4.2.1 Rescue medication, emergency procedures, and additional treatment(s)

The use of rescue medication will be permitted in this trial, and will be limited to pioglitazone, metformin, alpha-glucosidase inhibitor or basal insulin (i.e. intermediate or long-acting insulin such as insulin glargine, insulin determir, neutral protamine hagedorn [NPH] insulin) including during the FU period.

In specific situations (e.g. during hospitalisation) short-acting insulin may be given as rescue medication for up to two weeks in combination with the study medication.

The dose of rescue medication will be according to local labelling at the investigator's discretion. Rescue medication will not be provided as part of the clinical trial supplies, unless required by local laws and regulations. Particular rescue medication may not be available in countries (e.g. pioglitazone).

The use of rescue medication in case of hyperglycaemia will be permitted during the <u>randomised</u> treatment period of the trial only and only if one or more of the following criteria have met:

- During the <u>titration phase</u> (Visit 2 to Visit 6): The patient has a glucose level >240 mg/dl (>13.3 mmol/L) after an overnight fast.
- During the <u>maintenance phase</u> (Visit 6 to Final Visit): The patient has a glucose level >180 mg/dl (>10.0 mmol/L) after an overnight fast
- During the <u>maintenance phase</u> (Visit 6 to Final Visit): the patient has an HbA<sub>1c</sub> > 7.5% (58 mmol/mol)

The above results for fasting plasma glucose, which could be obtained from the HBGM device, should be confirmed, meaning that there is a minimum of two measurements, at least one of which should be performed after an overnight fast at the investigational site, and on a different day to the initial measurement.

In the case of repeated symptomatic hypoglycaemia or severe hypoglycaemia (criteria see Section <u>5.2.2.1.</u>); appropriate adjustment of oral antidiabetic therapy like dose reduction of metformin, alpha-glucosidase inhibitor, rescue therapy or study medication should be initiated.

The use of rescue medication has to be taken in accordance with the prescribing information and will be recorded in the eCRF. Patients who have to be treated with other rescue medication than the protocol defined rescue therapy should discontinue study treatment when the combined use of the study treatment and this rescue medication is contraindicated, but will remain in the trial.

Any additional treatment, that does not qualify as a rescue medication, and is considered necessary for the patient's welfare may be given at the discretion of the investigator. Exceptions to this are the restrictions described in Section 4.2.2.

All concomitant (additional) and/or rescue medication will be recorded on the appropriate pages of the eCRF.

There are no special emergency procedures to be followed.

#### 4.2.2 Restrictions

# 4.2.2.1 Restrictions regarding concomitant treatment

The use of other antidiabetic agents (next to background therapy and any rescue therapy) such as other oral agents, short-acting insulin\* or injectable GLP-1 analogue/agonists will be prohibited during the course of the study.

\*Short acting insulin may be given as rescue medication for up to two weeks (e.g. during hospitalisation).

Additionally treatment with anti-obesity drugs is prohibited.

In case metformin is used as background therapy and participants are in need for intravascular administration of iodine containing contrast agents: metformin is allowed to be discontinued according to local practice; usually before administration and 48 hours afterwards.

If any restricted treatments or any other concomitant drugs interfering with the study medication are given during the conduct of the trial, the study medication dose can be reduced, or the study medication can be discontinued temporarily, or if needed permanently (see also Section 3.3.4.1).

# 4.2.2.2 Restrictions on diet and life style

No restrictions given; all patients should be provided healthy lifestyle advice at baseline and also have this reinforced during the trial. Available educational material (e.g. from national diabetes associations or national health authorities) relevant for the country/region could be supplied by the site.

#### 4.3 TREATMENT COMPLIANCE

Patients will be asked to bring all trial medication (with or without any remaining tablets/capsules) with them to each trial Visit. The tablets/capsules will be counted by the investigator or his/her designate and compliance will be calculated. Compliance will be calculated according to the formula:

Compliance (%) =  $\frac{\text{Nr. of tablets/capsules actually taken since last tablet/capsule count}}{\text{Nr. of tablets/caps. which should have been taken in the same period}} \times 100\%$ 

Compliance during the open-label placebo run-in phase should be between 80% and 120%. If compliance is outside this range, the patient should be carefully interviewed and, if necessary, re-informed about the purpose and the conduct of the trial. Investigator may extend the placebo-run phase up to four weeks to meet this compliance requirement. Unreliable patients should be withdrawn from the study before randomisation at the discretion of the investigator.

Compliance during the randomised treatment phase should also be between 80% and 120%. Severe violation of treatment compliance is defined as an important protocol violation and will lead to the exclusion from the per protocol set (PPS).

Boehringer Ingelheim
BI Trial No.: 1218.74
20 April 2016

Patients who are not compliant with their medication should again be carefully interviewed and again re-informed about the purpose and the conduct of the trial.

# 5. VARIABLES AND THEIR ASSESSMENT

#### 5.1 EFFICACY

# 5.1.1 Endpoint(s) of efficacy

The primary endpoint in this trial is time to the first occurrence of any of the following adjudicated components of the primary composite endpoint: CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI) or non-fatal stroke

The key secondary efficacy endpoints are:

- time to the first occurrence of any of the following adjudicated components of CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI), non-fatal stroke or hospitalisation for unstable angina pectoris
- composite endpoint of (treatment sustainability defined as the proportion of patients that are on study treatment at study end, that at Final Visit maintain glycaemic control (HbA<sub>1c</sub>  $\leq$  7.0%) without need for rescue medication (between end of titration [Visit 6] and Final Visit) and patients without any moderate/severe hypoglycaemic episodes (between Visit 6 and Final Visit) and without  $\geq$  2% weight gain at Final Visit (between Visit 6 and Final Visit))
- composite endpoint of (treatment sustainability defined as the proportion of patients that are on study treatment at study end, that at Final Visit maintain glycaemic control (HbA $_{1c} \le 7.0\%$ ) without need for rescue medication (between Visit 6 and Final Visit) and patients without > 2% weight gain at Final Visit (between Visit 6 and Final Visit))

Whereas moderate/severe hypoglycaemic episodes are defined as:

- Moderate hypoglycaemic event: documented symptomatic hypoglycaemia with plasma glucose concentration ≤ 70 mg/dL. Event accompanied by typical symptoms of hypoglycaemia but no need for external assistance
- Severe hypoglycaemic event: documented hypoglycaemic episode requiring assistance of another person to actively administer carbohydrate, glucagon or other resuscitative actions need for external assistance

Additionally secondary efficacy endpoints are the change from baseline of HbA<sub>1c</sub>, FPG, proportion of patients that at Final Visit maintain glycaemic control without need for rescue medication (between end of titration [Visit 6] and Final Visit) to obtain HbA<sub>1c</sub>  $\leq$  7.0% or that obtain HbA<sub>1c</sub>  $\leq$  7.0% overall (see Section 7.1).

## 5.1.2 Assessment of efficacy

 $HbA_{1c}$ :

Blood samples for the determination of  $HbA_{1c}$  will be taken according to the <u>Flow Chart</u>. The blood sample can be taken at any time during the visit. The samples will be analysed at a central laboratory or its affiliates having a National Glycohemoglobin

20 April 2016

Standardization Program (NGSP) Level I certificate. Further details about sample handling, shipment, and assay procedures can be found in the Investigator's Site File (Lab manual).

*FPG*:

Blood samples for the determination of FPG will be taken according to the <u>Flow Chart</u> after an overnight fast (10 hours no food and only water). At all respective visits, the samples should be taken before breakfast <u>and</u> before trial drug administration. The samples will be measured at a central laboratory using validated assays. Further details about sample handling and shipment can be found in the Investigator Site File (Lab manual).

#### 5.2 SAFETY

# 5.2.1 Endpoint(s) of safety

Secondary and tertiary CV endpoints are described in <u>Section 7</u>.

In addition, incidence and intensity of adverse events, physical examination, vital signs, ECG and change from baseline in laboratory parameters will be assessed.

#### 5.2.1.1 Reporting waiver for cardiovascular outcome events

In accordance with ICH-guideline E2A and in order to maintain the integrity of this study, cardiovascular outcome events that occur after randomisation and represent a SAE, are exempted from expedited reporting to health authorities. The medication code will not be broken for the purpose of expedited reporting to regulatory authorities.

Cardiovascular outcome events are defined as the following components of the primary, secondary and tertiary cardiovascular endpoints:

- cardiovascular death
- non fatal myocardial infarction
- silent myocardial infarction
- non fatal stroke (ischemic/hemorrhagic/etiology unknown)
- hospitalisation for unstable angina
- heart failure requiring hospitalisation
- transient ischemic attack (TIA)
- coronary revascularisation procedures (PCI and CABG)

For definitions of the cardiovascular outcome events see Appendix 10.2.

The investigator must document immediately (within 24 hours or the next business day whichever is shorter) the outcome events on the appropriate eCRF page in the RDC.

In case of a stroke the disability or dependence in the daily activities will be collected with the grade of modified Rankin Scale (mRS) at day 7 or at hospital discharge (if duration of hospitalization is < 7 days) and 3-6 months after stroke onset.

#### 5.2.2 Assessment of adverse events

#### 5.2.2.1 Definitions of adverse events

#### Adverse event

An adverse event (AE) is defined as any untoward medical occurrence, including an exacerbation of a pre-existing condition, in a patient in a clinical investigation who received a pharmaceutical product. The event does not necessarily have to have a causal relationship with this treatment.

An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

#### Serious adverse event

A serious adverse event (SAE) is defined as any AE which results in death, is immediately life-threatening, results in persistent or significant disability / incapacity, requires or prolongs patient hospitalisation, is a congenital anomaly / birth defect, or is to be deemed serious for any other reason if it is an important medical event when based upon appropriate medical judgement which may jeopardise the patient and may require medical or surgical intervention to prevent one of the other outcomes listed in the above definitions.

Life-threatening in this context refers to an event in which the patient was at risk of death at the time of the event; it does not refer to an event that hypothetically might have caused death if more severe.

For Japan: An AE which possibly leads to disability will be reported as an SAE. Every new occurrence of cancer will be reported as a SAE regardless of the duration between discontinuation of the drug and the occurrence of the cancer.

#### Intensity of adverse event

The intensity of the AE should be judged based on the following:

Mild: Awareness of sign(s) or symptom(s) which is/are easily tolerated Moderate: Enough discomfort to cause interference with usual activity Severe: Incapacitating or causing inability to work or to perform usual activities

#### Causal relationship of adverse event

Medical judgment should be used to determine the relationship, considering all relevant factors, including pattern of reaction, temporal relationship, de-challenge or re-challenge, confounding factors such as concomitant medication, concomitant diseases and relevant history. Assessment of causal relationship should be recorded in the case report forms.

**Protocol Revision 6** 


For Japan: The reason for the decision on causal relationship needs to be provided in the CRF.

Yes: There is a reasonable causal relationship between the investigational product administered and the AE.

No: There is no reasonable causal relationship between the investigational product administered and the AE.

If a SAE is reported from a still blinded trial, the causal relationship must be provided by the investigator for all potential trial drugs, i.e. the BI trial drug linagliptin, active comparator glimepiride and placebo.

## Worsening of underlying disease or other pre-existing conditions

Worsening of the underlying disease or of other pre-existing conditions will be recorded as an (S)AE in the (e)CRF.

# Changes in vital signs, ECG, physical examination, and laboratory test results

Changes in vital signs including blood pressure, pulse rate, ECG\*, physical examination, and laboratory tests results will be recorded as (S)AEs in the eCRF if they are judged clinically relevant by the investigator.

\* Changes in the ECG indicating silent MI should be reported as cardiovascular outcome event (see also Section 10.5).

Clinically relevant abnormalities found at physical examination, vital signs or ECG that are not pre-existing prior to signing of informed consent (study inclusion) should be reported as adverse events, If such abnormalities already pre-exist prior study inclusion they should be considered as baseline conditions.

# Hypoglycaemic events

Hypoglycaemic events should be documented according to the following criteria:

- Asymptomatic hypoglycaemia: Event not accompanied by typical symptoms of hypoglycaemia but with a measured plasma glucose concentration ≤ 70 mg/dl (3.9 mmol/l)
- Documented symptomatic hypoglycaemia with glucose concentration  $\geq 54$  mg/dl and  $\leq 70$  mg/dl ( $\geq 3.0$  mmol/l and  $\leq 3.9$  mmol/l): Event accompanied by typical symptoms of hypoglycaemia
- Documented symptomatic hypoglycaemia with glucose concentration < 54 mg/dl (< 3.0 mmol/l): Event accompanied by typical symptoms of hypoglycaemia but no need for external assistance
- Severe hypoglycaemic episode: Event requiring the assistance of another person to actively administer carbohydrate, glucagon or other resuscitative actions

All symptomatic hypoglycaemic events, all asymptomatic events with glucose levels less than 3.0 mmol/L (or less than 54 mg/dL) and all asymptomatic hypoglycaemic

events that are considered as adverse events by the investigator have to be recorded as an adverse event.

#### Adverse Events of Special Interest (AESI)

The term AESI relates to any specific AE that has been identified at the project level as being of particular concern for prospective safety monitoring and safety assessment within this trial, e.g. the potential for AEs based on knowledge from other compounds in the same class. AESI need to be reported to the Sponsor's Pharmacovigilance Department within the same timeframe that applies to SAE.

The following events are considered as adverse events of special interest (AESI):

- Hypersensitivity reactions such as angioedema, angioedema-like events, and anaphylaxis
- Skin lesions such as exfoliative rash, skin necrosis, or bullous dermatitis
- Hepatic events such as  $\geq 3$  fold ULN of AST and/or ALT in combination with an elevation of total bilirubin  $\geq 2$  fold ULN measured in the same blood draw sample, hepatitis, hepatic injury, jaundice and potential Hy's Law cases.
- Renal adverse events such as acute renal failure,
- Pancreatitis (refer to ISF)
- Pancreatic cancer

Hepatic injury is defined by the following alterations of liver parameters: for patients with normal liver function at baseline: an elevation of AST and/or  $ALT \geq 3$  fold ULN combined with an elevation of total bilirubin  $\geq 2$  fold ULN measured in the same blood draw sample. Patients showing these lab abnormalities need to be followed up according to Section 10.6 of this clinical trial protocol and the "DILI checklist" provided in ISF.

#### Hepatic events:

If AST and/or ALT are increased  $\geq 3$  x ULN, follow-up laboratory tests of ALT, AST, total bilirubin (with differentiation of bilirubin in direct and indirect if total bilirubin is elevated) and additionally alkaline phosphates (ALP), CK (CK-MB if CK is elevated), amylase, lipase and INR must be initiated as soon as possible (ideally within 48 to 72 hours of the pathologic test result). Further follow-up investigations shall be initiated depending on the clinical course until the patient is recovered and/or a diagnosis was made. See for further details Section 10.6.2.

Laboratory Criteria for "Potential Hy's Law case":

- 1. AST and/or ALT > 3 x ULN and
- 2. Total bilirubin  $> 2 \times ULN$  and
- $3. ALP < 2 \times ULN$

#### Renal events:

If creatinine shows a  $\geq$  2-fold increase from baseline, the investigator should make arrangements for follow-up blood samples(s) to be collected for repeat analysis of creatinine.

Further follow-up investigations should be done according to medical judgement depending on the clinical course until the patient is recovered and/or a diagnosis is made.

#### Skin lesions:

If skin lesions (such as exfoliative rash, skin necrosis, or bullous dermatitis - see further detailed list in ISF): further follow-up investigations should be done according to medical judgement depending on the clinical course until the patient is recovered and/or a diagnosis is made.

Protocol-specified AESIs (as identified by the investigator based on the above definitions for adverse events of special interest) can be classified as serious or non-serious but all these AESIs once identified by the investigator must be reported on an SAE form in an expedited manner similar to SAEs, even if they do not meet any of the SAE seriousness criteria.

Beyond of this, and for the purposes of ongoing pharmacovigilance activities by the sponsor, adverse events based on additional searches for coded preferred terms of adverse events captured in the trial database (such as Special MedDRA Queries (SMQs), and user defined searches (BicMQs)) will be queried to verify with the investigator if the adverse event reported represent such a suspected or diagnosed protocol specific AESI. AESIs once identified by the investigator must be reported on a SAE form in an expedited manner similar to SAEs, even if they do not meet any of the SAE seriousness criteria.

These additional searches (summarised under the so called 'overview of protocol defined AESIs and safety topics of interest') may change according to active pharmacovigilance of linagliptin. The most up to date list of these searches will be included in the ISF/Remote Data Capture (RDC) system and changes will be communicated to all investigators.

# 5.2.2.2 Adverse event and serious adverse event reporting

Reporting will be done according to the specific definitions and instructions detailed in the 'Adverse Event Reporting' section of the Investigator Site File (ISF).

All adverse events, serious and non-serious and all AESIs, occurring during the course of the clinical trial (i.e., from signing the informed consent onwards through the residual effect period (REP) until the individual patient's end of trial) will be collected, documented and reported to the sponsor by the investigator on the appropriate eCRFs pages.

The REP (timeframe after last dose of study medication when measurable drug levels or pharmacodynamic effects are still likely to be present) is defined as 7 days after the last trial medication application. All AEs which occurred through the treatment phase and throughout the REP will be considered as on treatment please see <a href="section 7.3.3">section 7.3.3</a>. Events which occurred after the REP will be considered as post treatment events.

After the individual patient's end of trial the investigator does not need to actively monitor the patient for AEs but should only report relevant SAEs and relevant AESIs of which the investigator may become aware of.

However, if in an individual patient only vital status information is collected after premature discontinuation, from then on and until the individual patient's end of trial, the investigator does not need to actively monitor the patient for AEs but should only report fatal AEs, relevant SAEs and relevant AESIs of which the investigator may become aware of.

#### Immediate documentation of events:

The investigator must report immediately (within 24 hours of awareness the following events on the SAE form to the sponsor's unique entry point as specified in the ISF:

- All SAEs
- All serious and non-serious AESIs
- Non-serious AEs relevant for a reported SAE(s) and/or AESI(s)
- Potential Hy's Law cases (see Section 5.2.2.1)
- Cardiovascular outcome events if they represent a SAE and occur during the screening/run-in phase

The same timeline applies if follow-up information becomes available. In specific occasions the Investigator could inform the Sponsor upfront via telephone. This does not replace the requirement to complete and fax the BI SAE form.

# AEs considered "Always Serious"

In accordance with the European Medicines Agency initiative on Important Medical Events, Boehringer Ingelheim has set up a list of AEs, which by their nature, can always be considered to be "serious" even though they may not have met the criteria of an SAE as given above.

BI has established a list of AEs which are defined to be always serious. In order to support the investigator with the identification of these "always serious adverse events", if a non-serious AE is identified to be serious per BI definition, a query will be raised. The investigator must verify the description and seriousness of the event. If the event description is correct, the item "serious" needs to be ticked and a SAE has to be reported in expedited fashion following the same procedure as above.

The list of these adverse events can be found via the RDC-system.

For Japan: This information must be also reported immediately to the head of the trial site.

# Information required

For each AE, the Investigator should provide the information requested on the appropriate (e)CRF pages and the BI SAE form, e.g. onset, end date, intensity, treatment required, outcome, seriousness, and action taken with the investigational drug(s). The Investigator should determine the causal relationship to the trial medication, and any possible interactions between the investigational drug(s) and a Non-Investigational Medicinal Product (NIMP).

All (S)AEs, including those persisting after individual patient's end of trial must be followed up until they have resolved, have been sufficiently characterized, or no further information can be obtained.

This immediate report is required irrespective of whether the investigational product has been administered or not and irrespective of causal relationship. It also applies if new information to existing SAEs or protocol-specified AESIs becomes available.

#### **Pregnancy**

In rare cases, pregnancy might occur in clinical trials. Once a female subject has been enrolled into the clinical trial, after having taken study medication, the investigator must report immediately any drug exposure during pregnancy to the sponsor. Drug exposure during pregnancy has to be reported immediately (within 24 hours of awareness to the defined unique entry point for SAE forms of the respective BI OPU (country-specific contact details will be provided in the Investigator Site File). The outcome of the pregnancy associated with the drug exposure during pregnancy must be followed up. In the absence of an (S)AE, only the Pregnancy Monitoring Form for Clinical Trials and not the SAE form is to be completed. The ISF will contain the Pregnancy Monitoring Form for Clinical Trials (Part A and Part B).

# 5.2.2.3 Oncological adverse events

Epidemiological evidence suggests that people with diabetes are at a significantly higher risk of several forms of cancer compared with subjects without diabetes [R10-6495]. Currently it is unclear whether the association between cancer and diabetes is indirect and largely due to shared risk factors (such as the modifiable risk factors: e.g. obesity, diet, physical activity, tobacco smoking, alcohol, or non-modifiable risk factors: e.g. age, gender, race, and ethnicity), whether it is direct influence (e.g. due to hyperglycaemia), or whether diabetes is a marker of underlying biologic factors that alter cancer risk (e.g. insulin resistance and hyperinsulinemia) [R10-6496, R10-6498, R10-6536, R10-6497, R10-6494].

In order to assess patients with oncological adverse events (benign and malignant) in detail, detailed information will be requested and should be provided. The main focus on oncological adverse events is on the following organ systems, based on [R10-6638] where an increased risk for cancer in the population of patients with T2DM was described:

- Liver
- Pancreas
- Endometrium

- Colon and rectum
- Breast
- Bladder
- Thyroid
- Prostate

Request for detailed information (e.g. medical history, diagnostic result, laboratory results staging, genetics), will be mainly focused on the above listed organ systems, however is not restricted to them. For details refer to the oncology assessment charter.

# 5.2.3 Assessment of safety laboratory parameters

The parameters that will be determined are listed below. Analysis will be performed by a central laboratory:

## 5.2.3.1 Haematology

- Haematocrit
- Haemoglobin
- Erythrocyte count
- Platelet count

# 5.2.3.2 Clinical chemistry

- Amylase
- Lipase
- AST\*\* (aspartate transaminase, SGOT)
- ALT\*\* (alanine transaminase, SGPT)
- γ-GT (gamma-glutamyl-transferase)
- Alkaline phosphatase
- Lactic dehydrogenase (LDH)
- Total bilirubin\*\*
- Direct and indirect bilirubin if total bilirubin is elevated
- Total Protein
- Albumin
- Creatine kinase (CK)
- CK-MB, if CK is elevated

- Total and automates differential leukocyte counts (Neutrophils, Eosinophils, Basophils, Lymphocytes, Monocytes) in absolute counts
- Potassium
- Sodium
- Creatinine
- Urea
- Calcium
- Inorganic phosphorous
- Urid acid
- Cholesterol (total)\*\*\*
- HDL cholesterol\*\*\*
- LDL cholesterol\*\*\*
- Triglycerides\*\*\*
- Troponin

<sup>\*\*</sup>AST, ALT and Total bilirubin are combined in any lab assessment, with exception of Visit 1a.

\*\*\* Lipid profile, only obtained at Visits 2, 6, 9, 12, 15, 18, 21, 24, 27, and 30 and 32.

# 5.2.3.3 Urinalysis

- Albumin, Creatinine (spot urine quantitative measurement)
- Ketone
- Leucocytes

• Protein

Visit 1a safety laboratory only includes ALT (SGPT), AST (SGOT), alkaline phosphatase, serum creatinine, urine analysis and urine albumin and creatinine, in addition to HbA1c and does not need to be collected in fasted state.

Exact date and time of blood sampling should be recorded on the central laboratory requisition form.

Albumin/creatinine ratio will be calculated at the central lab.

Pregnancy testing (urine dipstick method) will be performed in female patients of child-bearing potential according to the <u>Flow Chart</u>. Testing will be performed locally, using pregnancy test kits provided by the central laboratory.

Immediately after the result of a pregnancy test is known, the pregnancy test kit will be discarded at the site. The result of the test <u>must</u> therefore be documented in the source documents available at site for future verification by the on-site monitor.

A negative pregnancy test result is required at Visit 2 for all female patients of childbearing potential to remain eligible for entry into the treatment phase of the trial.

#### 5.2.3.4 Renal function impairment

Renal function impairment will be assessed by the central lab based on the plasma creatinine value measured according to the Flow Chart.

Estimated Creatinine clearance will be calculated from serum creatinine using the following MDRD formula as specified in the Statistical Analysis Plan.

This formula considers the race as an adjustment factor, therefore, the race must be known (and will be collected) for accurate estimation.

Renal impairment will be classified in the following way:

- No renal function impairment: eGFR ≥ 90 mL/min/1.73m<sup>2</sup>;
- Mild renal function impairment: eGFR 60-89 mL/min/1.73m<sup>2</sup>;
- Moderate renal function impairment: eGFR 30-59 mL/min/1.73m<sup>2</sup>;
- Severe renal function impairment: eGFR 15-29 mL/min/1.73m<sup>2</sup>;
- Kidney failure: eGFR < 15 mL/min/1.73m<sup>2</sup>.


**Protocol Revision 6** 

## 5.2.4 Electrocardiogram (ECG)

12-lead ECGs (I, II, III, aVR, aVL, aVF, V1 - V6) will be recorded according to the Flow Chart.

The ECGs will be centrally analysed and stored by third party. Investigators will receive evaluated ECGs within 3 working days by third party, unless there are unresolved discrepancies. Additional ECGs may be collected by the investigator for safety reasons. Clinically relevant abnormal findings will be reported as AEs, if they are newly discovered after inclusion in the trial.

The recordings will be checked for pathological results by the investigator. Any ECG abnormalities will be carefully monitored and, if necessary, the patient will be removed from the trial and medically treated.

# 5.2.5 Assessment of other safety parameters

Vital signs and height

Systolic and diastolic blood pressure as well as pulse rate (electronically or by palpation, count for 1 minute) will be measured after 5 minutes of rest in the seated position according to the <u>Flow Chart</u>. All recordings should be made using a similar type of blood pressure recording instrument (i.e., approved sphygmomanometer or an approved blood pressure meter utilizing liquid mercury) on the same arm. See for further details <u>Section 10.3</u>.

Height (metres, m) will be measured according to the <u>Flow Chart</u>. Body mass index (BMI kg/m<sup>2</sup>) will be calculated for determination of eligibility at Visit 1a.

Weight and Waist circumference

Weight measurements (kilogram, kg) should always be done using a similar approved type of scale for one patient. In order to get comparable body weight values, it should be performed in the following way:

- fasting (except for the screening visit),
- after the urine sampling (weight after bladder voiding),
- shoes and coat/jackets should be taken off
- pockets should be emptied of heavy objects (i.e. keys, coins etc.).

Waist circumference measurements should be made around a patient's bare midriff, after the patient exhales while standing without shoes and with both feet touching and arms hanging freely. The measuring tape should be made of a material that is not easily stretched, such as fibreglass. The tape should be placed perpendicular to the long axis of the body and horizontal to the floor and applied with sufficient tension to conform to the measurement surface [R07-4080].

Waist circumference should be determined by measuring the midpoint between the lowest rib and the iliac crest [ $\underline{R07-4080}$ ].


#### Physical examination

A complete physical examination will be performed by the investigator according to <u>Flow Chart</u>. Documentation of, and findings from the physical examination, must be part of the source documents available at the site.

#### Home Blood Glucose Monitoring

All patients will be provided with Home Blood Glucose Monitoring (HBGM) equipment and supplies for use at home during the 2 up to 4 week run-in phase. HBGM testing should be performed at least once a week after an overnight fast during the placebo run-in phase of the trial and when patient experiences signs/symptoms of hypo- or hyperglycaemia. Once the patient is randomised, weekly testing is no longer required for study purposes and may be discontinued, however the patients will be instructed to bring their HBGM devices to a visit for an additional measurement of fasted glucose if required (see flow chart). HBGM measurements at visits during the titration phase are mandatory to efficaciously uptitrate dosing of the glimepiride/glimepiride placebo arm.

More frequent testing can be done if deemed necessary by the investigator or required by local authorities. The respective procedure for illiterate patients (if included) is described in the Appendix 10.1.1.

Instruction on the proper use of the HBGM will be provided by the study staff. The patient will be asked to record the results of the HBGM test on a HBGM Testing Log that will be included in the patient's source document file. Only in the case of linked adverse events or of asymptomatic hypoglycaemia with a measured plasma glucose concentration >=3.0 and <=3.9mmol/L (>=54 and <=70 mg/dL), if not considered as adverse event, the single HBGM values will be recorded in the CRF.

If the results of a HBGM test reveal blood plasma glucose value of > 240 mg/dL (>13.3 mmol/L) after an overnight fast during the titration phase or > 180 mg/dL (>10.0 mmol/L) after an overnight fast during the maintenance phase or > 400 mg/dl (22.2 mmol/L) randomly determined and confirmed by a second HBGM (not on the same day) the patient should contact the site for further advice.

During the trial, the patient should also contact the site for advice if the results of a HBGM test reveal blood plasma glucose value of  $< 70 \ (3.9 \ \text{mmol/L})$  after an overnight fast. If the blood glucose level is  $< 54 \ \text{mg/dL}$  (3.0 mmol/L), the patient should be instructed to eat/drink something containing carbohydrate.

HBGM (i.e. fasting glucose) will be measured in the morning of the visit prior the cognitive function testing (see <u>Flow Chart</u>).

The HBGM diary should be brought to each visit for review by investigator/trial staff. Patient HBGM diary should be collected at the visit (if completed) and a new HBGM diary should be given to the patient.

Boehringer Ingelheim
BI Trial No.: 1218.74
20 April 2016

 **Protocol Revision 6** 

20 April 2016 

# 5.4 APPROPRIATENESS OF MEASUREMENTS

All measurements performed during this trial are standard measurements and will be performed in order to monitor efficacy and safety aspects in an appropriate way.

The scheduled measurements are appropriate to see drug induced changes in vital signs, standard laboratory values,

and ECG. The endpoints are standard and accepted for evaluation of efficacy and safety of an oral antidiabetic drug, and they are widely used in this kind of study.

Therefore, the appropriateness of all measurements applied in this trial is given.

Boehringer Ingelheim
BI Trial No.: 1218.74
20 April 2016

# 6. INVESTIGATIONAL PLAN

#### 6.1 VISIT SCHEDULE

All trial visits should take place preferably between 7:00 AM and 11:00 AM. If a patient mistakenly takes trial medication on the morning of a visit before attending the clinic (excluding visits starting before randomisation) or comes in non-fasted where a fasting condition is required (all visits except Visit 1a), the visit should be rescheduled for another day as soon as possible reminding the patient about the expected conditions. The rescheduled visit must take place in a short enough time-frame so that the patient has sufficient trial medication available.

All patients are to adhere to the visit schedule as specified in the <u>Flow Chart</u>. Some flexibility is allowed in scheduling the visits according to visit time windows as specified in the <u>Flow Chart</u>. If any visit has to be rescheduled, subsequent visits should follow the original visit date schedule (calculated from randomisation Visit 2). The trial medication packs contain sufficient medication to allow for these time windows.

#### 6.2 DETAILS OF TRIAL PROCEDURES AT SELECTED VISITS

The <u>Flow Chart</u> summarizes the investigational procedures to be done at each visit. The procedures are further described below.

#### 6.2.1 Screening and Placebo run-in period

After informed consent process is complete and written informed consent is obtained, the patients will be assessed for study eligibility (Visit 1a) including central laboratory assessments: ALT (SGPT), AST (SGOT), alkaline phosphatase, serum creatinine, urinalysis and urine albumin and creatinine, in addition to HbA<sub>1c</sub>. Visit 1b should occur within one week after Visit 1a once it has been confirmed that the patient is eligible to continue to Visit 1b.

Those patients who qualify at screening (as determined at Visit 1a and Visit 1b), will undergo a 2 up to 4 week placebo run-in phase (Visit 1b to Visit 2). During the run-in phase the patients will continue receiving their background therapy and they will be given a Home Blood Glucose Monitor and all the necessary supplies to use it. The HBGM will be used according to Section <u>5.2.5</u>. Patients requiring rescue therapy during the screening and/or placebo run-in phase will not be eligible.

Patients must satisfy all inclusion and exclusion criteria prior to randomisation (see Sections 3.3.2 and 3.3.3). In addition, if during the run-in phase there is any indication that the patient is not stable enough, in terms of their type 2 diabetes, to complete the study or that the patient will be non-compliant with the study medication or restrictions, then these patients should not be randomised. The placebo-run phase could be extended up to 4 weeks to satisfy patients' successful completion of run-in phase.

20 April 2016

#### **6.2.2** Treatment phase

Randomisation will occur at Visit 2 using IXRS.

The patients will return to the clinic for regularly scheduled visits as specified in the <u>Flow Chart</u>. These visits will assess the occurrence of safety and efficacy endpoints, study medication compliance and accountability, concomitant therapy or intervention. Between Visit 2 and Visit 6 glimepiride/glimepiride placebo will be uptitrated up to maximal 4 mg/day (refer to section 4.1.4).

At each visit trial medication compliance will be calculated and new supplies from a new medication kit assigned via IXRS will be dispensed.

This is an outcome study. All patients, including those who discontinue treatment must be followed up until the end of the study. Patients who prematurely discontinue treatment will continue to be contacted by the investigator at regular intervals (according to the original visit schedule or an alternative reduced schedule negotiated with the patient). If a patient who prematurely discontinued study drug is not willing to return at the pre-defined regular visit schedule, at minimum a yearly telephone call (preferably every 6 months) and a telephone call at study end (through the patient or alternative person designated by the patient) will be required, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit should be recorded. Every attempt will be made by the investigator to ensure patients continue participating in the study during study drug interruptions and after discontinuation of study drug.

Patients who prematurely discontinued study medication during the Maintenance Phase are allowed to restart the study medication at any time. Every attempt should be made by the investigator to have the patient restart study medication, even if the dose must be down titrated.

## 6.2.3 End of trial and Follow-up period

A patient has the right to withdraw informed consent for participation at any time for any reason. However, withdrawal of consent from study participation should be very rare and unusual. Because of this, the investigator must be involved in the discussions with the patient regarding a withdrawal of consent.

If the patient withdrew informed consent the patient should stop taking study medication and should be asked to complete the study ending tests and procedures as described in the <u>Flow Chart</u> for End of Treatment Visit and Visit 33 (Follow up visit). Completing these procedures is strongly recommended for the patient's safety.

For patients that have withdrawn informed consent, the patient will be asked to resign an informed consent form, which will allow to enquire at least about the patient's vital status and occurred outcome events through contacts to relatives, acquaintances, family physicians, hospital records, etc.

Boehringer Ingelheim 20 April 2016 BI Trial No.: 1218.74

End of Treatment Visit (EOT) activities will be performed when a patient discontinues study medication treatment permanently. A follow-up visit will take place 30 days after the EOT visit.

The follow-up visit may be performed as a phone visit for patients who completed the planned treatment period (only adverse events/outcome events and changes in concomitant therapy, details on trial completion and vital status to be obtained).


**Protocol Revision 6** 

# 7. STATISTICAL METHODS AND DETERMINATION OF SAMPLE SIZE

#### 7.1 STATISTICAL DESIGN - MODEL

#### **Design**

This is a multicentre, multinational, randomised, double blind, parallel group, comparator-controlled safety study of linagliptin versus glimepiride. The trial is event driven and will run with an estimated number of 6000 patients for approximately 432 weeks beginning with the randomisation of the first patient. In the case the numbers of events is not or may not be reached within this period the trial duration and/or the number of patients enrolled will be increased until the defined number of adjudicated primary events is reached. We plan a 2 to 4 weeks run-in phase.

## **Objectives**

The study objectives are described in Section 2.2.

For the primary objective the upper bound of the two-sided (1-2\*alpha)\*100% confidence interval which equals the upper bound of the one-sided (1-alpha)\*100% confidence interval will be used to investigate non- inferiority of linagliptin versus glimepiride regarding the primary endpoint. The non-inferiority margin is chosen as 1.3 (FDA Guidance for Industry - Diabetes Mellitus - Evaluating Cardiovascular Risk in New Antidiabetic Therapies to Treat Type 2 Diabetes, R09-2151). The overall significance level is 2.5%. The alpha for each analysis depends on the alpha-spending function and the schedule of interim analyses.

#### Primary endpoint

The primary endpoint used in the primary analysis is time to the first occurrence of any of the following adjudicated components of the primary composite endpoint: CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI) or non-fatal stroke.

If patients do not experience a primary endpoint event, they will be considered censored at their last documented study visit. If a patient died and has no primary outcome event, the patient will be censored at the date of death.

# Key Secondary endpoints

As key secondary endpoints will be analysed:

 time to the first occurrence of any of the following adjudicated components of the composite endpoint: CV death (including fatal stroke and fatal MI), nonfatal MI (excluding silent MI), non-fatal stroke or hospitalisation for unstable angina pectoris.

2) composite endpoint of (treatment sustainability defined as the proportion of patients that are on study treatment at study end, that at Final Visit maintain glycaemic control (HbA1c ≤ 7.0%) without need for rescue medication\* (between end of titration [Visit 6] and Final Visit) and patients without any moderate/severe hypoglycaemic episodes (between Visit 6 and Final Visit) and without > 2% weight gain at Final Visit (between Visit 6 and Final Visit)).

- 3) composite endpoint of (treatment sustainability defined as the proportion of patients that are on study treatment at study end, that at Final Visit maintain glycaemic control (HbA1c  $\leq$  7.0%) without need for rescue medication\* (between Visit 6 and Final Visit) and patients without  $\geq$  2% weight gain at Final Visit (between Visit 6 and Final Visit))
- \* Any dose increase of anti-diabetic background medication or introduction of new anti-diabetic treatment <u>during</u> study medication treatment will be counted as rescue medication. Short term use of any insulin- up to two weeks (e.g. during hospitalisation) won't count as rescue medication in the definition of treatment sustainability.

# Secondary cardiovascular endpoints

In additional analyses the occurrence of the primary and first key secondary endpoint will be evaluated, resulting in the number of patients with at least one of the events above and the relative frequency with respect to the number of patients in the full analysis set (FAS).

Further secondary CV-endpoints are the occurrence of and time to:

• Composite endpoint of all CEC confirmed adjudicated events (see tertiary cardiovascular endpoints)

# Secondary diabetes related endpoints

Secondary <u>diabetes related</u> endpoints include change from baseline to Final Visit in the following laboratory parameters:

- HbA<sub>1c</sub>
- fasting plasma glucose
- Total cholesterol
- LDL cholesterol
- HDL cholesterol
- Triglycerides
- Creatinine
- eGFR (MDRD formula)
- Urinary albumin

In addition any transition in albuminuria classes will be investigated.
Boehringer Ingelheim
BI Trial No.: 1218.74
20 April 2016

### 7.2 NULL AND ALTERNATIVE HYPOTHESES

For the primary objective, <u>first</u> a non-inferiority hypothesis is tested with respect to time to first occurrence of any of the adjudicated components of the primary composite endpoint.

 $H_{0(NonInf)}$ :  $HR_{linagliptin \ vs. \ glimepiride} \ge \delta$ 

 $(H_{0(NonInf)})$ : Linagliptin is inferior to glimepiride by at least  $\delta$  regarding the risk of the primary composite endpoint of cardiovascular events.)

VS.

 $H_{1(NonInf)}$ :  $HR_{Linagliptin \ vs. \ glimepiride} < \delta$ 

 $(H_{1(NonInf)}$ : Linagliptin is non-inferior to glimepiride by the margin  $\delta$  regarding the risk of the primary composite endpoint of cardiovascular events.)

The non-inferiority margin  $\delta$  is chosen to be 1.3 [R09-2151]

If the non-inferiority hypothesis with margin 1.3 has revealed a significant result, then secondly, a superiority hypothesis is tested with respect to time to first occurrence of any of the adjudicated components of the primary composite endpoint.

 $H_{0(Superiority)}$ :  $HR_{linagliptin \ vs. \ glimepiride} \ge 1$  vs.

 $(H_{0(Superiority)})$ : Linagliptin is inferior to glimepiride regarding the risk of the composite primary endpoint of cardiovascular events.)

VS.

H<sub>1</sub>(Superiority): HR<sub>linagliptin vs. glimepiride</sub> < 1

 $(H_{1(Superiority)}:$  Linagliptin is superior to glimepiride regarding the risk of the composite primary endpoint of cardiovascular events.)

If the superiority hypothesis has revealed a significant result, then thirdly, a superiority hypothesis is tested with respect to the first key secondary endpoint

 $H_0(Superiority)$ :  $HR_{linagliptin \ vs. \ glimepiride} \ge 1$  vs.

 $(H_{0(Superiority)})$ : Linagliptin is inferior to glimepiride regarding the risk of the first key secondary endpoint.)

VS.

H<sub>1</sub>(Superiority): HR<sub>linagliptin</sub> vs. glimepiride < 1

(H<sub>1(Superiority)</sub>: Linagliptin is superior to glimepiride regarding the risk of the first key secondary endpoint.)


If the superiority hypothesis has revealed a significant result, then fourthly the second key secondary endpoint will be analysed hierarchically. The second key secondary endpoint (see Section 7.1) will be tested regarding the following hypothesis (p: probability for composite endpoint)

```
H_{0\text{(key secondary 2)}}: p_{\text{linagliptin}} - p_{\text{glimepiride}} = 0 vs
```

 $(H_{0(key\ secondary2\ )}$ : Linagliptin is equal to glimepiride regarding the occurrence of the second key secondary endpoint.)

```
H_{1(\text{key secondary 2})}: p_{\text{linagliptin}} - p_{\text{glimepiride}} \neq 0
```

 $(H_{1(key\ secondary\ 2)}$ : Linagliptin is unequal to glimepiride regarding the occurrence of the second key secondary endpoint.)

If this hypothesis has revealed a significant result, then fifthly the third key secondary endpoint will be tested hierarchically regarding the following hypothesis:

```
H_{0\text{(key secondary 3: }p_{\text{linagliptin}}} - p_{\text{glimepiride}} = 0 vs
```

 $(H_{0(key\ secondary\ 3)}$ : Linagliptin is equal to glimepiride regarding the occurrence of the third key secondary endpoint.)

```
H_{1(key\ secondary\ 3)}: p_{linagliptin} - p_{glimepiride} \neq -0
```

 $(H_{1(key\ secondary\ 3)}:$  Linagliptin is unequal to glimepiride regarding the occurrence of the third key secondary endpoint.)

Any confirmatory hypothesis test will be performed on the full analysis set.

### 7.3 PLANNED ANALYSES

The primary analysis will be performed on the full analysis set (FAS). The FAS will consist of all randomised patients who were treated with at least one dose of study drug.

For the primary and key secondary endpoints a 'classical intention to treat (ITT) analysis on the FAS' will be done. That means that:

- the patient set consists of the FAS,
- the allocated study treatment at randomisation will be used for the FAS of patients for analysis ('as randomised')
- all events which occurs until study end will be taken into account.

A per protocol set (PPS) of patients following the trial protocol in essential criteria will be created for sensitivity analyses. Patients included in the FAS who have important protocol violations will be excluded from the PPS. A protocol violation will be considered important if it can be expected to have a distorting influence on the assessment of the primary endpoint and/or first key secondary endpoints.

Important protocol violations include:

- Randomised study drug: incorrect active study drug taken.
- Severe violation of treatment compliance (defined as less than 50% of visits from Visit 3 on (excluding placebo run-in phase) with treatment compliance outside 80-120% range.
- Non-adherence to other specifications of the protocol that could bias the primary endpoint

Additionally 30-days-treatment set of patients will be created for sensitivity analysis. The 30-days-treatment set will include all randomised patients with a minimum treatment duration of 30 days.

All patients treated with at least one dose of study drug (the Treated Set) will be included in the safety evaluation.

### 7.3.1 Primary analyses

The one-sided overall significance level will be alpha=2.5%. For the primary analysis a 'classical ITT-analysis on the FAS will be performed as described above. For the primary analysis a cox proportional hazards regression model of time to the first event with factor treatment will be conducted. The non-inferiority margin will be 1.3.

As described in Section 7.3.4 the DMC will perform formal interim analyses. The overall significance level of 2.5% will be allocated to the DMC-interim analyses and the final analysis according to the O'Brien & Fleming alpha-spending function. The O'Brien & Fleming alpha-spending function defined the significance level for the first interim analysis on 4P-MACE.

Due to the change of the primary endpoint after the first DMC interim analysis a Bonferroni adjustment will be applied in addition, to control the overall alpha-level. That means, the alpha spent at the first DMC interim analysis (performed for 4P-MACE and based on the O'Brien & Fleming alpha-spending function) is subtracted from the initial overall alpha. The O'Brien & Fleming alpha-spending function based on the new overall alpha (after additional Bonferroni adjustment) defines the allocation of the still available overall significance level for the second interim analysis and the final analysis.

The significance levels for the analyses are denoted by  $\alpha_i$ , i=1,...,3. The total number of analyses is three, including 2 interim analyses.

In the i-th analysis,  $i=1,\ldots,3$ , the upper limit of the two sided  $(1-2*\alpha_i)*100\%$ -confidence interval of the hazard ratio will be compared with the non-inferiority margin. Also the one-sided p-value of the non-inferiority test based on the Wald chi-squared statistic will be given. If the non-inferiority test satisfies the non-inferiority margin, a superiority test (Wald chi-squared statistic) will be performed. If the superiority test has revealed a significant result, a superiority test on the first key secondary endpoint will be performed on the same significance level as for the primary endpoint. If the superiority test has revealed a significant result, the second and third key secondary endpoints will be tested hierarchically (see Section 7.2.). The second and third key secondary endpoints will be analysed with Chi-Square test on the same significance level  $(2*\alpha_i)*100\%$  as the primary endpoint.

No centre effect is included into the model, as the centre size is expected to be small. Furthermore, due to the low event rate there would not be a sufficient number of events per centre for the analysis of a centre effect and a centre by treatment interaction.

For the primary endpoint sensitivity analyses will be done on the PPS, the 30-days-treatment set and as an 'on-treatment analysis' as described below. For the first key secondary endpoint sensitivity analyses will be done on the PPS and as an 'on-treatment analysis' as described below. These sensitivity analyses will be performed based on the corresponding patient sets for the time patients are on-treatment + 30 days after permanent treatment discontinuation or end of observation, whichever comes first.

The 'on-treatment analysis' will be performed on the FAS (consisting of all randomised patients who were treated with at least one dose of study drug) with censoring at the time patients are on treatment + 30 days after permanent treatment discontinuation or end of observation, whichever comes first.

For all these sensitivity analyses the allocated study treatment at randomisation will be used for treatment assignment.

For the second and third key secondary endpoints sensitivity analyses will be done on the PPS and the 30-days-treatment set. For the sensitivity analysis on the 30-days-treatment set patients who prematurely discontinue study treatment will not be counted as non-responders as in the primary analysis for the second and third key secondary endpoints. The measurement of Final Visit will be used. For the sensitivity analysis on the PPS patients who prematurely discontinue study treatment will be counted as non-responders as in the primary analysis. For both sensitivity analyses the allocated study treatment at randomisation will be used for treatment assignment.

### 7.3.2 Secondary analyses

All other secondary analyses are of exploratory nature, no correction for multiple hypotheses testing will be made. All statistical tests and confidence intervals are two-sided with a significance level of alpha=0.05 and will include the factor treatment, unless stated otherwise.

For all cardiovascular endpoints that include time-to-event data the same models and testing procedures as the primary analysis will be applied to compare the two treatment groups.

For continuous secondary diabetes related endpoints with several on-treatment measurements change from baseline will be evaluated with a restricted maximum likelihood (REML) based mixed model repeated measures (MMRM) approach with fixed, categorical effects of treatment, week, treatment-by-week interaction, with the continuous covariates of baseline and baseline-by-week interaction. For those continuous secondary diabetes related endpoints with only one measurement on treatment an analysis of covariance (ANCOVA) model with the factor treatment and the baseline value of the respective variable as covariate will be performed. For qualitative secondary diabetes related endpoints, a Chi-Square test is used to compare the two treatment groups.

### 7.3.3 Safety analyses

All safety data will be displayed and analysed using descriptive statistical methods. No formal inferential analysis is planned for safety comparison. AEs will be coded using the MedDRA coding dictionary. All events with an onset after the first dose of study medication up to a period of seven days after the last dose of study medication will be assigned to the treatment phase for evaluation. Other AEs will be assigned either to the screening or follow-up phase as appropriate. Laboratory values taken after the first dose of randomised treatment up to a period of seven days after the last

intake of treatment will be assigned to the treatment phase for evaluation. Laboratory values will be compared to their reference ranges and frequency tables will be provided for the number of patients within and outside the reference range. Changes from baseline in blood pressure and pulse rate will be summarised by treatment group.

### 7.3.4 Interim analyses

An independent Data Monitoring Committee (DMC) will review safety and efficacy data and make recommendations whether to continue the study, continue the study with modifications, or terminate the study. As described in Section 3.1.1 the DMC analyses and operations will be formally separated from the sponsor, the investigators and the Steering committee.

The DMC will perform formal interim analyses of the primary endpoint for non-inferiority and superiority. The trial team and Steering Committee stay blinded for these interim analyses. The sponsor will perform the final analysis. To prevent an inflation of the significance level a group sequential design according to the alphaspending approach [R97-0643] is chosen. The O'Brien & Fleming alpha-spending function defines the allocation of the overall significance level to the analyses.

The O'Brien & Fleming alpha-spending function defined the significance level for the first interim analysis on 4P-MACE. Due to the change of the primary endpoint after the first DMC interim analysis a Bonferroni adjustment will be applied in addition, to control the overall alpha-level. That means, the alpha spent at the first DMC interim analysis (performed for 4P-MACE and based on the O'Brien & Fleming alpha-spending function) is subtracted from the initial overall alpha. The O'Brien & Fleming alpha-spending function based on the new overall alpha (after additional Bonferroni adjustment) defines the allocation of the still available overall significance level for the second interim analysis and the final analysis.

The second interim analysis will be performed based on approximately 411 primary endpoint events. The final analysis will take place after the observation of a minimum of 631 primary endpoint events.

The trial will be terminated after a formal DMC-interim analysis, if superiority for linagliptin can be shown with respect to cardiovascular safety, with particular emphasis on CV mortality. The trial should be terminated after DMC interim analysis for futility, if superiority of glimepiride with respect to the primary endpoint can be shown prematurely or if a futility assessment shows that the 1.3 non-inferiority margin likely will not be met.

The criteria for stopping the trial after a DMC-interim analysis in favour for the alternative hypothesis are given by the alpha-spending function according to O'Brien and Fleming and an additional Bonferroni adjustment applied after the first DMC interim analysis for 4P-MACE and the following analyses regarding 3P-MACE to control the overall alpha-level, with the possibility to stop the trial in favour for the alternative. The bounds of the group sequential design  $(\alpha_i, i=1,...3)$  result from an overall  $\alpha=2.5\%$ , number of events for final analysis= 631 and the chosen alpha-

spending function [R10-2517] and the additional Bonferroni adjustment for the second interim and final analysis.

The first formal DMC-interim analysis of the primary endpoint should be based on a minimum number of 80 adjudicated primary outcome events and a minimum duration of 1.5 years after the randomisation of the first patient. The Power of such an interim analysis would be > 80%, if the true HR is extraordinary low.

The DMC will perform periodic safety reviews with an emphasis on cardiovascular and neurological events and CV mortality. The frequency of these reviews is detailed in the DMC charter, but additional looks may be scheduled as needed by the DMC. In addition, the Steering Committee may also request the DMC to meet for a safety review.

### 7.4 HANDLING OF MISSING DATA

Patients with temporary or permanent study treatment termination will be followed up for cardiovascular events.

### Cardiovascular safety and other safety endpoints

With respect to safety evaluations, it is not planned to impute missing values.

### Diabetes related endpoints

The REML based MMRM analysis will handle missing data for continuous diabetes related endpoints for patients who discontinue the study treatment prematurely or miss a visit. This approach is valid, if missing observations are missing at random. Missing data for binary efficacy endpoints for patients who discontinue the study treatment prematurely will be considered as non-responders (worst case-scenario).

Methods to handle any other exceptional cases will be considered before unblinding the data and will be applied in a manner consistent with other trials of this type. The evaluability of patients with deviations from the protocol likely to confound the primary endpoint will be decided prior to unblinding.

The last observation carried forward (LOCF) approach will be performed in a sensitivity analysis on diabetes related endpoints.

### 7.5 RANDOMISATION

The sponsor will arrange for the randomisation as well as packaging and labelling of study medication. Eligible patients will be randomly assigned to one of the two treatment groups, with equal allocation of treatments The randomisation list will be generated using a validated system, which involves a pseudo-random number generator so that the resulting treatment sequence will be both reproducible and non-predictable.

The randomisation will be performed in blocks. The block size will be reported in the CTR. Stratification by centre will be achieved by allocating complete blocks for each site. The allocation process will be performed on Visit 2 through an interactive voice and web-based response system (IXRS).

Except for the DMC, access to the code will be restricted to dedicated randomisation personnel and any exceptional access to the code (in case of an emergency) will be documented according to the sponsor's SOPs.

The study will only be unblinded after all CRF / electronic data have been entered into the trial database, after queries have been resolved and after the database has been locked. Access to the codes will be controlled and documented by a signed confidentiality statement, which will be stored in the CTMF.

Practical aspects of the treatment allocation process and methods to carry out blinding are detailed in Sections 4.1.2 and 4.1.5, respectively.

### 7.6 DETERMINATION OF SAMPLE SIZE

A group sequential design with according to the alpha-spending approach [R97-0643] was chosen. The critical values and the test characteristics of the group sequential test design are calculated according to the O'Brien & Fleming alpha-spending function with an additional Bonferroni adjustment applied after the first DMC interim analysis for 4P-MACE and the following analyses based on 3P-MACE.

The overall Power depends on the number and time points of interim analyses. Therefore the overall Power cannot be calculated explicitly. Therefore the Power will be given for a one-stage design without any interim analyses.

In a one-stage trial, for specified  $\alpha$ = 2.5%, and assuming equal risk between the two treatments (HR = 1.0) the Power for showing non inferiority (non-inferiority margin=1.3) will be 90.9% if the log rank test is performed at 631 number of accumulated events.

The computation assumes an allocation ratio of 1:1.

Assuming 1-year event rates of 0.018 for the glimepiride group and 0.018 for the linagliptin group and an accrual time of 2 years and a follow-up time of 5.4 years and a 1-year loss to follow-up rate of 1.5% a total of 6000 patients is expected to yield the necessary number of events.

In a one-stage trial, with 1-year event rates of 0.018 for the glimepiride group and 0.0144 for the linagliptin group (HR = 0.8) the Power for showing superiority will be 80% if the log rank test is performed at 631 number of accumulated events. Assuming an accrual time of 2 years and a follow-up time of 6.2 years and a 1-year loss to follow-up rate of 1.5% a total of 6000 patients is expected to yield the necessary number of events.

The sample size calculations were calculated with Addplan 4.0.3 [R10-2517].

**Boehringer Ingelheim** 

## 8. INFORMED CONSENT, DATA PROTECTION, TRIAL RECORDS

The trial will be carried out in compliance with the protocol, the principles laid down in the Declaration of Helsinki in accordance with the ICH Harmonised Tripartite Guideline for Good Clinical Practice (GCP) and relevant BI Standard Operating Procedures (SOPs). Standard medical care (prophylactic, diagnostic and therapeutic procedures) remains in the responsibility of the treating physician of the patient.

The investigator should inform the sponsor immediately of any urgent safety measures taken to protect the study patients against any immediate hazard, and also of any serious breaches of the protocol/ICH GCP.

For Japan: and the Japanese GCP regulations (Ministry of Health and Welfare Ordinance No. 28, March 27, 1997).

The rights of the investigator (for Japan: trial site) and of the sponsor with regard to publication of the results of this trial are described in the investigator contract (for Japan: trial site). As a general rule, no trial results should be published prior to finalisation of the Clinical Trial Report.

<u>Insurance Cover:</u> The terms and conditions of the insurance cover are made available to the investigator and the patients via documentation in the ISF (Investigator Site File).

### 8.1 STUDY APPROVAL, PATIENT INFORMATION, AND INFORMED CONSENT

This trial will be initiated only after all required legal documentation has been reviewed and approved by the respective Institutional Review Board (IRB) / Independent Ethics Committee (IEC) and competent authority (CA) according to national and international regulations. The same applies for the implementation of changes introduced by amendments.

Prior to patient participation in the trial, written informed consent must be obtained from each patient (or the patient's legally accepted representative) according to ICH GCP and to the regulatory and legal requirements of the participating country. Each signature must be personally dated by each signatory and the informed consent and any additional patient-information form retained by the investigator as part of the trial records. A signed copy of the informed consent and any additional patient information must be given to each patient or the patient's legally accepted representative.

For Japan: The investigator must give a full explanation to trial patients by using the patient information form, which is prepared avoiding the use of technical terms and expressions. The patient is given sufficient time to consider participation in the trial. The investigator obtains written consent of the patient's own free will with the informed consent form after confirming that the patient understands the contents. The investigator must sign (or place a seal on) and date the informed consent form. If a trial collaborator has given a supplementary explanation, the trial collaborator also signs (or places a seal on) and dates the informed consent.

The respective procedure for illiterate patients is described in the Appendix <u>10.1</u>.

The patient must be informed that his/her personal trial-related data will be used by Boehringer Ingelheim in accordance with the local data protection law. The level of disclosure must also be explained to the patient.

The patient must be informed that his / her medical records may be examined by authorised monitors (CML/CRA) or Clinical Quality Assurance auditors appointed by Boehringer Ingelheim, by appropriate IRB / IEC members, and by inspectors from regulatory authorities.

### 8.2 DATA QUALITY ASSURANCE

In order to achieve a high level of standardised processes, data collection of efficacy and safety endpoints is coordinated centrally:

- Central lab analysis of efficacy endpoints and safety lab
- Central ECG collection
- Central IXRS for randomisation and kit allocation at each visit
- Central Outcome event adjudication process

The data management procedures to ensure the quality of the data are described in detail in the trial data management and analysis plan (TDMAP) available in CTMF.

A quality assurance audit/inspection of this trial may be conducted by the sponsor or sponsor's designees or by IRBs/IECs or by regulatory authorities. The quality assurance auditor will have access to all medical records, the investigator's trial-related files and correspondence, and the informed consent documentation of this clinical trial.

### 8.3 RECORDS

Case Report Forms (CRFs) for individual patients will be provided by the sponsor, either on paper or via remote data capture. See Section <u>4.1.5.2</u> for rules about emergency code breaks. For drug accountability, refer to Section <u>4.1.8.</u>

### 8.3.1 Source documents

Source documents provide evidence for the existence of the patient and substantiate the integrity of the data collected. Source documents are filed at the investigator's site.

Data reported entered in the eCRFs that are transcribed from source documents must be consistent with the source documents or the discrepancies must be explained. The investigator may need to request previous medical records or transfer records, depending on the trial; also current medical records must be available.

For eCRFs all data must be derived from source documents.

#### 8.3.2 Direct access to source data and documents

The investigator / institution will permit trial-related monitoring, audits, IRB / IEC review and regulatory inspection, providing direct access to all related source data / documents. CRFs/eCRFs and all source documents, including progress notes and

copies of laboratory and medical test results must be available at all times for review by the sponsor's clinical trial monitor, auditor and inspection by health authorities (e.g. FDA). The Clinical Research Associate (CRA) / on site monitor and auditor may review all CRFs/eCRFs, and written informed consents. The accuracy of the data will be verified by reviewing the documents described in Section 8.3.1.

### 8.3.3 Storage of records

For Japan:

Storage period of records:

*Trial site(s):* 

The trial site(s) must retain the source documents and essential documents for a period defined by the Japanese GCP regulation and the Sponsor's SOP.

Sponsor:

The sponsor must retain the essential documents according to the Sponsor's SOP.

When it is no longer necessary for the trial site to retain source documents and essential documents, the sponsor must notify the head of the trial site.

### 8.4 LISTEDNESS AND EXPEDITED REPORTING OF ADVERSE EVENTS

### 8.4.1 Listedness

To fulfil the regulatory requirements for expedited safety reporting, the sponsor evaluates whether a particular adverse event is "listed", i.e. is a known side effect of the drug or not. Therefore a unique reference document for the evaluation of listedness needs to be provided. For linagliptin this is the current version of the Investigator's Brochure [U04-1767]. For glimepiride this is the EU SPC (Amaryl). The current versions of these reference documents are to be provided in the ISF. No AEs are classified as listed for matching placebo, study design, or invasive procedures.

### 8.4.2 Expedited reporting to health authorities and IECs/IRBs

Expedited reporting of serious adverse events, e.g. suspected unexpected serious adverse reactions (SUSARs) to health authorities and IECs/IRBs, will be done according to local regulatory requirements. Cardiovascular outcome events that occur after randomisation and represent a SAE, are exempted from expedited reporting to health authorities. Further details regarding this reporting procedure are provided in the Investigator Site File.

### 8.5 STATEMENT OF CONFIDENTIALITY

Individual patient medical information obtained as a result of this trial is considered confidential and disclosure to third parties is prohibited with the exceptions noted below. Patient confidentiality will be ensured by using patient identification code numbers.

Treatment data may be given to the patient's personal physician or to other appropriate medical personnel responsible for the patient's welfare. Data generated as a result of the trial need to be available for inspection on request by the participating physicians, the sponsor's representatives, by the IRB / IEC and the regulatory authorities. For EU, i.e. the CA.

### 8.6 COMPLETION OF TRIAL

For Japan: When the trial is completed, the investigator should inform the head of the trial site of the completion in writing, and the head of the trial site should promptly inform the IRB and sponsor of the completion in writing.

For EU member states: The EC/competent authority in each participating EU member state needs to be notified about the end of the trial (last patient/patient out, unless specified differently in Section 6.2.3 of the CTP) or early termination of the trial.

### 8.7 PROTOCOL VIOLATIONS

The investigator should document any deviations from the protocol regardless of their reasons. Only when the protocol was not followed in order to avoid an immediate hazard to trial subjects or for other medically compelling reason, the principal investigator should prepare and submit the records explaining the reasons thereof to the sponsor, and retain a copy of the records.

For Japan: The investigator or sub-investigator should record all CTP violations. The investigator should provide and submit the sponsor and the head of the trial site the records of violations infringing the Japanese GCP or violations to eliminate an immediate hazard to trial patients and for other medically inevitable reasons.

## 8.8 COMPENSATION AVAILABLE TO THE PATIENT IN THE EVENT OF TRIAL RELATED INJURY

For Japan only: In the event of health injury associated with this trial, the sponsor is responsible for compensation based on the contract signed by the trial site.

#### 9. REFERENCES

#### 9.1 PUBLISHED REFERENCES

- P08-01788 Ryden L. Standl E. Bartnik M. Berghe G van den. Betteridge J. Boer MJ de, Cosentino F, Jonsson B, Laakso M, Malmberg K, Priori S, Ostergren J, Tuomilehto J, Thrainsdottir I. Guidelines on diabetes, prediabetes, and cardiovascular diseases: full text: the Task Force on Diabetes and Cardiovascular Diseases of the European Society of Cardiology (ESC) and of the European Association for the Study of Diabetes (EASD). Eur Heart J 9 (Suppl C), C3 - C74 (2007)
- R10-0116 Vaccaro O, Eberly LE, Neaton JD, Yang L, Riccardi G, Stamler J, Multiple Risk Factor Intervention Trial (MRFIT) Research Group. Impact of diabetes and previous myocardial infarction on long-term survival: 25-year mortality follow-up of primary screenees of the Multiple Risk Factor Intervention Trial. Arch Intern Med 164, 1438 -1443 (2004)
- R10-0117 Gu K, Cowie CC, Harris MI. Mortality in adults with and without diabetes in a national cohort of the U.S. population, 1971 - 1993. Diabetes Care 21 (7), 1138 – 1145 (1998)
- R07-1076 International Diabetes Federation, Clinical Guidelines Task Force. Global guideline for type 2 diabetes. Brussels: International Diabetes Federation (2005)
- R09-6397 Asian-Pacific Type 2 Diabetes Policy Group. Type 2 diabetes: practical targets and treatments. 4th ed. Melbourne, Singapore: International Diabetes Institute, In Vivo Communications (Asia) (2005)
- AACE Diabetes Mellitus Clinical Practice Guidelines Task Force R08-1310 American association of clinical endocrinologists medical guidelines for clinical practice for the management of diabetes mellitus. Endocr Pract 13 (Suppl 1), 3 - 68 (2007)
- R10-4077 National Institute for Health and Clinical Excellence. Type 2 diabetes: newer agents for blood glucose control in type 2 diabetes (this short clinical guideline partially updates NICE clinical guideline 66. The recommendations have been combined with unchanged recommendations from CG66 in NICE clinical guideline 87 (NICE short clinical guideline 87, issue date: May 2009). weblink: nice.org.uk ; London: National Institute for Health and Clinical Excellence (2009)
- P08-06509 Johansen OE. Cardiovascular disease and type 2 diabetes mellitus: a multifaceted symbiosis. Scand J Clin Lab Invest 2007;67(8):786-800.

| Boehringer Ingelheim | 20 April 2016 |
|-----------------------|---------------|
| BI Trial No.: 1218.74 | |

| R10-2212 | Williams R, Van Gaal L, Lucioni C, Advisory Board. Assessing the |
|---|---|
| | impact of complications on the costs of Type II diabetes. Diabetologia |
| | 2002;45:S13-7 |

- P10-00533 Canadian Diabetes Association Clinical Practice Guidelines Expert Committee. Canadian Diabetes Association 2008 clinical practice guidelines for the prevention and management of diabetes in Canada. Can J Diabetes 32(suppl 1), S1-S201. 2008
- R09-1164 Nathan DM, Buse JB, Davidson MB, Ferrannini E, Holman RR, Sherwin R, Zinman B; American Diabetes Association; European Association for Study of Diabetes. Medical management of hyperglycemia in type 2 diabetes: a consensus algorithm for the initiation and adjustment of therapy: a consensus statement of the American Diabetes Association and the European Association for the Study of Diabetes. Diabetes Care. 2009;32:193-203.
- R10-0133 Hoerger TJ, Segel JE, Gregg EW, Saaddine JB. Is glycemic control improving in U.S. adults? Diabetes Care 2008;31:81-86
- R10-0134 Liebl A, Mata M, Eschwege E, Advisory Board. Evaluation of risk factors for development of complications in Type II diabetes in Europe. Diabetologia 2002;45:S23-8
- R10-0657 Turner RC, Cull CA, Frighi V, Holman RR. Glycemic control with diet, sulfonylurea, metformin, or insulin in patients with type 2 diabetes mellitus: progressive requirement for multiple therapies (UKPDS 49). UK Prospective Diabetes Study (UKPDS) Group. JAMA. 1999;281:2005-12.
- R09-6400 Kahn SE, Haffner SM, Heise MA, Herman WH, Holman RR, Jones NP, Kravitz BG, Lachin JM, O'Neill MC, Zinman B, Viberti G; ADOPT Study Group. Glycemic durability of rosiglitazone, metformin, or glyburide monotherapy. N Engl J Med. 2006;355:2427-43
- R09-6405 Effect of intensive blood-glucose control with metformin on complications in overweight patients with type 2 diabetes (UKPDS 34). UK Prospective Diabetes Study (UKPDS) Group. Lancet. 1998;352:854-65
- R09-6409 Holman RR, Paul SK, Bethel MA, Matthews DR, Neil HA. 10-year follow-up of intensive glucose control in type 2 diabetes. N Engl J Med. 2008;359:1577-89
- R09-6407 Action to Control Cardiovascular Risk in Diabetes Study Group.

  Effects of Intensive Glucose Lowering in Type 2 Diabetes. N Engl J
  Med 2008; 358(24): 2545-2559

| Boehringer Ingelheim | 20 April 2016 |
|----------------------------------------------|---------------|
| NT TO 1 1 NT 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 1 | |

| R09-6408 | Duckworth W, Abraira C, Moritz T, Reda D, Emanuele N, Reaven PD, Zieve FJ, Marks J, Davis SN, Hayward R, Warren SR, Goldman S, McCarren M, Vitek ME, Henderson WG, Huang GD; VADT Investigators. Glucose control and vascular complications in veterans with type 2 diabetes. N Engl J Med. 2009 Jan 8;360(2):129-139 |
|---|---|
| R10-2210 | Nissen SE, Wolski K, Topol EJ.Effect of muraglitazar on death and major adverse cardiovascular events in patients with type 2 diabetes mellitus. JAMA. 2005;294:2581-6. |
| R10-2211 | Nissen SE, Wolski K. Effect of rosiglitazone on the risk of myocardial infarction and death from cardiovascular causes. N Engl J Med. 2007;356:2457-71 |
| R09-2151 | Guidance for industry: diabetes mellitus - evaluating cardiovascular risk in new antidiabetic therapies to treat type 2 diabetes (December 2008). Silver Spring: U.S.Department of Health and Human Services, Food and Drug Administration, Center for Drug Evaluation and Research (CDER) 2008 |
| R09-6409 | Meier JJ, Nauck MA. Glucagon-like peptide 1 (GLP-1) in biology and pathology. Diabetes Metab Res Rev 2005;21:91–117 |
| R09-6410 | Monami M, Iacomelli I, Marchionni N, Mannucci E. Dipeptydil peptidase-4 inhibitors in type 2 diabetes: a meta-analysis of randomized clinical trials. Nutrition, Metabolism and Cardiovascular Diseases, article in press, doi: 10.1016/j.numecd.2009.03.015 Nutr Metab Cardiovasc Dis 2009 |
| R04-2173 | Turner RC, Holman RR, Cull CA, Stratton IM, Matthews DR, Fright V, Manley SE, Neil A, McElroy H, Wright D, Kohner E, Fox C, Hadden D, UK Prospective Diabetes Study Group. Intensive blood-glucose control with sulphonylureas or insulin compared with conventional treatment and risk of complications in patients with typ 2 diabetes (UKPDS 33). Lancet 1998;352:837-853. |
| R09-6394 | Bell DSH. Practical considerations and guidelines for dosing sulfonylureas as monotherapy or combination therapy. Clin Ther 2004;26(11):1714-1727. |
| R09-6395 | Dormandy JA, et al, PROactive Investigators. Secondary prevention of macrovascular events in patients with type 2 diabetes in the PROactive Study (PROspective pioglitAzone Clinical Trial In macroVascular Events): a randomised controlled trial. Lancet 2005;366:1279-1289. |
| D00 (20) | A 1 D11 A 1 |

R09-6396 American Diabetes Association Workgroup on Hypoglycemia.

Defining and reporting hypoglycaemia in diabetes: a report from the American Diabetes Association Workgroup on Hypoglycemia.

Diabetes Care 2005;28(5):1245-1249.

| R10-2517 | ADDPLAN, 2007. Software for Adaptive Designs and Analyses: |
|----------|------------------------------------------------------------|
| | Release 4. ADDPLAN GmbH, Cologne, Germany. |

| R97-0643 | Lan KKG, DeMets DL. Discrete sequential boundaries for clinical |
|----------|-----------------------------------------------------------------|
| | trials. Biometrika 1983;70(3):659-663. |

- P96-4362 Harrower ADB. Pharmacokinetics of oral antihyperglycaemic agents in patients with renal insufficiency. Clin Pharmacokinet 31 (2), 111 119 (1996)
- R10-4375 Glucophage (metformin hydrochloride tablets), Glucophage XR (metformin hydrochloride extended-release tablets) (Bristol-Myers Squibb Company) (NDA 20-357/S-031, NDA 21-202/S-016, version: 08/27/2008).
- R07-4080 Klein S, Allison DB, Heymsfield SB, Kelley DE, Leibel RL et al. Waist circumference and cardiometabolic risk: a consensus statement from Shaping America's Health: Association for Weight Management and Obesity Prevention; NAASO, The Obesity Society; the American Society for Nutrition; and the American Diabetes Association. Am J Clin Nutr 2007;85:1197-202.
- R10-6494 Vigneri P, FF, Sciacca L, PG, Vigneri R. Diabetes and cancer. Endocr Relat Cancer 2009;16:1103-1123.
- R10-6495 Hemminki K, Li X, Sundquist J, Sundquist K. Risk of cancer following hospitalization for type 2 diabetes. Oncologist 2010;15:548-555.
- R10-6496 Giovannucci E, Michaud D. The role of obesity and related metabolic disturbances in cancers of the colon, prostate, and pancreas.

  Gastroenterology 2007;132(6):2208-2225.
- R10-6497 Smith U, Gale EAM. Does diabetes therapy influence the risk of cancer? Diabetologia 2009;52:1699-1708.
- Xue F, Michels KB. Diabetes, metabolic syndrome, and breast cancer: a review of the current evidence. Am J Clin Nutr 2007;86(Suppl):823S 835S.
- R10-6536 Hjartaker A, Langseth H, Weiderpass E. Obesity and diabetes epidemics: cancer repercussions. In: Berstein LM, Santen RJ, editors.Innovative endocrinology of cancer.Austin: Landes Bioscience 2008:72-93.

| R10-6638 | Giovannucci E, Harlan DM, Archer MC, Bergenstal RM, Gapstur SM, |
|---|---|
| | Habel LA, Pollak M, Regensteiner JG, Yee D. Diabetes and cancer: a |
| | consensus report. Diabetes Care 33 (7), 1674 - 1685 (2010). |

- P15-02848 Marx N, Rosenstock J, Kahn SE, Zinman B, Kastelein JJ, Lachin JM, Espeland MA, Bluhmki E, Mattheus M, Ryckaert B, Patel S, Johansen OE, Woerle HJ Design and baseline characteristics of the CARdiovascular Outcome Trial of LINAgliptin versus glimepiride in type 2 diabetes (CAROLINA). Diabetes Vasc Dis Res 12 (3), 164-174 (2015).
- P13-02826 Rosenstock J, Marx N, Kahn SE, Zinman B, Kastelein JJ, Lachin JM, Bluhmki E, Patel S, Johansen OE, Woerle HJ Cardiovascular outcome trials in type 2 diabetes and the sulphonylurea controversy: rationale for the active-comparator CAROLINA trial. Diabetes Vasc Dis Res 10 (4), 289-301 (2013).
- P16-04169 Pocock SJ. Design of major randomized trials: part 3 of a 4-part series on statistics for clinical trials. J Am Coll Cardiol 2015. 66(24):2757.
- R13-3903 Scirica BM, Bhatt DL, Braunwald E, Steg PG, Davidson J, Hirshberg B, Ohman P, Frederich R, WiviottSD, Hoffman EB, Cavender MA, Udell JA, Desai NR, Mozenson O, McGuire DK, Ray KK, Leiter LA, Raz I, SAVOR-TIMI 53 Steering Committee and Investigators. Saxagliptin and cardiovascular outcomes in patients with type 2 diabetes mellitus.N Engl J Med 369, 1317 1326 (2013).
- White WB, Cannon CP, Heller SR, Nissen SE, Bergenstal RM, Bakris GL, Perez AT, Fleck PR, Mehta CR, Kupfer S, Wilson C, Cushman WC, Zannad F, EXAMINE Investigators. Alogliptin after acute coronary syndrome in patients with type 2 diabetes.N Engl J Med 369 (14), 1327 1335 (2013).
- R16-1123 Pfeffer MA, Claggett B, Diaz R, Dickstein K, Gerstein HC, Kober LV, Lawson FC, Ping L, Wei X, Lewis EF, Maggioni AP, McMurray JJV, Probstfield JL, Riddle MC, Solomon SD, Tardif JC, ELIXA Investigators. Lixisenatide in patients with type 2 diabetes and acute coronary syndrome.N Engl J Med 373 (23), 2247 2257 (2015).
- R15-3017 Green JB, Bethel MA, Armstrong PW, Buse JB, Engel SS, Garg J, Josse R, Kaufman KD, Koglin J, Korn S, Lachin JM, McGuire DK, Pencina MJ, Standl E, Stein PP, Suryawanshi S, Werf F van de, Peterson ED, Holman RR, TECOS Study Group. Effect of sitagliptin on cardiovascular outcomes in type 2 diabetes.N Engl J Med, (2015)
- R09-2151 Guidance for industry: diabetes mellitus evaluating cardiovascular risk in new antidiabetic therapies to treat type 2 diabetes (December 2008). Silver Spring: U.S. Department of Health and Human Services,

Food and Drug Administration, Center for Drug Evaluation and Research (CDER) (2008)

R12-3960 European Medicines Agency (EMA) Committee for Medicinal

Products For Human Use (CHMP): guideline on clinical investigation

of medicinal products in the treatment or prevention of diabetes

mellitus (14 May 2012, CPMP/EWP/ 1080/00 Rev. 1).

### 9.2 UNPUBLISHED REFERENCES

U04-1767 Linagliptin Investigator's Brochure. Current Version.

### 10. APPENDICES

### 10.1 INCLUSION OF ILLITERATE PATIENTS

### 10.1.1 Home blood glucose monitoring

In the event of recruiting an illiterate patient, the following process should be followed with respect to HBGM and documenting the results:

- at Visit 1b, the person assisting the patient with this process (e.g. the patient's caregiver or relative) will attend the clinic together with the patient
- the site staff should confirm that this individual will be present with the patient, whenever he/she is likely to need to perform HBGM
- the site staff should then train both the patient and above-mentioned individual with respect to the correct use of the HBGM equipment during each period of the trial. This will include the use of the glucose meter itself and the test strips, lancet device and control solution(s). Furthermore, if whole blood referenced test strips are standard in the country(ies) where illiterate patients are being recruited, the site staff must ensure that both the patient and the person assisting the patient with the HBGM, have understood that plasma referenced test strips are used in the trial, and that there may be differences in the results obtained via these two methods. A training letter is available to support this process
- the site staff should also train both the patient and the above-mentioned individual with respect to the completion of the HBGM testing log. As for all other patients, the results of all per-protocol HBGM that is performed by/on illiterate patients should be documented on a HBGM testing log that will be included in the patients source document file. In the event of hyper or hypoglycaemia, the person assisting the patient should record symptoms on the HBGM testing log in accordance with the patients' description

HGBM tests can be performed either by the patient him/herself, or by the person assisting the patient with this aspect of the trial.

### 10.1.2 Patient information and informed consent

In the event of recruiting an illiterate patient, the following process should be followed with respect to patient information and informed consent:

- The designated site personnel performing the informed consent process will read the trial-approved patient information sheet and informed consent form to the patient, and explain the details of the trial, all in the presence of an impartial witness
- This impartial witness must be literate, and can be the patient's relative or caregiver, or a member of staff employed by the clinic but not part of the immediate trial team. In addition, if there are any further local regulations with respect to the consent of illiterate patients, these should also be followed

- The requirements of the trial will be explained thoroughly and the patient will be given ample time to ask questions and consider his/her participation. If he/she wishes, the patient can take the patient information sheet and informed consent form home for further consideration
- If patient agrees to take part in the trial, he/she would then return to the clinic for the consent process to be completed. The site designated personnel responsible for this process will confirm that the patient has no further questions in the presence of the same impartial witness (if the patient returns on another day). If a different impartial witness is present, the entire informed consent process must be repeated
- Participating patients will provide a thumb impression or make a mark (or signature if the patient is able to sign him/herself) on the signature section of the informed consent form
- The date of the patient's signature will be left blank as the patient is illiterate. However, if the patient is able, he/she will date the mark/signature personally
- The impartial witness or the site designated personnel may write the name of the patient on the informed consent form
- The impartial witness should enter his/her name, sign and personally date the witness section of the informed consent form. In countries where local data protection regulation permits it, the address or identification number of the impartial witness should also be entered. The signature then attests that the content of the patient information sheet and informed consent form was accurately explained to the patient, who apparently understood and freely gave consent to participate in the trial
- The designated site personnel also signs and personally dates the informed consent form

### 10.2 DEFINITIONS OF ENDPOINT EVENTS

Definitions of the adjudicated endpoints events and the principles of standardised data collection in the centralised CEC adjudication process are outlined in the current CEC Charter and process guideline.

### 10.3 BLOOD PRESSURE MEASUREMENT PROCEDURE AND TREATMENT RECOMMENDATIONS

Initially, blood pressure should be taken three times in both arms. The arm with the mean higher pressure (either systolic - if needed to decide- or diastolic) should be used for subsequent measurements.

Blood pressure measurements can be performed with either a standard mercury sphygmomanometer or an electronic device, i.e. either electronic or manual measurements of blood pressure are acceptable, depending on the standard practice at each study site - Note: Boehringer Ingelheim will not provide electronic devices to sites that use the standard manual sphygmomanometers.

Blood pressure measurements should be performed on the same arm and, if possible, by the same person. The same method must be used throughout the trial, for a given patient, i.e. if a patient receives the first blood pressure measurement for example with an electronic device, the same method and a similar type of device should be used throughout the study for this patient (without switching to manual blood pressure measurement). On the other hand, inter-patients variability is acceptable, i.e. a study site is allowed to consistently use an electronic device to measure the blood pressure in a given patient throughout the study and a manual technique in another patient.

After patients have rested quietly, in the seated position for five minutes, three blood pressure measurements will be taken approximately two minutes apart. The seated pulse rate will be taken during the two-minute interval between the second and third blood pressure reading. If an electronic blood pressure device is used the pulse rate at time of the second or third blood pressure reading may be used.

Blood pressure measurements should be recorded to the nearest 2 mmHg only when measured with a manual sphygmomanometer; when digital devices are used the value from the device should be rounded to the nearest 1 mmHg.

For calculation of mean values, decimal places should be rounded to integers (e.g. a DBP of 94.5 would be rounded to 95 mmHg and a DBP of 109.4 would be rounded to 109 mmHg).

It has been clearly established that the co-existence of hypertension and diabetes increases the risk of developing renal and other organ damage, leading to a much greater incidence of stroke, coronary heart disease, congestive heart failure, peripheral artery disease and cardiovascular mortality. Reduction of high blood pressure could decrease the risk of stroke, heart disease and reduce the likelihood of dementia, heart failure, and death.

Treatment recommendations of hypertension in diabetic patients are described in several guidelines, e.g. the current "Guidelines on Diabetes, pre-diabetes, and cardiovascular diseases of the European Society of Cardiology (ESC) and the European Association for the Study of Diabetes" [P08-01788], also accessible at weblink: escardio.org.

### 10.4 TREATMENT RECOMMENDATIONS FOR DYSLIPIDAEMIA

Increased cardiovascular risk in T2DM patients is independently associated with their hyperglycemia together with high blood pressure (BP) and dyslipidaemia, the last typically the high-density lipoprotein cholesterol (HDL-C) and raised triglyceride (TG) levels found as components of the metabolic syndrome. Although low-density lipoprotein cholesterol (LDL-C) levels are not particularly higher in T2DM patients,

the opportunity to reduce cardiovascular risk is currently greatest through lipid lowering management by reducing LDL-C. There is almost a linear relationship between the absolute risk reduction in LDL-C and the proportional reductions in the incidence of cardiovascular events.

Treatment recommendations of dyslipidaemia in diabetic patients are described in several guidelines, e.g. the current "Guidelines on Diabetes, pre-diabetes, and cardiovascular diseases of the European Society of Cardiology (ESC) and the European Association for the Study of Diabetes" [P08-01788], also accessible at weblink: escardio.org.

### 10.5 SILENT MYOCARDIAL INFARCTION

Incidence and impact of silent MI will be assessed in this study.

Definition of relevant ECG abnormalities related to silent MI is the presence of:

- Any Q-wave in leads  $V2-V3 \ge 0.02$  seconds or QS complex in leads V2 and V3
- Q-wave ≥ 0.03 seconds and ≥ 0.1 mV deep or QS complex in leads I, II, aVL, aVF, or V4-V6 in any two leads of a contiguous lead grouping (I, aVL, V6; V4-V6; II, III, and aVF)
- R-wave  $\geq 0.04$  seconds in V1-V2 and R/S  $\geq 1$  with a concordant positive T-wave in the absence of a conduction defect

An MI will only be classified as silent if 1) the ECG criteria's are fulfilled, 2) the ECG changes were absent from baseline or previous ECGs and 3) no preceding clinical history of MI (including stent thrombosis and other coronary events) during study follow-up occurred and 4) investigator reporting of silent MI.

### 10.6 CLINICAL EVALUATION OF LIVER INJURY

### 10.6.1 Introduction

Alterations of liver laboratory parameters, as described in Section <u>5.2.2.1</u> (protocol specific adverse events of special interest) are to be further evaluated using the following procedures:

### 10.6.2 Procedures

Repeat the following lab tests: ALT, AST, total bilirubin (with differentiation of bilirubin in direct and indirect) and additionally alkaline phosphates (ALP), CK (CK-MB, if CK is elevated), amylase, lipase, INR - within 48 to 72 hours and provide additional blood sample to the central laboratory for automatic reflex testing of the below listed laboratory parameters. Only in case whereby the central laboratory is not immediately available (e.g. if the logistics are such that the patient's repeat specimen would not reach the central laboratory in a reasonable timeframe), ALT, AST, total bilirubin (with differentiation of bilirubin in direct and indirect) and additionally alkaline phosphates (ALP), CK (CK-MB, if CK is elevated), amylase, lipase, INR will be evaluated by local laboratory and results are made available to the investigator


Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19

and to BI as soon as possible. If in such a case ALT and/or AST  $\geq 3$  fold ULN combined with an elevation of total bilirubin  $\geq 2$  fold ULN are confirmed, results of the laboratory parameters described below must be made available to the investigator and to BI as soon as possible.

### In addition,

- initiate close observation of subjects by repeat testing of ALT, AST, alkaline phosphates (ALP), CK (CK-MB, if CK is elevated), total bilirubin (with differentiation of bilirubin in direct and indirect), amylase, lipase, INR with repeated testing of these parameters at least weekly until ALT and or AST abnormalities stabilize or return to normal, then according to the protocol. Depending on further laboratory changes, additional parameters identified e.g. by reflex testing will be followed up based on medical judgement and Good Clinical Practices (GCP).
- initiate examination for alternative reasons for elevation of liver parameters:
  - obtain a detailed history of current symptoms and concurrent diagnoses and medical history according to the "DILI checklist" provided in the ISF
  - obtain history of concomitant drug use (including non-prescription medications and herbal and dietary supplement preparations), alcohol use, recreational drug use, and special diets according to the "DILI checklist" provided in the ISF
  - obtain a history of exposure to environmental chemical agents (consider home and work place exposure) according to the "DILI checklist" provided in the ISF

### and report these via the CRF.

- obtain further lab tests to evaluate for alternative causes (need to be done once):
  - Hepatitis-Serology:
    - Anti-HAV-IgM,
    - HBsAg, HBcAg, anti-HBs (for documentation of probably non-acute infection) (if any are positive then HBV DNA by PCR),
    - Anti-HCV (if positive then HCV RNA by PCR);
    - Anti-HDV IgM;
    - Anti-HEV (if positive then Anti-HEV IgM or HEV-RNA by PCR);
    - Epstein-Barr-Virus: VCA-IgG, VCA-IgM, or early antigen
    - Cytomegalovirus (anti CMV-IgG and anti CMV-IgM)
    - Herpes Simples virus (IgG, IgM)

### ${\bf Proprietary\ confidential\ information.}$

- Parvovirus (IgG, IgM)
- Toxoplasmosis (IgG, IgM)
- Screen for autoimmune hepatitis (ANA, SMA, AMA, anti-LKM)
- Metabolic screen (glucose, cholesterol, triglycerides)
- Coeruloplasmin, alpha-a antitrypsin,
- obtain further information on medical history and additional data as far as possible, use the 'DILI' checklist in the ISF for collecting the information.
- Provide abdominal ultrasound to rule out biliary tract, pancreatic or intrahepatic pathology, e.g. bile duct stones or neoplasm.

### 10.6.3 Decision to Stop Drug Administration

Based on the potential risk for a patient, it can be necessary to discontinue study drug treatment. This decision should be made in close cooperation between the investigator and Boehringer Ingelheim.

# 11. SUMMARY OF CLINICAL TRIAL PROTOCOL MODIFICATIONS

**Summary of Clinical Trial Protocol Modifications Sheet (SOMS)** 

| Number of CTP modification | 1 |
|---|---|
| Date of CTP modification | 21 July 2011 |
| EudraCT number | 2009-013157-15 |
| BI Trial number | 1218.74 |
| BI Investigational Product(s) | Linaglitin |
| Title of protocol | A multicentre, international, randomised, parallel group, double blind study to evaluate Cardiovascular safety of linagliptin versus glimepiride in patients with type 2 diabetes mellitus at high cardiovascular risk. The CAROLINA Trial. |
| To be implemented only | |
| after approval of the | |
| IRB/IEC/Competent Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Can be implemented without | |
| IRB/IEC/ Competent | |
| Authority approval as | |
| changes involve logistical or | |
| administrative aspects only | |
| Section to be changed | Protocol synopsis (objectives) |
| Description of change | Description of treatment sustainability |
| Rationale for change | To correct definition of treatment sustainability |
| Section to be changed | Protocol synopsis (inclusion criteria) |

Protocol Revision 6 

| Description of shares | Changa 1: |
|---|---|
| Description of change | Change 1: Inclusion of patients with background |
| | medication of |
| | - sulphonylurea + alpha-glucosidase |
| | inhibitor or |
| | - glinide + alpha-glucosidase inhibitor |
| | Change 2: Documented coronary artery disease (≥50% luminal diameter narrowing of left main |
| | coronary arteries in angiogram). |
| | Change 3: Peripheral occlusive arterial disease will include stenting as inclusion criterion. |
| | Change 4: Since blood pressure and LDL are not measured at V1a, these values should be known prior study enrolment if used for inclusion (values < 6 months old prior V1a). |
| | Change 5:<br>BMI $\leq$ 45 kg/m <sup>2</sup> at Visit 1b |
| | Change 6: Addition of inclusion criterion: stable antidiabetic background medication (unchanged daily dose) for at least 8 weeks prior V1a and without short term use of insulin. Background medication should be stable during screening/run-in phase to allow randomisation |
| | Change 7: Limitation of recruitment of patients of Category C and D. |
| Rationale for change | Change 1: |
| | Combination therapy of sulphonylurea/glinide + alpha-glucosidase |
| | inhibitor is a suitable combination therapy for the protocol target population |
| | Change 2: |
| | To clarify that $\geq 50\%$ luminal diameter narrowing is documented in at least two |

20 April 2016

Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19

**Protocol Revision 6** 


| | major coronary arteries Including note for |
|---|---|
| | major coronary arteries. Including note for further clarification. |
| | Change 3: To allow stenting cardiovascular risk |
| | Change 4: (inclusion criterion 3) To clarify current blood pressure and LDL measurements if used for inclusion. |
| | Change 5: BMI will be measured at V1b |
| | Change 6: Medication should be stable 8 weeks prior V1a to allow enrolment) and during screening/run-in phase (to allow randomisation) |
| | Change 7: Since the cardiovascular risk is relatively lower for patients of category C and D compared to category A and B, recruitment of patients of category C will be limited to approximately 25% and recruitment of patients of category D will be limited to approximately 25% of total amount of randomised patients. This will be arranged on regional/country level. |
| Section to be changed | Protocol synopsis (duration of treatment) |
| Description of change | Observational study duration is clarified |
| Rationale for change | To clarify observational study duration |
| Section to be changed | Protocol synopsis (Criteria for efficacy) |
| Description of change | Description of primary efficacy endpoint |
| Rationale for change | To be in line with section 5.1.1. |
| Section to be changed | Protocol synopsis (main exclusion |
| | criteria) |
| Description of change | Change 1: Treatment with other diabetic drugs (as specified in inclusion criteria) prior informed consent is excluded. This included also clinical trials where these antidiabetic drugs have been provided to patients. |
| | Change 2:<br>Sibutramine and orlistat were removed as specifically named anti-obesity drugs |

20 April 2016

**Protocol Revision 6** 


| | Changa 2: |
|---|---|
| | Change 3: Pre-planned coronary artery revascularisation (PCI, CABG) within next 6 months after V1a or any previous PCI ≤ 6 months prior informed consent or any previous CABG < 3 months prior informed consent |
| | Change 4: (new exclusion criterion) Exclusion of acute coronary syndrome ≤ 6 weeks prior to informed consent |
| | Change 5: (new exclusion criterion) Exclusion of stroke or TIA ≤ 3 months prior to informed consent |
| Rationale for change | Change 1: To ensure other antidiabetic drugs are also excluded if prescribed in another clinical trial. |
| | Change 2: To remove specific anti-obesity medication and prevent need for future revisions when available products of this class may chance. |
| | Change 3: To exclude recent PCI and CABG |
| | Change 4: (new exclusion criterion) To ensure that patients with acute coronary syndrome ≤ 6 weeks prior to informed consent are not included. |
| | Change 5: (new exclusion criterion) To ensure that patients with stroke or TIA ≤ 3 months prior to informed consent are not included. |
| Section to be changed | Flow Chart |
| Description of change | Change 1: Interactive Voice and Web-based Response System will be used, so called IXRS |
| | Change 2: At Visit 15 and Visit 30 (EOT/EOS) cognition testing will be performed. As a |

| | 1, 1 |
|---|---|
| | result at these visit also HBGM will be done prior testing. |
| | Change 3: (footnote L) The FPG range is more specified for cognitive testing. |
| | Change 4: (footnote J) Between V1a and V1b AEs should also be collected in screen failures prior V1b. |
| | Change 5: (new footnote J) Maximal time window between visits is specified. |
| | Change 6: (footnote M) Clinically relevant abnormalities found at physical examination, vital signs or ECG that are not pre-existing prior to signing of informed consent (study inclusion) should be reported as adverse events. |
| | <u>Change 7</u> : (footnote O) |
| Rationale for change | Change 1: To clarify that Interactive Voice and Webbased Response System will be used, so called IXRS |
| | Change 2: To ensure FPG levels are within range to measure cognition data. |
| | Change 3: (footnote L) The HBGM results at certain FPG concentrations may allow repeated HBGM after at least one hour. |
| | Change 4: (footnote J) To ensure all AEs will be captured, also in screen failures prior V1b. |
| | Change 5: (new footnote J) To ensure patient will not run-out of study medication |
| | <u>Change 6</u> : (footnote M) |


**Protocol Revision 6** 

| | To ensure that clinically relevant |
|-----------------------|------------------------------------------------|
| | abnormalities will be reported as adverse |
| | events if not pre-existing prior signing of |
| | informed consent. |
| | informed consent. |
| | <u>Change 7</u> : (footnote O) |
| Section to be changed | 2.1 |
| Description of change | Inclusion of patients with background |
| | medication of |
| | - sulphonylurea + alpha-glucosidase |
| | inhibitor or |
| | - glinide + alpha-glucosidase inhibitor |
| Rationale for change | Combination therapy of |
| | sulphonylurea/glinide + alpha-glucosidase |
| | inhibitor is a suitable combination therapy |
| | for the protocol target population |
| Section to be changed | 2.2 |
| Description of change | Change 1: |
| | Description of primary objectives |
| | Change 2: |
| | Description of treatment sustainability |
| Rationale for change | Change 1: |
| | Description of primary objectives was |
| | missing in this Section |
| | Change 2: |
| | To correct the definition of treatment |
| | sustainability. |
| Section to be changed | 2.3 |
| Description of change | Reference to linagliptin's phase III program. |
| Rationale for change | Linagliptin's phase III program has been |
| | completed for registration. |
| Section to be changed | 3.1.1 |
| Description of change | Change 1: |
| 1 2 2 3 | Steering Committee (SC) and Data |
| | Monitoring (DMC) Charters won't be |
| | provided in ISF |
| | 1 |
| | Change 2: |
| | Description of inclusion of treatment naïve |
| | T2DM patients. |
| Rationale for change | Change 1: |
| Radionale for change | SC and DMC procedures are not required |
| | for sites. If required, the Charter(s) will be |
| | 101 sites. If required, the Charter(s) will be |

 $\label{proprietary confidential information.} Proprietary \ confidential \ information.$ 

**Protocol Revision 6** 


| | submitted to IEC/IRB or Health Authority |
|---|---|
| | for notification. |
| | Change 2: |
| | To clarify that treatment naive T2DM |
| | patients should be offered first line therapy (e.g. metformin) before allowing them for |
| | study inclusion, unless they have specific |
| | contra-indications to its use. |
| Section to be changed | 3.2 |
| Description of change | Treatment goal for HbA1c is <7% and |
| | rescue medication is encouraged if HbA1c is >7.5%. However, the decision to initiate |
| | rescue medication remains with the |
| | investigator and the appropriate local |
| | treatment guidelines. |
| Rationale for change | To provide clarification of treatment goal |
| | and use of rescue medication to be in line with section 4.2.1 |
| Section to be changed | 3.3 |
| Description of change | Permission to randomise more than 30 |
| | patients will only be allowed after a careful |
| | review of enrolment status, resources and |
| Dationals for shangs | data quality of the site. Site should have sufficient resources and |
| Rationale for change | data quality to allow randomisation of more |
| | than 30 patients. |
| Section to be changed | 3.3.1 |
| Description of change | Change 1: |
| | Background medication should also be stable during screening/run-phase to allow |
| | randomisation. |
| | Change 2: |
| Dationals for shangs | Deletion of sentence. Change 1: |
| Rationale for change | To clarify that background medication |
| | should also be stable during screening/run- |
| | in phase to allow randomisation. |
| | Change 2: |
| | Background medication is already |
| | highlighted in section 4.1.4. |
| Section to be changed | 3.3.2 |
| Description of change | Change 1: |

20 April 2016

Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19

**Protocol Revision 6** 


| | Order of inclusion criteria has changed, i.e. T2DM is now a specific inclusion criterion number 1. |
|---|---|
| | Change 2: (inclusion criterion 2) Inclusion of patients with background medication of - sulphonylurea + alpha-glucosidase inhibitor or - glinide + alpha-glucosidase inhibitor |
| | Change 3: (inclusion criterion 2) Documented coronary artery disease ( $\geq$ 50% luminal diameter narrowing of left main coronary artery or $\geq$ 50% in at least two major coronary arteries in angiogram). |
| | Change 4: (inclusion criterion 3) Peripheral occlusive arterial disease will include stenting as inclusion criterion. |
| | Change 5: Since blood pressure and LDL are not measured at V1a, these values should be known prior study enrolment if used for inclusion (values < 6 months old prior V1a). |
| | Change 6: (inclusion criterion 5) BMI ≤ 45 kg/m <sup>2</sup> at Visit 1b |
| | Change 7: (new inclusion criterion 7) Stable anti-diabetic background medication (unchanged daily dose) for at least 8 weeks prior V1a and without short term use of insulin. Background medication should be stable during screening/run-in phase to allow randomisation |
| | Change 8: Limitation of recruitment of patients of Category C and D. |
| Rationale for change | Change 1: To clearly identify T2DM as inclusion criterion and to be in line with CRF. |
| | Change 2: (inclusion criterion 2) Combination therapy of sulphonylurea/glinide + alpha-glucosidase |

20 April 2016


**Protocol Revision 6** 

| | inhibitor is a suitable combination therapy for the protocol target population |
|---|---|
| | Change 3: (inclusion criterion 3) To clarify that ≥ 50% luminal diameter narrowing is documented in at least two major coronary arteries. Including note for further clarification. |
| | Change 4: (inclusion criterion 3) To allow stenting cardiovascular risk |
| | Change 5: (inclusion criterion 3) To clarify current blood pressure and LDL measurements if used for inclusion. |
| | Change 6: (inclusion criterion 5) BMI will be measured at V1b |
| | Change 7: (new inclusion criterion) Medication should be stable 8 weeks prior V1a to allow enrolment) and during screening/run-in phase (to allow randomisation) |
| | Change 8: Since the cardiovascular risk is relatively lower for patients of category C and D compared to category A and B, recruitment of patients of category C will be limited to approximately 25% and recruitment of patients of category D will be limited to approximately 25% of total amount of randomised patients. This will be arranged on regional/country level. |
| Section to be changed | 3.3.3 |
| Description of change | Change 1: (exclusion criterion 2) Treatment with other diabetic drugs (as specified in inclusion criteria) prior informed consent is excluded. This included also clinical trials where these antidiabetic drugs have been provided to patients. |
| | Change 2: (exclusion criterion 3) Sibutramine and orlistat were removed as specifically named anti-obesity drugs |
| | Change 3: (exclusion criterion 7) |

Protocol Revision 6 

| | Pre-planned coronary artery revascularisation (PCI, CABG) within next 6 months after V1a or any previous PCI ≤ 6 months prior informed consent or any previous CABG < 3 months prior informed consent |
|---|---|
| | Change 4: (exclusion criterion 17) Sexual abstinence (if allowed by local authorities) and double barrier added to list of acceptable method of birth control |
| | <u>Change 5: (new exclusion criterion 19)</u> Exclusion of acute coronary syndrome ≤ 6 weeks prior to informed consent |
| | Change 6: (new exclusion criterion 20) Exclusion of stroke or TIA ≤ 3 months prior to informed consent |
| Rationale for change | Change 1: (exclusion criterion 2) To ensure other antidiabetic drugs are also excluded if prescribed in another clinical trial. |
| | Change 2: (exclusion criterion 3) To remove specific anti-obesity medication and prevent need for future revisions when available products of this class may chance. |
| | Change 3: (exclusion criterion 7) To exclude recent PCI and CABG |
| | Change 4: (exclusion criterion 17) In certain countries sexual abstinence is allowed by local authorities as acceptable method of birth control. Double barrier is an acceptable method of birth control. |
| | Change 5: (new exclusion criterion 19) To ensure that patients with acute coronary syndrome ≤ 6 weeks prior to informed consent are not included. |
| | Change 6: (new exclusion criterion 20) |

| | T d. d. d. d. d. TIA |
|---|---|
| | To ensure that patients with stroke or TIA $\leq$ |
| | 3 months prior to informed consent are not |
| | included. |
| Section to be changed | 3.3.4.1 |
| Description of change | Change 1: |
| | Updated procedures for patients who |
| | withdraw informed consent. |
| | <u>Change 2</u> : Indicating that all study |
| | procedures, e.g. lab measurements should |
| | be done in patients who discontinued study |
| | medication prematurely. |
| | Change 3: |
| | Addition of minimal requirements for |
| | patients who discontinued study treatment. |
| | patients who discontinued study treatment. |
| | Change 4: |
| | Background medication should be kept |
| | stable for the course of the trial unless |
| | medical emergencies, or other plausible |
| | reasons (e.g. hyper -or hypoglycaemia) |
| | necessitate changes at the discretion of the |
| | investigator |
| Rationale for change | Change 1: |
| _ | To clarify procedures for patients who |
| | withdraw informed consent |
| | Change 2: |
| | To clarify that study procedures should be |
| | done as much as possible in patients who |
| | discontinued study medication prematurely. |
| | p |
| | Change 3: |
| | To capture minimal data (i.e. primary |
| | endpoint events and vital status) of patients |
| | who discontinued study treatment. |
| | Change 4 |
| | • |
| Section to be changed | 1 0 |
| Section to be changed | 4.1.4 |
| Section to be changed Description of change Rationale for change | who discontinued study treatment. Change 4: To allow treatment flexibility for background medication in this long term trial, as you may expect that diabetes will progress over time. 4.1.3 Linagliptin marketed dose is 5mg Linagliptin 5mg is marketed in countries |
| Daniel dia C 1 | Change 1. |
|---|---|
| Description of change | Change 1: Background medication should be kept stable for the course of the trial unless medical emergencies, or other plausible reasons (e.g. hyper -or hypoglycaemia) necessitate changes at the discretion of the investigator. Change 2: |
| | Rephrase of uptitration. |
| | Change 3: Patients on previous glimepiride will start the randomisation phase at same glimepiride dose. |
| | Change 4: Uptitration of glimepiride becomes more flexible and will be allowed at (un) scheduled visits during maintenance phase. |
| | Change 5: During the maintenance phase it is investigator judgement to change the study and/or background medication dose. Rescue medication could also be initiated provided protocol criteria are met. |
| | Change 6: Study medication should be taken shortly before or during a meal (except on visit days) |
| | Change 7: Background and/or rescue medication will be taken as prescribed including visit days. |
| Rationale for change | Change 1: To allow treatment flexibility for background medication in this long term trial, as you may expect that diabetes will progress over time. |
| | Change 2: To clarify that during titration phase uptitration is mandatory at certain FPG levels, provided there is no risk for hypoglycaemia (investigator's judgement). |

|------|-----|----|-----|

| | Change 3: |
|---|---|
| | To clarify those patients on previous |
| | glimepiride will start study medication on same glimepiride dose. |
| | Sum gameparae acce. |
| | Change 4: |
| | To increase flexibility of study medication. |
| | Instructions for uptitration of glimepiride are indicated. |
| | are mareasea. |
| | Change 5: |
| | To clarify that it is investigator judgement |
| | to change study and/or background medication dose or to initiate rescue |
| | medication. |
| | Change 6: |
| | According to prescription guidelines glimepiride should be taken shortly before |
| | or during a meal. |
| | or during a mount |
| | Change 7: |
| | To clarify that background and/or rescue |
| | medication will be taken as usual on visit days. |
| Section to be changed | 4.1.5.2 |
| Description of change | A patient could continue with study |
| | medication after site or global unblinding. |
| Rationale for change | To clarify that patient could continue on |
| | study medication after site or global |
| Section to be changed | unblinding. 4.2.1 |
| Description of change | Change 1: |
| 1 | Alpha-glucosidase inhibitors will be |
| | allowed as rescue medication |
| | Change 2: |
| | Adding sentence regarding rescue |
| | medication |
| Rationale for change | Change 1: |
| | To increase potential rescue medication in |
| | countries where alpha-glucosidase inhibitors are prescribed. |
| | minoriors are presented. |
| | Change 2: |
| | Particular rescue medication may not be |
| | available in countries (e.g. pioglitazone). |


| Section to be changed | 4.2.2.1 |
|---|---|
| Description of change | If any restricted medication are given to the patient, the study medication <b>can</b> be discontinued temporarily, or if needed permanently. |
| Rationale for change | Discontinuation of study medication is medical judgement by investigator. To ensure this paragraph is in line with section 3.3.4.1 |
| Section to be changed | 4.2.2.2 |
| Description of change | All patients should be provided with healthy advice and relevant educational material to be used for this purpose will be supplied |
| Rationale for change | To ensure patients will receive advice and educational material regarding healthy advice. |
| Section to be changed | 5.2.1.1 |
| Description of change | Exemption of cardiovascular outcome events (heartfailure requiring hospitalisation, TIA. PCI and CABG) from expedited and unblinded SUSAR reporting. |
| Rationale for change | To avoid unblinding of these cardiovascular outcome events to maintain the integrity of the trial. |
| Section to be changed | 5.2.2.1 (hepatic events) |
| Description of change | Section has been updated regarding procedures for follow-up of lab parameters. |
| Rationale for change | To be in line with section 10.6.2. |
| Section to be changed | 5.2.2.2 |
| Description of change | Change 1: Clinically relevant abnormalities found at physical examination, vital signs or ECG that are not pre-existing prior to signing of informed consent (study inclusion) should be reported as adverse events. |
| | Change 2: Cardiovascular outcome events if they represent an SAE should be reported as SAE if occurred during screening/run-in phase. |
| | Change 3: Cardiovascular outcome events should be reported as outcome event if occurred after randomisation. |


| oc No.: c01618200-19 | Protocol |
|-----------------------|----------|
| 1 1 riai No.: 1218./4 | |

| Rationale for change | <u>Change 1</u> : To ensure that clinically relevant abnormalities will be reported as adverse |
|---|---|
| | events if not pre-existing prior signing of informed consent. |
| | <u>Change 2</u> : To ensure prior randomisation |
| | cardiovascular outcome events will be reported as SAE. |
| | Change 3: To ensure the integrity of the trial, cardiovascular outcome events should be reported as outcome event if occurred after randomisation, i.e. no unblinding will occur. |
| Section to be changed | 5.2.2.3 |
| Description of change | New paragraph regarding oncology adverse events is added |
| Rationale for change | In order to assess patients with oncology adverse events in detail, detailed information will be requested and has to be provided. |
| Section to be changed | 5.2.3.2 |
| Description of change | Change 1: |
| | Change 2: AST, ALT and Total bilirubin are combined in any lab assessment |
| Rationale for change | Change 1: |
| | Change 2: To fulfil the FDA Drug Induce Liver Injury guideline |
| Section to be changed | 5.2.5 |
| Description of change | Change 1: Section vital signs and height has been updated. Reference to section 10.3 |
| | Change 2: Weight should be measured on same type of scale |
| | <u>Change 3</u> :<br>Further instructions for use of HBGM diary. |

Boehringer Ingelheim 20 April 2016

| Rationale for change | Change 1: |
|----------------------|---------------------------------------|
| _ | To be in line with Flow Chart and to |
| | highlight section 10.3 |
| | Change 2: |
| | To allow flexibility for weight |
| | measurements. |
| | Change 3: |
| | To clarify instructions of HBGM diary |

| Page 1 | 114 | of | 17 | 3 |
|--------|-----|----|----|---|
|--------|-----|----|----|---|

| Section to be changed | 6.2.2 |
|---|---|
| Description of change | Addition of minimal requirements for patients who discontinued study treatment. |
| Rationale for change | To capture minimal data (i.e. primary endpoint events and vital status) of patients who discontinued study treatment. |
| Section to be changed | 6.2.3 |
| Description of change | Deletion of sentence regarding discontinued patients. |
| Rationale for change | Information is already indicated in section 3.3.4.1 and 6.2.2 |
| Section to be changed | 7.1 (tertiary diabetes related endpoints) |
| Description of change | Change 1: Change of endpoint: proportion of patients with moderate/severe hypoglycaemic episodes. |
| | Change 2: Change of endpoint: Proportion of patients with treatment sustainability (defined as the proportion of patients that are on study treatment at study end without rescue medication) with ≤ 2% weight gain at Final Visit (with or without rescue medication during maintenance phase) (between Visit 6 and Final Visit)) |
| | Change 3: Short term use of basal insulin- up to two weeks - (e.g. during hospitalisation) won't count as rescue medication in the definition of treatment sustainability. |
| Rationale for change | Change 1: Definitions of hypoglycaemic episodes in line with section 5.1.1. |
| | Change 2: To ensure weight endpoint will be based on population with treatment sustainability |
| | Change 3: Short term use of basal insulin is a common treatment option when dual oral therapy failed. Per definition it will be seen as (new) |

|------|-----|----|-----|
|------|-----|----|-----|

| | rescue treatment if given more than two |
|-----------------------|----------------------------------------------|
| | weeks. |
| | , |
| Section to be changed | 7.1 (other endpoints) |
| Description of change | Incidence of particular adverse events will |
| | be analysed as "other endpoint". |
| Rationale for change | To fulfil safety requirements of health |
| 8 | authorities. |
| Section to be changed | 7.3.4. |
| Description of change | Change 1: |
| Description of change | The DMC will perform formal interim |
| | analyses of the primary endpoint for non- |
| | inferiority and superiority |
| | interiority and superiority |
| | Change 2: |
| | Sentence deleted, regarding stopping rule |
| | for futility. |
| Detionals for shares | - |
| Rationale for change | Change 1: |
| | To clarify formal interim analyses by DMC. |
| | Change 2. |
| | Change 2: |
| | Stopping rules for futility are already |
| | indicated in same paragraph. |
| Section to be changed | 8.4.2 |
| Description of change | Cardiovascular outcome events should be |
| | reported as outcome event if occurred after |
| | randomisation |
| Rationale for change | To ensure the integrity of the trial. |
| Section to be changed | 9.1 |
| Description of change | References added |
| Rationale for change | References added regarding oncology |
| | adverse events and new standardised |
| | definitions for endpoint events in |
| | cardiovascular trials (October 2010) |
| Section to be changed | 10.2 (and sub-sections) |
| Description of change | Sub-sections in 10.2 are updated according |
| - compron or enunge | to new standardised definitions for endpoint |
| 1 | to non sumantibod definitions for enapoint |


| | <del></del> |
|-------------------------|--------------------------------------------|
| | events in cardiovascular trials (October |
| | 2010) |
| D 4: 1 C 1 | Ti 1- 41 - 1-6:-:4: 641 - |
| Rationale for change | To provide the definitions of the |
| | cardiovascular outcome events based on the |
| | current "Standardised Definitions for |
| | endpoint events in cardiovascular trials, |
| | Final recommendations (2010). |
| Section to be changed | 10.3 |
| Description of change | Clarification on blood pressure |
| | measurements |
| Rationale for change | Clarification on blood pressure |
| | measurements |
| Section to be changed | Several sections throughout the protocol |
| Description/rational of | Typo's, minor errors has been corrected |
| change | throughout the protocol |
| Section to be changed | 10.6.3 |
| Description of change | No check-list will be provided in the ISF |
| _ | supporting the collecting of further |
| | information. |
| Rationale for change | Patients who discontinued study medication |
| ge | should be followed as much as possible. |
| <u> </u> | bilders of folia The do filed do possible. |

20 April 2016

Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19

**Protocol Revision 6** 


| Number of CTP modification | 2 |
|---|---|
| Date of CTP modification | 6 March 2012 |
| EudraCT number | 2009-013157-15 |
| BI Trial number | 1218.74 |
| BI Investigational Product(s) | Linaglitin |
| Title of protocol | A multicentre, international, randomised, |
| Title of protocor | parallel group, double blind study to |
| | evaluate Cardiovascular safety of linagliptin |
| | versus glimepiride in patients with type 2 |
| | diabetes mellitus at high cardiovascular |
| | risk. The CAROLINA Trial. |
| To be implemented only | |
| after approval of the | |
| IRB/IEC/Competent | |
| Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Section to be changed | Protocol synopsis (objectives) |
| Description of change | Change 1: |
| | Exclusion of silent MI from primary |
| | endpoint |
| | Change 2: |
| | Change 2: Correction of confidence interval |
| Dationals for shange | Change 1: |
| Rationale for change | Silent MI will be reported as tertiary |
| | cardiovascular endpoint |
| | cardiovasculai chaponit |
| | Change 2: |
| | Confidence interval is determined based on |
| | the alpha from the alpha-spending function. |
| Section to be changed | · |
| ~ COULDIE OF NO CHIMILEUM | Protocol synopsis (criteria for safety) |
| | Protocol synopsis (criteria for safety) Change 1: |
| Description of change | Change 1: |
| | Change 1: Summarization of non-fatal and fatal MI, as well as non-fatal and fatal stroke for |
| | Change 1: Summarization of non-fatal and fatal MI, as well as non-fatal and fatal stroke for evaluation of time to and occurrence of |
| | Change 1: Summarization of non-fatal and fatal MI, as well as non-fatal and fatal stroke for |
| | Change 1: Summarization of non-fatal and fatal MI, as well as non-fatal and fatal stroke for evaluation of time to and occurrence of |

|-------|-----|----|-----|
| 1 420 | 110 | UI | 1,0 |

| | Deletion of stable angina pectoris as study |
|-----------------------|-------------------------------------------------|
| | endpoint. |
| Rationale for change | Change 1: |
| Rationale for change | To allow for an analysis of single |
| | 1 1 |
| | components with inclusion of death |
| | resulting from such a component. |
| | Change 2: |
| | Stable angina pectoris will not be |
| | adjudicated as tertiary cardiovascular |
| | endpoint. |
| Section to be changed | Protocol synopsis (inclusion criteria) |
| Description of change | Change 1: |
| Description of change | Addition of the statement in the inclusion |
| | criteria that anti-diabetic treatment naïve |
| | patients are only eligible for study |
| | enrolment if they are intolerant or contra- |
| | indicated to first line anti-diabetic |
| | treatment. |
| | Change 2: |
| | In consultation with the Steering |
| | Committee, enrolment of patients currently |
| | 1 1 |
| D (* 1 C 1 | at least on SU or glinide may be limited. |
| Rationale for change | Change 1: |
| | To clarify this criterion for naïve patients in |
| | the inclusion criteria as stated in protocol |
| | section 3.3.1. |
| | Change 2: |
| | To ensure an early/moderate disease |
| | population with short to moderate diabetes |
| | duration. To allow assessment of the CV |
| | safety profile of linagliptin versus |
| | glimepiride. |
| Section to be changed | Protocol synopsis (main criteria for |
| | exclusion) |
| Description of change | Change 1: |
| 1 | The wording any history and/or current |
| | treatment with other antidiabetic drugs |
| | added to inclusion criteria |
| | Change 2: |
| | Current treatment with systemic |
| | corticosteroids will exclude a patient of |
| | study enrolment |
| | Change 2: |
| | Change 3: |


| | T ', C1' '11 , , |
|-----------------------|------------------------------------------------|
| | Inappropriateness of glimepiride treatment |
| | for other issues (e.g. allergy) according to |
| | local prescribing information. |
| Rationale for change | Change 1: |
| Rationale for change | To clarify that any history and/or current |
| | treatment of anti-diabetic drugs as specified |
| | in the inclusion criteria will exclude a |
| | patient from study enrolment |
| | patient from study emorment |
| | Change 2: |
| | Clinical relevant drug-drug interaction of |
| | the study medication is limited to |
| | corticosteroids |
| | <u>Change 3:</u> |
| | To avoid patients being enrolled with |
| | allergies to the SU class |
| Section to be changed | Flowchart |
| Description of change | <u>Change 1:</u> |
| | Addition of maximal/minimal days from |
| | randomisation for screening to be |
| | performed. |
| | Change 2: |
| D 4: 1 6 1 | Visit time window of visit 6 is +/- 7 days |
| Rationale for change | Change 1: |
| | To clarify that maximal 42 days and |
| | minimal 15 days should be between |
| | screening and randomisation |
| | Change 2: |
| | Since patient received at visit 5 medication |
| | up to maximal 5 weeks, the time window |
| | for visit 6 is limited to +/- 1 week. |
| Section to be changed | 1.1 (medical background) |
| Description of change | Change of reference number |
| Rationale for change | Incorrect reference number |
| Section to be changed | 1.2 (drug profile) |
| Description of change | Updated drug profile |
| Rationale for change | To add new clinical trial data |
| Section to be changed | 2.1 (rationale for performing the trial) |
| Description of change | Addition of the statement that anti-diabetic |
| | treatment naïve patients are only eligible for |
| | study enrolment if they are intolerant or |
| | contra-indicated to first line anti-diabetic |
| | treatment. |

| Rationale for change | To clarify this criterion for naïve patients as |
|-----------------------|-------------------------------------------------|
| | stated in protocol section 3.3.1. |
| Section to be changed | 2.2 (trial objectives) |
| Description of change | Correction of confidence interval |
| Rationale for change | Confidence interval is determined based on |
| _ | the alpha from the alpha-spending function. |
| Section to be changed | 2.3 (benefit – Risk assessment) |
| Description of change | Change 1: |
| | Add description of alpha-glucosidase |
| | inhibitor as possible rescue medication (as |
| | indicated in section 4.2.1) |
| | Change 2: |
| | Updated list of anti-diabetic drugs (given as |
| | study medication or allowed as rescue |
| | medication) which are not approved for use |
| | in pregnancy. |
| Rationale for change | Change 1: |
| | To provide background of alpha- |
| | glucosidase inhibitor as possible rescue |
| | medication |
| | Change 2: |
| | To update list of antidiabetic drugs (given |
| | as study medication or allowed as rescue |
| | medication) which are not approved for use |
| | in pregnancy. |
| Section to be changed | 3.3 (selection of trial population) |
| Description of change | Change 1: |
| Description of change | Change 1. |
| | Change 2: |
| | Addition of procedures for re-screening and |
| Detionals for the | re-testing |
| Rationale for change | Change 1: |
| | Change 2. |
| | Change 2: |

|------|-----|--------|

| | Procedures for re-screening and re-testing |
|---|---|
| | are permitted under certain circumstances |
| Section to be changed | 3.3.1 (main diagnosis for study entry) |
| Description of change | Change 1: |
| Description of change | Change of wording "therapy" into "anti- |
| | diabetic treatment" |
| | Change 2: |
| | Adding of wording "intolerances" |
| | Change 3: |
| | Adding wording "whereas if medications |
| | such as metformin and alpha-glucosidase |
| | inhibitor are being used, these should be |
| | continued". |
| Rationale for change | Change 1: |
| | To clarify that treatment naïve T2DM |
| | patients should be offered first line anti- |
| | diabetic treatment before patients are |
| | eligible for study inclusion |
| | Change 2. |
| | Change 2: |
| | To clarify that anti-diabetic treatment naïve |
| | patients are only eligible for study enrolment if they are intolerant or contra- |
| | indicated to first line anti-diabetic |
| | treatment. |
| | treatment. |
| | Change 3: |
| | To clarify that background anti-diabetic |
| | medication such as metformin and alpha- |
| | glucosidase inhibitor should be continued at |
| | Visit 2. |
| Section to be changed | 3.3.2 (inclusion criteria) |
| <b>Description of change</b> | Change 1: |
| | Addition of the statement in the inclusion |
| | criteria that anti-diabetic treatment naïve |
| | patients are only eligible for study |
| | enrolment if they are intolerant or contra- |
| | indicated to first line anti-diabetic |
| | treatment. |
| | Change 2: |
| | Change 2: |
| | In consultation with the Steering |
| | Committee, enrolment of patients currently |
| | at least on SU or glinide may be limited. |
| Rationale for change | Change 1: |

|------|-----|--------|

| | To clarify this criterion for naïve patients in |
|-----------------------|-------------------------------------------------|
| | the inclusion criteria as stated in protocol |
| | section 3.3.1. |
| | Change 2: |
| | To ensure an early/moderate disease |
| | population with short to moderate diabetes |
| | duration. To allow assessment of the CV |
| | safety profile of linagliptin versus |
| | glimepiride. |
| Section to be changed | 3.3.3 (exclusion criteria) |
| Description of change | Change 1: |
| Description of change | The wording any history and/or current |
| | treatment with other antidiabetic drugs |
| | added to exclusion criteria |
| | added to exclusion effective |
| | Change 2: |
| | Adding wording "any" insulin. |
| | rading wording uny mounn. |
| | Change 3: |
| | Clinical relevant drug-drug interaction of |
| | the study medication is limited to |
| | corticosteroids |
| | Corticosteroids |
| | Change 4: |
| | Add wording "SU class "to exclusion |
| | criterion 8. |
| Rationale for change | Change 1: |
| Turionale for enange | To clarify that any history and/or current |
| | treatment of anti-diabetic drugs as specified |
| | in the exclusion criteria will exclude a |
| | patient from study enrolment |
| | r |
| | Change 2: |
| | To clarify that short term us of any insulin |
| | (up to two weeks) is allowed. |
| | (CF to the heart) is uno hear. |
| | Change 3: |
| | Clinical relevant drug-drug interaction of |
| | the study medication is limited to |
| | corticosteroids |
| | Change 4: |
| | To clarify that also known allergy to SU |
| | treatment will exclude the patient for study |
| | enrolment. |
| Section to be changed | 3.3.4 (removal of patients from therapy |
| | or assessments) |
| | 1 |


| D | C1 1 |
|---|---|
| Description of change | Change 1: |
| | Addition of the definition of Lost-To- |
| | Follow-Up |
| | Change 2: |
| | Study medication can be discontinued |
| | temporarily. Investigators are encouraged to |
| | re-administer study medication to a |
| | randomised patient if there are no further |
| | safety concerns. |
| Rationale for change | Change 1: |
| | Clarification which patients are considered |
| | Lost-To-Follow-Up |
| | Lost to rollow op |
| | Change 2: |
| | Change 2: |
| | Since this is an outcome study, the primary |
| | analysis will be performed based on all |
| | randomised patients who were treated with |
| | at least one dose of study drug. Therefore |
| | investigators are encouraged to re- |
| | administer study medication to a |
| | randomised patient if there are no further |
| | safety concerns. |
| Section to be changed | 4.1.4 (drug assignment and |
| | administration of doses for each patient) |
| Section to be changed Description of change | |
| | administration of doses for each patient) Change 1: |
| | administration of doses for each patient) Change 1: The average HBGM value of previous |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study medication has been further |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study medication has been further clarified/described |
| | administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study medication has been further |
| | Administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study medication has been further clarified/described Change 3: |
| | Administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study medication has been further clarified/described Change 3: To add wording that "The above principle |
| | Administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study medication has been further clarified/described Change 3: To add wording that "The above principle also applies for patients being included on a |
| | Administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study medication has been further clarified/described Change 3: To add wording that "The above principle |
| | Administration of doses for each patient) Change 1: The average HBGM value of previous recent fasting HBGM measurements prior to the day of visit (from the patient's HBGM diary) could also be used to guide uptitration at the discretion of the investigator, if there is a meaningful discrepancy between the single fasted HBGM value at the day of the visit in the clinic and this average HBGM value. Change 2: The titration process of the study medication has been further clarified/described Change 3: To add wording that "The above principle also applies for patients being included on a |

Boehringer Ingelheim 20 April 2016

| | To allow to use additional HBGM values if there is a meaningful discrepancy between the HBGM value at the day of visit in the clinic and the HBGM values in patient's HBGM diary <u>Change 2:</u> To clarify the titration phase in more detail to ensure titration process will be followed. |
|---|---|
| | Change 3: |
| | To clarify that the principle also applies for |
| | patients being included on a background of |
| Section to be shanged | alpha-glucosidase inhibitor. |
| Section to be changed | 4.2.1 (rescue medication, emergency procedures, and additional treatment(s)) |
| Description of change | Change 1: |
| r r | Short-acting insulin may be given as rescue |
| | medication for up to two weeks in |
| | combination with the study medication (e.g. |
| | during hospitalisation). |
| | Change 2: |
| | The results for fasting plasma glucose to |
| | initiate rescue medication could be obtained |
| | from the HBGM device. |
| | Change 3: |
| | Add alpha-glucosidase inhibitor |
| | Change 4: |
| | Adding wording "the protocol defined rescue therapy" |
| Rationale for change | Change 1: |
| g | In practice short-acting insulin is given as |
| | rescue medication to T2DM patients (e.g. |
| | during hospitalization). Such treatment may |
| | be given in combination with the study |
| | medication for up to two weeks. |
| | Change 2: |
| | To clarify that the results for fasting plasma |
| | glucose to initiate rescue medication could |
| | be obtained from the HBGM device. |
| | Change 3: |
| | To be consistent since alpha-glucosidase |
| | inhibitor could be described as anti-diabetic |
| | background medication |


| Section to be changed Description of change G S Rationale for change T C S T C S T C S T C S T T T T T T T T T T T T | Change 4: To clarify that there is specific protocol defined rescue medication 1.2.2.1 (restrictions) Change 1: Short acting insulin may be given as rescue medication up to two weeks (e.g. during hospitalisation) |
|---|---|
| Section to be changed Description of change G S Rationale for change T C S T C S T C S T C S T T T T T T T T T T T T | Fo clarify that there is specific protocol defined rescue medication 1.2.2.1 (restrictions) Change 1: Short acting insulin may be given as rescue medication up to two weeks (e.g. during |
| Section to be changed Description of change G S Rationale for change T C S T C S T C S T C S T T T T T T T T T T T T | Fo clarify that there is specific protocol defined rescue medication 1.2.2.1 (restrictions) Change 1: Short acting insulin may be given as rescue medication up to two weeks (e.g. during |
| Section to be changed Description of change G G G G G G G G G G G G G | lefined rescue medication 1.2.2.1 (restrictions) Change 1: Short acting insulin may be given as rescue medication up to two weeks (e.g. during |
| Section to be changed Description of change G I Rationale for change 4 4 4 C I C I C I C I C I C I C I I | Change 1: Short acting insulin may be given as rescue medication up to two weeks (e.g. during |
| Description of change G S T | Change 1: Short acting insulin may be given as rescue nedication up to two weeks (e.g. during |
| Rationale for change | Short acting insulin may be given as rescue medication up to two weeks (e.g. during |
| Rationale for change | nedication up to two weeks (e.g. during |
| Rationale for change | , , , |
| Rationale for change | , |
| Rationale for change I | |
| Rationale for change I | Change 2: |
| Rationale for change I | f any restricted treatments or any other |
| Rationale for change CI | concomitant drugs interfering with the |
| Rationale for change G | tudy medication, the study medication dose |
| I I | ean be reduced. |
| r | Change 1: |
| | n practice short-acting insulin is given as |
| | escue medication to T2DM patients (e.g. |
| | during hospitalization). Such treatment may |
| | be given in combination with the study |
| r | nedication for up to two weeks. |
| | Change 2: |
| | To clarify that study medication dose can be |
| | changed if concomitant drugs interfere with |
| | he study medication. |
| | 5.1.1 (endpoint(s) of efficay) |
| | Exclusion of silent MI from primary |
| | endpoint |
| | To clarify that silent MI will be reported as |
| | ertiary cardiovascular endpoint |
| Section to be changed 5 | 5.2.1.1 (reporting waver for |
| | eardiovascular events) |
| | Silent MI is added to list of cardiovascular |
| | outcome events |
| | To avoid unblinding of patient with silent |
| | MI to ensure the integrity of the trial. |
| | (1) ( ) |
| 8 - | 5.2.2 (assessment of adverse events) |
| | Change 1: |
| | Change 1:<br>Change of adverse event reporting in case |
| | Change 1: Change of adverse event reporting in case of worsening of the underlying disease or |
| | Change 1:<br>Change of adverse event reporting in case |
| | Change 1: Change of adverse event reporting in case of worsening of the underlying disease or other pre-existing conditions |
| | Change 1: Change of adverse event reporting in case of worsening of the underlying disease or other pre-existing conditions Change 2: |
| e | Change 1: Change of adverse event reporting in case of worsening of the underlying disease or other pre-existing conditions |
| | Change 1: Change of adverse event reporting in case of worsening of the underlying disease or other pre-existing conditions Change 2: |

| | Change 3: |
|-----------------------|-------------------------------------------------|
| | Updated reporting of clinical evaluation of |
| | hepatic injury |
| Rationale for change | <u>Change 1:</u> |
| | To clarify the criteria for (S)AE reporting. |
| | Change 2: |
| | To expand the criteria for (S)AE reporting. |
| | Change 3: |
| | To incorporate clinical evaluation of hepatic |
| | injury according to BI standards |
| Section to be changed | 5.2.2.2 (adverse event and serious adverse |
| Section to be changed | event reporting) |
| Description of abanga | • |
| Description of change | Change 1: The change and 20 days often |
| | The observational phase ends 30 days after |
| | the patient has completed the study. |
| | Change 2: |
| | The following paragraph has been added to |
| | the protocol: "BI has established a list of |
| | AEs which are defined to be always serious. |
| | In order to support the investigator with the |
| | identification of these "always serious |
| | adverse events", if a non serious AE is |
| | identified to be serious per BI definition, a |
| | query will be raised. The investigator must |
| | verify the description and seriousness of the |
| | event. If the event description is correct, the |
| | item "serious" needs to be ticked and an |
| | SAE has to be reported in expedited fashion |
| | following the same procedure as above. |
| | The list of these adverse events can be |
| | found via the RDC-system." |
| Rationale for change | <u>Change 1:</u> |
| | To clarify that the he observational phase |
| | ends 30 days after the patient has completed |
| | the study (with or without study |
| | medication). |
| | Change 2: |
| | To expand the definition of SAEs. |
| Section to be changed | 5.2.5 (assessment of other safety |
| | parameters) |
| Description of change | To add wording "something containing" |
| Rationale for change | For further clarification |
| Tanonaic IVI Change | 1 of farmer claimeation |
| į l | |


| Description of change | |
|---|---|
| D ( 1 C 1 | <del></del> |
| Rationale for change | |
| | <del></del> |
| Section to be changed | 7.1 (objectives) Addition of "*100" to reflect percentage |
| Description of change Rationale for change | Typo correction |
| Section to be changed | 7.1 (primary endpoint) |
| Description of change | Exclusion of silent MI from primary |
| Description of change | endpoint |
| Rationale for change | Silent MI will be reported as tertiary |
| | cardiovascular endpoint. |
| Section to be changed | 7.1 (key secondary endpoints) |
| Description of change | Change 1: |
| | Definition of rescue medication for |
| | evaluation of key secondary endpoints was |
| | added. |
| | Charras 2: |
| | Change 2: Both short acting and basal insulin may be |
| | used as rescue medication. Short acting |
| | insulin only up to two weeks (e.g. during |
| | hospitalisation). Therefore the word "basal" |
| | was deleted. |
| Rationale for change | Change 1: |
| | To clarify definition of rescue therapy for |
| | evaluation of key secondary endpoints. |
| | Change 2: |
| | Short-acting insulin may also be used as |
| | rescue medication up to two weeks. Use of insulin up to two weeks will not count as |
| | rescue medication in the definition of |
| | treatment sustainability. |
| Section to be changed | 7.1 (secondary cardiovascular endpoints) |
| Description of change | Change 1: |
| | Replace treated patients by patients in the |
| | full analysis set. |
| | Change 2: |
| | Exclusion of silent MI from primary |
| Dational for a | endpoint Change 1: |
| Rationale for change | Change 1: |


| | According to Section 7.3 the primary |
|-----------------------|-----------------------------------------------|
| | analysis is performed on the patients in the |
| | FAS. |
| | Change 2: |
| | Silent MI will be reported as tertiary |
| | cardiovascular endpoint. |
| Section to be changed | 7.1 (tertiary cardiovascular endpoints) |
| Description of change | Change 1: |
| Description of change | Summarization of non-fatal and fatal MI, as |
| | well as non-fatal and fatal stroke for |
| | evaluation of time to and occurrence of |
| | tertiary cardiovascular endpoints. |
| | Change 2: |
| | Refine wording of tertiary cardiovascular |
| | endpoint. |
| | Cl 2 |
| | Change 3: |
| | Addition of silent MI as tertiary |
| | cardiovascular endpoint. |
| Rationale for change | Change 1: |
| | To allow for an analysis of single |
| | components with inclusion of death |
| | resulting from such a component. |
| | Change 2: |
| | Improve wording |
| | Change 3: |
| | To clarify that silent MI will be analysed as |
| | tertiary cardiovascular endpoint. |
| Section to be changed | 7.1 (secondary diabetes related |
| | endpoints) |
| Description of change | Addition of any transitions in albuminuria |
| | classes and change from baseline in |
| | albuminuria as secondary diabetes related |
| | endpoints. |
| Rationale for change | Albuminuria and change of albuminuria are |
| 8. | important diabetes related endpoints, which |
| | results may be different between the two |
| | treatment arms. These endpoints are added |
| | to allow any publication of the results. |
| Section to be shanged | |
| Section to be changed | 7.1 (tertiary diabetes related endpoints) |
| Description of change | Change 1: |
| | Addition of time to rescue medication |
| | intake as tertiary diabetes related endpoint. |


| | Change 2: Addition of proportion of patients with rescue therapy intake as tertiary diabetes related endpoint. |
|---|---|
| | Change 3: Definition of rescue medication for evaluation of tertiary endpoints was added. |
| | Change 4: Deletion of stable angina pectoris as study endpoint. |
| Rationale for change | <u>Change 1:</u><br>Definition of new endpoints |
| | Change 2: Definition of new endpoints |
| | Change 3: To clarify definition of rescue therapy for evaluation of tertiary diabetes related endpoints. |
| | Change 4: Stable angina pectoris will not be adjudicated as tertiary cardiovascular endpoint. |
| Section to be changed | 7.1 (other endpoints) |
| Description of change | Change 1: Add proportion of patients with hypoglycaemia and time to first hypoglycaemia as other endpoint. |
| | Change 2: Delete all-cause mortality from other endpoints. |
| Rationale for change | <u>Change 1:</u> Definition of new endpoints |
| | Change 2: All-cause mortality is already included in tertiary cardiovascular endpoints. |
| Section to be changed | 7.2 (null and alternative hypotheses) |
| Description of change | Adopt hypotheses for key secondary endpoints. |

|------|-----|----|-----|

| Rationale for change | As Fisher's exact test will be replaced by Chi-Square test, the two-sided p-value will be reported and hence hypotheses needed to be changed. |
|---|---|
| Section to be changed | 7.3 (planned analyses) |
| Description of change | Change 1: Definition of severe violation of treatment compliance refined. Change 2: The definition of the on-treatment set was |
| | refined to be more precise. |
| Rationale for change | Change 1: Refine definition of violation of compliance |
| | Change 2: Clarify the definition of the on-treatment set in detail. |
| Section to be changed | 7.3.1 (primary analyses) |
| Description of change Rationale for change | Change 1: Addition of "*100" to reflect percentage Change 2: Change of the test for evaluation of key secondary endpoints to Chi-Square test, on the same significance level (2*α <sub>i</sub> )*100% as the primary endpoint. Change 1: Typo correction. |
| | Change 2: Use of Chi-Square test instead of Fisher's exact test as this test is more powerful. Use of two-sided p-values. |
| Section to be changed | 7.3.2 (secondary analyses) |
| Description of change | Change 1: For all cardiovascular endpoints that include occurrence of an event, Chi-Square test is used to compare the two treatment groups. |
| | Change 2: A logistic regression with factor treatment is performed for cardiovascular endpoints. |

| | Change 3: There will not be any one-sided tests (test for superiority of linagliptin versus glimepiride, alpha= 0.025) be performed for diabetes related endpoints. Change 4: For continuous secondary diabetes related endpoints with several on-treatment measurements change from baseline will be evaluated with a restricted maximum likelihood (REML) based mixed model repeated measures (MMRM) approach. For those continuous secondary diabetes related endpoints with only one measurement on treatment an analysis of covariance (ANCOVA) model with the factor treatment and the baseline value of the respective variable as covariate will be performed. Change 5: For qualitative secondary diabetes related endpoints, Chi-Square test is used to compare the two treatment groups. |
|---|---|
| Rationale for change | Change 1: Use of Chi-Square test instead of Fisher's exact test as this test is more powerful. Change 2: The logistic regression will be performed |
| | additionally to report odds ratios. Change 3: In order to provide a consistent picture, all binary and continuous diabetes related endpoints will be investigated in the same way, respectively. Change 4: The MMRM approach will be performed to allow dealing with missing values and to |
| | account for correlations between repeated measurements. Change 5: |

| | Use of Chi-Square test instead of Fisher's |
|---|---|
| | exact test as this test is more powerful. |
| Section to be changed | 7.3.4 (interim analyses) |
| <b>Description of change</b> | Deleted filing of DMC charter in ISF. |
| Rationale for change | The DMC charter will not be filed in the ISF. |
| Section to be changed | 7.4 (handling of missing data) |
| Description of change | Change 1: The REML based MMRM analysis will handle missing data for continuous diabetes related endpoints. |
| | Change 2: The last observation carried forward (LOCF) approach will be performed in a sensitivity analysis on diabetes related endpoints. |
| Rationale for change | Change 1: This analysis will deal with missing values. |
| | Change 2: As the MMRM approach will be used to deal with missing observations of continuous diabetes related endpoints, LOCF will be performed in a sensitivity analysis. |
| Section to be changed | 8 and 8.1 (study approval, patient information, and informed consent) |
| Description of change | Additional wording/paragraph for Japan |
| Rationale for change | To fulfil Japanese requirements |
| Section to be changed | 8.2 (data quality assurance) |
| Description of change | Additional paragraph regarding data quality assurance |
| Rationale for change | To clarify data quality assurance |
| Section to be changed | 8.4.1 (listedness and expedited reporting of adverse events) |
| Description of change | Change of required SPC references |
| Rationale for change | Unique reference documents for metformin and pioglitazone are no longer required, since rescue medication is not pre-specified. Per protocol there are several options for rescue medication (investigator's judgement). |

| Section to be changed | 8.7 (protocol violations) |
|---|---|
| Description of change | Addition of paragraph regarding reporting of protocol violations |
| Rationale for change | To clarify requirement of reporting of protocol violations |
| Section to be changed | 9.1 (published references) |
| Description of change | Deletion of reference R11-2713 |
| Rationale for change | Reference R11-2713 is not needed anymore. |
| Section to be changed | 10.2 (definitions of endpoint events) |
| Description of change | Definitions of the adjudicated endpoints events and the principles of standardised data collection in the centralised CEC adjudication process are outlined in the current CEC Charter and process guideline. The endpoint definitions are deleted from the protocol. |
| Rationale for change | To reflect that the CEC charter will be maintained throughout the course of current definitions for cardiovascular endpoints. |
| Section to be changed | 10.3 (blood pressure measurement procedure and treatment recommendations) |
| Description of change | Addition of further guidance of blood pressure measurements |
| Rationale for change | To clarify blood pressure measurements |
| Section to be changed | Section 10.6 (clinical evaluation of liver injury) |
| Description of change | Updated paragraphs of clinical evaluation of liver injury |
| Rationale for change | To incorporate clinical evaluation of liver injury according to BI standards |

| Number of CTP modification | 3 |
|---|---|
| Date of CTP modification | 1 August 2012 |
| EudraCT number | 2009-013157-15 |
| BI Trial number | 1218.74 |
| BI Investigational Product(s) | Linagliptin |
| Title of protocol | A multicentre, international, randomised, |
| | parallel group, double blind study to |
| | evaluate Cardiovascular safety of linagliptin |
| | versus glimepiride in patients with type 2 |

20 April 2016

Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19

**Protocol Revision 6** 


| | diabetes mellitus at high cardiovascular risk. The CAROLINA Trial. |
|---|---|
| | The CAROLINA That. |
| To be implemented only | |
| after approval of the | |
| IRB/IEC/Competent | |
| Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for approval | |
| арргочаг | |
| Section to be changed | Title page |
| Description of change | Trial Clinical Monitor name and address |
| Description of enange | details updated. |
| Rationale for change | New TCM assigned and address change. |
| Section to be changed | Protocol synopsis (Objectives) |
| Description of change | Inclusion of the fifth test within hierarchical |
| | testing procedure. |
| Rationale for change | As the classical MACE endpoint will be |
| g- | introduced as first key secondary endpoint, |
| | the testing hierarchy will include 5 |
| | hypothesis tests. |
| Section to be changed | Protocol synopsis (Methodology) |
| Description of change | Safety was crossed out as the study's focus |
| | lies on efficacy and safety. |
| Rationale for change | For clarification. |
| Section to be changed | Protocol synopsis (No. of patients) |
| Description of change | "At least" was changed into "An estimated |
| D.C. L.C. L | number of". |
| Rationale for change | To clarify that the study is event driven and |
| | that the required number of patients is an estimation. |
| Section to be abanged | Protocol synopsis (inclusion criteria) |
| Section to be changed Description of change | Change 1: |
| Description of change | |
| | - Myocardial infarction (≥ 6 weeks prior |
| | to |
| | informed consent) |
| | - Percutaneous Coronary Intervention |
| | (PCI) ≥ 6 weeks prior informed consent |
| | - Coronary Artery By-pass Grafting (CABG) ≥ 4 years prior to informed |

| | consent or with recurrent angina pectoris following surgery |
|---|---|
| | - Ischemic or hemorrhagic stroke (≥ 3 months prior to informed consent) |
| | Was changed to: |
| | - Myocardial infarction (> 6 weeks prior to informed consent) |
| | - Percutaneous Coronary Intervention (PCI) > 6 weeks prior informed consent |
| | - Coronary Artery By-pass Grafting (CABG) > 4 years prior to informed consent or with recurrent angina pectoris following surgery |
| | - Ischemic or hemorrhagic stroke (> 3 months prior to informed consent). |
| | Change 2: |
| | Treatment compliance requirement in the placebo-run was added. |
| Rationale for change | To be consistent with section 3.3.2 inclusion |
| | criteria. |
| Section to be changed | Protocol synopsis (criteria for exclusion) |
| Description of change | Change 1: Duration of short term insulin (up to two weeks) is allowed, if taken at least 8 weeks prior informed consent |
| | was changed into: |
| | Duration of short term insulin (up to two consecutive weeks) is allowed, if taken at least 8 weeks prior informed consent. |
| | Change 2: All exclusion criteria have been added. |
| Rationale for change | <u>Change 1:</u> For clarification and |
| | Change 2: |
| | to be consistent with section 3.3.3 exclusion |
| | criteria. |
| Section to be changed | Protocol synopsis (duration of treatment) |
| Description of change | 2 to 4 weeks placebo run-in phase followed<br>by up to 400 weeks treatment + 1 week |
| | follow-up after study drug termination. |


| | Observational study duration is up to 30 days after date of patients Final Visit. |
|---|---|
| | Was changed into: |
| | 2 up to 4 weeks placebo run-in phase |
| | followed by up to an estimated 400 weeks |
| | treatment period and 1 week follow-up after |
| | study drug termination. Observational study |
| | duration is up to 30 days after date of |
| | patients Final Visit. |
| Rationale for change | To clarify duration of treatment. |
| Section to be changed | Protocol synopsis (Criteria for efficacy) |
| Description of change | Inclusion of classical MACE endpoint as first key secondary endpoint and shift of previous first and second key secondary endpoints to second and third position. |
| Rationale for change | This endpoint was defined as first key secondary endpoint. |
| Section to be changed | Protocol synopsis (Criteria for safety) |
| Description of change | Change 1: |
| Description of enange | non- fatal MI, non- fatal stroke, |
| | non- ratar ivii, non- ratar stroke, |
| | Was shapped into |
| | Was changed into: |
| | (non)- fatal MI, (non)- fatal stroke, |
| | Change 2: |
| | Silent myocardial infarction added as |
| | criteria for safety; |
| | Change 3: |
| | Reference to section 5.2 added. |
| Rationale for change | To be consistent with section 5.2.1 |
| | endpoints and tertiary cardiovascular |
| | endpoints as described in section 7.1 |
| Section to be changed | Protocol synopsis (Statistical methods) |
| Description of change | Inclusion of analysis methods for key |
| | secondary endpoints. |
| Rationale for change | According to Annotated clinical trial |
| | protocol instructions the model used for the |
| | analysis of key secondary endpoints should |
| | be mentioned. |
| Section to be changed | Flow chart |
| Description of change | |
| | l l |

## Change 1: Maximum number of days from screening (V1a) to randomisation changed from -42 into -35; Change 2: demographics obtained at Visits 1a and 1b, footnote added that the race of the patient will be collected; Change 3: additional footnotes added, re-ordered or revised; Change 4: added that placebo run-in medication will be dispensed by the IXR system; Change 5: Change 6: Change 7: additional laboratory parameters added to footnote h; Change 8: added that the MDRD considers race as an adjustment factor; Change 9: Change 10:


| | Change 11. |
|---|---|
| | Change 11: clarification of end of trial activities and guidance on re-institution of glimepiride/glimepiride placebo added. |
| Rationale for change | Changa 1: |
| Kationale for change | Change 1: To clarify maximum number of days between screening and randomisation; |
| | CI 2 |
| | Change 2: to clarify that demographic data is obtained at |
| | Visit 1a and Visit 1b and that race will be captured in the eCRF, because T2DM treatment |
| | results maybe race sensitive. Furthermore, the |
| | renal function will be assessed using the MDRD |
| | formula. This formula considers the race as |
| | an |
| | adjustment factor, therefore, the race must be |
| | known for accurate estimation; |
| | Change 3: |
| | to adapt the footnotes to the changes in the flowchart; |
| | Change 4: |
| | to clarify that placebo run-in medication is dispensed by IXRS; |
| | <u>Change 5:</u> |
| | Change 6: |
| | Change 7: to clarify obtained laboratory parameters at Visit 1a; Change 8: |


| | to state that MDRD formula considers race as an adjustment factor; Change 9: to clarify that the number of to be obtained questionnaires is an approximation; Change 10: Change 11: to clarify end of trial activities and to add guidance on re-institution of trial medication. |
|---|---|
| Section to be changed | Abbreviations |
| Description of change | Several abbreviations added. |
| Rationale for change | To list all abbreviations used in the protocol. |
| Section to be changed | 2.2 Trial Objectives |
| Description of change | Inclusion of classical MACE endpoint as first key secondary endpoint. Inclusion of the fifth test within hierarchical testing procedure. |
| Rationale for change | As the classical MACE endpoint will be introduced as first key secondary endpoint, the testing hierarchy will include 5 hypothesis tests. |
| Section to be changed | 3.1 Overall trial design and trial |
| | population |
| Description of change | Change 1: The first paragraph was aligned with the methodology section in the protocol synopsis; |
| | Change 2: the minimum number of patients of 6000 was changed into an estimated number of 6000 patients, in addition it was added that the 400 weeks treatment duration is an estimated treatment duration; Change 3: |

**Protocol Revision 6** 

| | treatment compliance criterion was added to the definition of successfully completed at least two weeks of the placebo run-in; Change 4: added that SU/glinide should not be taken in the morning of Visit 2. Change 5: |
|---|---|
| | the end of trial activities and requirements were clarified and |
| | Change 6: trial stop procedures, including timeframe to stop the trial and to perform last patient visits clarified. |
| Rationale for change | Change 1: To be consistent with the methodology section in the synopsis; |
| | Change 2: to clarify that the study is event driven and that the required number of patients and the treatment duration is an estimation; |
| | Change 3: to clarify that the treatment compliance criterion is a placebo-run requirement; |
| | Change 4: to clarify that no double doses should be taken at Visit 2; |
| | Change 5: to clarify end of trial activities and |
| | Change 6: to clarify trial stop procedures. |
| Section to be changed | 3.1.1 Administrative structure of the trial |
| Description of change | Pancreatic adjudication was added. |
| Rationale for change | To set-up an adjudication committee for pancreatic events. |

| Section to be changed | 3.2 Discussion of trial design, including the choice of control group |
|---|---|
| Description of change | The treatment duration was clarified e.g. by adding that the 400 week treatment duration is estimation. |
| Rationale for change | To clarify treatment duration. |
| Section to be changed | 3.3 Selection of trial population |
| Description of change | Change 1: The number of patients to be screened was increased from 9000 to 10.000 patients; |
| | Change 2: at least 6000 patients Was changed to: estimated number of 6000 patients; |
| | Change 3: clarification of expected number of patients per site and |
| | Change 4: Requirement to obtain approval from the TCM to randomise more than 30 patients was removed. |
| Rationale for change | Change 1: To reflect the expected number of screened patients based on actual data and current percentage of screen failures; |
| | Change 2: to clarify that the study is event driven and that the required number of patients is an estimation; |
| | Change 3: to clarify that sites could end up with less than 8 patients due to competitive recruitment and |
| | Change 4: approval to continue recruitment beyond 30 patients in a certain sites is given by the |

|-------|----|
| - "5" | • |

| | TCM to the CML and therefore will be |
|---|---|
| 0 4 4 7 7 | transferred to the monitoring manual. |
| Section to be changed | 3.3.3 Exclusion criteria |
| Description of change | Duration of short term insulin (up to two weeks) is allowed, if taken at least 8 weeks prior informed consent |
| | Was changed to: |
| | Duration of short term insulin (up to two |
| | consecutive weeks) is allowed, if taken at |
| | least 8 weeks prior informed consent. |
| Rationale for change | For clarification |
| Section to be changed | 3.3.4.1 Removal of individual patients |
| Description of change | Change 1: End of study was changed into end of trial; |
| | Change 2: inappropriateness of glimepiride treatment for renal safety issues according to local prescribing information was added as a withdrawal criterion; |
| | Change 3: the end of treatment requirements and follow-up procedures have been updated and |
| | Change 4: added that SU/glinide should not be taken in the morning of Visit 2. |
| Rationale for change | Change 1: To use consistent terminology in line with the protocol flow chart; |
| | Change 2: for clarification; |
| | Change 3: to clarify end of treatment activities and follow-up requirements and |
| | Change 4: |

| | to clarify that no double doses should be taken at Visit 2. |
|---|---|
| Section to be changed | 4.1.2 Method of assigning patients to treatment groups |
| Description of change | Added that sites will receive an information manual describing all steps to randomise a patients, obtain a medication kit assignment and to acknowledge study drug. |
| Rationale for change | For clarification. |
| Section to be changed | 4.1.4 Drug assignment and administration of doses for each patient |
| Description of change | Change 1: The titration requirements have been rewritten; |
| | Change 2: "If applicable" was added to the sentence that patients will continue their standard metformin therapy throughout the study; |
| | Change 3: investigator judgement to change study medication was changed into investigators judgement to change glimepirde/glimepiride placebo; |
| | Change 4: added that patients should be instructed to take trial medication once daily with water; |
| | Change 5: guidance on re-institution of glimepiride/ glimepiride placebo added and |
| | Change 6: Guidance on timing of in clinic visit added. |
| Rationale for change | Change 1: To clarify that glimepiride/glimepiride placebo is uptitrated and not study medication, which included linagliptin/linagliptin placebo (double dummy); |


| | Change 2: |
|---|---|
| | to clarify that treatment naive patients are |
| | eligible if intolerant or contra-indicated to |
| | first line anti-diabetic treatment; |
| | Change 3 and change 4: |
| | for clarification; |
| | Change 5: |
| | to add guidance on re-institution of trial |
| | medication and |
| | Change 6: |
| | To be consistent with instruction given in |
| | section 6.1. |
| Section to be changed | 4.1.7 Storage conditions |
| Description of change | <u>Change 1:</u> |
| | Added that in addition to wallets, blisters |
| | are provided; |
| | Change 2: |
| | added that a temperature log must be |
| | maintained at site and |
| | Change 3: |
| | medication return requirements were moved |
| | to the correct section in the protocol, section |
| | 4.1.8. |
| Rationale for change | <u>Change 1:</u> |
| | To clarify the use of wallets and blisters; |
| | Change 2: |
| | to clarify temperature monitoring |
| | requirements for study medication and |
| | Change 3: |
| | to move the drug accountability |
| | requirements to the corresponding section in |
| | the protocol. |
| Section to be changed | 4.1.8 Drug accountability |
| Description of change | Drug accountability requirements was shifted from Section 4.1.7 to this Section. |
| <b>Protocol Revision 6</b> | |
|----------------------------|---------------------|
| | _ |
| | Protocol Revision 6 |

| Rationale for change | To add drug accountability requirement to |
|---|---|
| | the correct clinical trial protocol section. |
| Section to be changed | 4.3 Treatment compliance |
| Description of change | Change 1: |
| | The requirement to use a worksheet to |
| | document treatment compliance was removed and |
| | Tomo you und |
| | Change 2: |
| | It was clarified that severe violation of |
| | compliance is seen as important protocol |
| | violation. |
| Rationale for change | Change 1: |
| | Treatment compliance should be reflected in the patient source documents and |
| | the patient source documents and |
| | Change 2: |
| | for clarification. |
| Section to be changed | 5.1.1 Endpoint(s) of efficacy |
| Description of change | Inclusion of classical MACE endpoint as |
| | first key secondary endpoint. |
| Rationale for change | This endpoint was defined as first key secondary endpoint. |
| Section to be changed | 5.1.2 Assessment of efficacy |
| Description of change | The definition of overnight fast was made |
| | consistent with the definition given in the |
| | protocol synopsis. |
| Rationale for change | For consistency. |
| Section to be changed | 5.2.1 Endpoint(s) of safety |
| Description of change | Change 1: |
| | The reporting requirements for outcome events was moved from section 5.2.2.2 to |
| | this section, describing the outcome events |
| | and |
| | Change 2: |
| | added that in case of a stroke the disability |
| | or dependence in daily activities will be collected with the modified Rankin Scale |
| | (mRS). |
| Rationale for change | Change 1: |
| 8. | _ <del></del> |

|------|-----|----|-----|

| | To reflect the outcome reporting requirements in the correct section of the clinical trial protocol and <a href="Change 2">Change 2</a> : to clarify that the grade of mRS is collected in case of a stroke. |
|---|---|
| Section to be changed | 5.2.2.1 Definitions of adverse events |
| Description of change | Change 1: Added that all symptomatic hypoglycaemic events, all asymptomatic hypoglycaemic events with glucose levels less than 3.0 mmol/L and all asymptomatic hypoglycaemic events considered an AE by the investigator should be reported as adverse event and |
| | Change 2: clarification that hepatic injury is to be reported as SAE added. |
| Rationale for change | Change 1: To clarify reporting procedures for hypoglycaemic events. Change 2: To be in line with Boehringer Ingelheim |
| Section to be changed | standard operating procedures. 5.2.2.2 Adverse event and serious adverse |
| | event reporting |
| Description of change | The reporting requirements for outcome events have been moved to section 5.2.1 of the clinical trial protocol. |
| Rationale for change | To reflect the reporting requirements of outcome events and AESI in the correct sections of the clinical trial protocol. |
| Section to be changed | 5.2.3 Assessment of safety laboratory parameters |
| Description of change | Change 1: Added that the lipid profile will only be obtained at Visits: 2, 6, 9, 12, 15, 18, 21, 24, 27 and 30; Change 2: |


| | added that bilirubin is not measured at Visit |
|---|---|
| | 1a; |
| | , |
| | Change 3: |
| | Change 3: |
| | Change 4. |
| | Change 4: |
| | additional laboratory parameters added to Visit 1a and |
| | Visit 1a and |
| | Change 5: |
| | added that the MDRD considers race as an |
| Dationals for shares | adjustment factor. |
| Rationale for change | Change 1: |
| | To clarify laboratory requirements; |
| | <u>Change 2:</u> |
| | to clarify that bilirubin is not measured a |
| | Visit 1a; |
| | Change 3: |
| | Change 4: |
| | Change 4: to clarify obtained laboratory parameters at |
| | to clarify obtained laboratory parameters at |
| | to clarify obtained laboratory parameters at Visit 1a and |
| | to clarify obtained laboratory parameters at Visit 1a and Change 5: |
| | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race |
| Section to be changed | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. |
| Section to be changed Description of shange | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. 5.2.4 Electrocardiogram (ECG) |
| Section to be changed Description of change | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. 5.2.4 Electrocardiogram (ECG) Added that in case of unresolved |
| - J | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. 5.2.4 Electrocardiogram (ECG) Added that in case of unresolved discrepancies investigators will not receive |
| Description of change | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. 5.2.4 Electrocardiogram (ECG) Added that in case of unresolved discrepancies investigators will not receive evaluated ECG reports from the vendor. |
| - J | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. 5.2.4 Electrocardiogram (ECG) Added that in case of unresolved discrepancies investigators will not receive evaluated ECG reports from the vendor. To clarify that in case of discrepancies the |
| Description of change Rationale for change | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. 5.2.4 Electrocardiogram (ECG) Added that in case of unresolved discrepancies investigators will not receive evaluated ECG reports from the vendor. To clarify that in case of discrepancies the processing timelines will be > 3 days. |
| Description of change | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. 5.2.4 Electrocardiogram (ECG) Added that in case of unresolved discrepancies investigators will not receive evaluated ECG reports from the vendor. To clarify that in case of discrepancies the processing timelines will be > 3 days. 5.2.5 Assessment of other safety |
| Description of change Rationale for change | to clarify obtained laboratory parameters at Visit 1a and Change 5: to state that MDRD formula considers race as an adjustment factor. 5.2.4 Electrocardiogram (ECG) Added that in case of unresolved discrepancies investigators will not receive evaluated ECG reports from the vendor. To clarify that in case of discrepancies the processing timelines will be > 3 days. |

20 April 2016

**Protocol Revision 6** 


| | The requirement to use the same blood |
|---|---|
| | pressure instrument and weight |
| | measurement scale throughout the study |
| | was changed into a similar type of blood pressure instrument and weight scale; |
| | pressure instrument and weight scare, |
| | Change 2: |
| | the procedure for HBGM devices and |
| | corresponding reporting and site contact |
| | requirements have been clarified and |
| | Change 3: |
| | a requirement to collect the HBGM diary at |
| | each visit was added. |
| Rationale for change | <u>Change 1:</u> |
| | Use of the same blood measure instrument |
| | or weight scale device is from operational perspective not feasible taking into account |
| | treatment duration. A similar type of |
| | instrument or scale is acceptable; |
| | Change 2: |
| | to clarify HBGM procedures and |
| | corresponding reporting and contact requirements and |
| | requirements and |
| | Change 3: |
| | to avoid potential loss of source data. |
| Rationale for change | |
| Section to be changed | |
| Description of change | The second paragraph was deleted. |
| Rationale for change | To remove duplicate text. |
| Section to be changed | 6.2.1 Screening an placebo run-in period |
| Description of change | Change 1: |
| | Transaminases was defined as ALT (SGPT) |
| | and AST (SGOT) and urine albumin and |
| | urine creatinine was added; |
| | Change 2: |
| | <u> </u> |


| | the placebo run-in duration was changed from 2 to weeks into 2 up to 4 weeks and |
|---|---|
| | Change 3: it was clarified that patient requiring rescue therapy during the placebo run-in are not eligible. |
| Rationale for change | Change 1: To clarify obtained laboratory parameters at Visit 1a; |
| | Change 2: to clarify the placebo-run in duration and |
| | Change 3: to clarify that rescue medication during placebo run-in is allowed, although the patient would not be eligible. |
| Section to be changed | 6.2.2 Treatment phase |
| Description of change | It was clarified that glimepiride/glimepiride placebo will be uptitrated between visits 2-6 and all end of trial activities have been transferred to section 6.2.3. |
| Description of change Rationale for change | placebo will be uptitrated between visits 2-6 and all end of trial activities have been |
| . 0 | placebo will be uptitrated between visits 2-6 and all end of trial activities have been transferred to section 6.2.3. To clarify that glimepiride/glimepiride placebo is uptitrated during Visits 2-6 and to transfer end of trial activities to the corresponding section of the clinical trial |
| Rationale for change | placebo will be uptitrated between visits 2-6 and all end of trial activities have been transferred to section 6.2.3. To clarify that glimepiride/glimepiride placebo is uptitrated during Visits 2-6 and to transfer end of trial activities to the corresponding section of the clinical trial protocol. |
| Rationale for change Section to be changed | placebo will be uptitrated between visits 2-6 and all end of trial activities have been transferred to section 6.2.3. To clarify that glimepiride/glimepiride placebo is uptitrated during Visits 2-6 and to transfer end of trial activities to the corresponding section of the clinical trial protocol. 6.2.3 End of trial and follow-up period Change 1: End of study was changed into end of trial |
| Rationale for change Section to be changed | placebo will be uptitrated between visits 2-6 and all end of trial activities have been transferred to section 6.2.3. To clarify that glimepiride/glimepiride placebo is uptitrated during Visits 2-6 and to transfer end of trial activities to the corresponding section of the clinical trial protocol. 6.2.3 End of trial and follow-up period Change 1: End of study was changed into end of trial and Change 2: the end of treatment requirements and |

| 1 426 130 01 173 | Page | 150 | of | 173 |
|------------------|------|-----|----|-----|
|------------------|------|-----|----|-----|

| | to clarify end of treatment activities and |
|---|---|
| | follow-up requirements. |
| Section to be changed | 7.1 Design |
| Description of change | The minimum number of patients of 6000 was changed into an estimated number of 6000 patients. |
| Rationale for change | To clarify that the study is event driven and that the required number of patients is an estimation. |
| Section to be changed | 7.1 Primary endpoint |
| Description of change | Patients without events will be considered censored at the end of study or at lost to follow-up, whichever comes first. |
| | Was changed to: If patients do not experience a primary endpoint event, they will be considered censored at their last documented study visit. If a patient died and has no primary outcome event, the patient will be censored at the date of death. |
| Rationale for change | Correction of description |
| Section to be changed | 7.1 Key secondary endpoints |
| Description of change | Definition of time to the first occurrence of any of the adjudicated components of the classical MACE composite endpoint as first key secondary endpoint. |
| | Definition of previous first and second key secondary endpoints as second and third key secondary endpoints. |
| Rationale for change | To include the testing for superiority on the time to the first occurrence of any of the adjudicated components of the classical MACE composite endpoint into the testing hierarchy as the third test. |
| Section to be changed | 7.1 Secondary cardiovascular endpoints |
| Description of change | Delete time to first occurrence of any of the adjudicated components of the classical MACE composite endpoint from secondary endpoints. |
| Rationale for change | This endpoint was defined as first key secondary endpoint. |

|--|------|-----|----|-----|
|--|------|-----|----|-----|

| Section to be changed | 7.2 Null and alternative hypotheses |
|---|---|
| Description of change | Change 1: Inclusion of the superiority hypothesis with respect to time to first occurrence of any of the adjudicated components of the classical MACE endpoint to be tested thirdly. |
| | The hypotheses on second and third key secondary endpoints will be tested fourthly and fifthly, respectively, if previous tests have revealed significant results. |
| | Change 2: Any confirmatory hypothesis test will be performed on the full analysis set. |
| Rationale for change | Change 1: Change of testing hierarchy to include also superiority testing for classical MACE endpoint. |
| | Change 2: According to Annotated clinical trial protocol instructions the patient population should be stated in this subsection. |
| Section to be changed | 7.3 Planned analysis |
| Description of change | Change 1: A protocol violation will be considered important if it can be expected to have a distorting influence on the assessment of the primary endpoint and/or key secondary endpoints. |
| | Change 2: The name of the on-treatment set was changed to 30-days-treatment set. |
| Rationale for change | Change 1: Explaining the details on important protocol violations. |
| | Change 2: Ensuring the name of the patient analysis set reflects the definition. |


| Section to be changed | 7.3.1 Primary analyses |
|---|---|
| Description of change | Change 1: It was clarified, that the Steering Committee, which is blinded, will decide on the number and time points of the interim analyses. |
| | <u>Change 2:</u> Change description of testing hierarchy according to Section 7.2 and |
| | Change 3: inclusion of description of sensitivity analyses of first key secondary endpoint. Clarification of sensitivity analyses for second and third key secondary endpoints. |
| | Change 4: The name of the on-treatment set was changed to 30-days-treatment set. |
| | Change 5: In the sensitivity analyses censoring will be done at time patients are on-treatment + 30 days after permanent treatment discontinuation or end of observation, whichever comes first. |
| | <u>Change 6:</u> The definition of the on-treatment analysis was included. |
| Rationale for change | Change 1: To ensure the decision on the number and time points for the formal interim analyses are made by the steering committee, which is blinded. |
| | Change 2: Inclusion of the superiority hypothesis with respect to time to first occurrence of any of the adjudicated components of the classical MACE endpoint to be tested thirdly and |
| | Change 3: |

| Page | 153 | of | 1 | 7 | 3 |
|------|-----|----|---|---|---|

| | Clarification of sensitivity analyses of key secondary endpoints. |
|---|---|
| | Change 4: Ensuring the name of the patient analysis set reflects the definition. |
| | Change 5: Clarification that in the sensitivity analyses the censoring will be performed at the time patients are on-treatment + 30 days after permanent treatment discontinuation or end of observation, whichever comes first. |
| | Change 6: The definition of the on-treatment analysis was included based on FDA request. |
| Section to be changed | 7.3.4 Interim analyses |
| Description of change | It was clarified, that the Steering Committee will decide on the number and time points of the interim analyses. The DMC will perform periodic safety reviews with a frequency as detailed in the DMC charter, but additional looks may be scheduled as needed by the DMC. In addition, the Steering Committee may also request the DMC to meet for a safety review. |
| Rationale for change | To ensure the decision on the number and time points for the formal interim analyses are made by the steering committee, which is blinded. It was clarified that the DMC performs periodic safety reviews. |
| Section to be changed | 7.5 Randomisation |
| Description of change | DMC will have access to randomisation code. |
| Rationale for change | To clarify the role of the DMC. |
| Section to be changed | 7.6 Determination of sample size |
| Description of change | The sentence on the decision about number and time points of the interim analyses was deleted. |

| Rationale for change | These details are clarified in Section 7.3.1 |
|---|---|
| | and 7.3.4. |
| Section to be changed | 8 informed consent, data protection, trial records |
| Description of change | The version as of October 1996 of the declaration of Helsinki was removed. |
| Rationale for change | To be in line with corporate standard operating procedures. |
| Section to be changed | 10.3 Blood pressure measurement procedure and treatment recommendations |
| Description of change | The requirement to use the same blood pressure instrument measurement scale throughout the study was changed into a similar type of blood pressure instrument. |
| Rationale for change | Use of the same blood measure instrument is from operational perspective not feasible taking into account treatment duration. A similar type of instrument or scale is acceptable. |
| Section to be changed | 10.5 Silent myocardial infarction |
| Description of change | Reference to section 10.2.4 deleted. |
| Rationale for change | No longer a valid reference. |
| Section to be changed | 10.6.2 procedures |
| Description of change | The procedures and testing requirement in case of clinical evaluation of liver injury have been aligned with the Boehringer Ingeheim standard operating procedure. |
| Rationale for change | To be in line with Boehringer Ingelheim standard operating procedures. |

| Number of CTP modification | 4 |
|---|---|
| Date of CTP modification | April 2013 |
| EudraCT number | 2009-013157-15 |
| BI Trial number | 1218.74 |
| BI Investigational Product(s) | Linagliptin |
| Title of protocol | A multicentre, international, randomised, parallel group, double blind study to evaluate Cardiovascular safety of linagliptin versus glimepiride in patients with type 2 diabetes mellitus at high cardiovascular risk. The CAROLINA Trial. |

20 April 2016

Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19

**Protocol Revision 6** 


| To be implemented only after | |
|---|---|
| approval of the | |
| IRB/IEC/Competent Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for | |
| approval | |
| Section to be changed | Title page |
| Description of change | Trial Clinical Monitor name and address |
| | details updated. |
| Rationale for change | New TCM assigned and address change. |
| Section to be changed | <b>Protocol synopsis (Duration of</b> |
| | treatment) |
| Description of change | Introduction of the term follow-up period |
| Rationale for change | To be in line with current Boehringer |
| | Ingelheim standard operating procedures |
| Section to be changed | Flow chart |
| Description of change | Flow chart |
| | Flow chart |
| Description of change | Abbreviations |
| Description of change Rationale for change | |
| Description of change Rationale for change Section to be changed | Abbreviations |
| Description of change Rationale for change Section to be changed Description of change | Abbreviations LADA was added to the list. |
| Description of change Rationale for change Section to be changed Description of change Rationale for change | Abbreviations LADA was added to the list. For clarification |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change Rationale for change | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently Typo correction |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change Rationale for change Rationale for change Section to be changed | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently Typo correction 3.3.4.1 Removal of individual patients |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change Rationale for change Rationale for change Section to be changed | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently Typo correction 3.3.4.1 Removal of individual patients Change 1: The possibility of vital status and outcome events follow up after informed consent |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change Rationale for change Rationale for change Section to be changed | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently Typo correction 3.3.4.1 Removal of individual patients Change 1: The possibility of vital status and outcome |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change Rationale for change Rationale for change Section to be changed | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently Typo correction 3.3.4.1 Removal of individual patients Change 1: The possibility of vital status and outcome events follow up after informed consent withdrawal was added. |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change Rationale for change Rationale for change Section to be changed | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently Typo correction 3.3.4.1 Removal of individual patients Change 1: The possibility of vital status and outcome events follow up after informed consent withdrawal was added. Change 2: |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change Rationale for change Rationale for change Section to be changed | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently Typo correction 3.3.4.1 Removal of individual patients Change 1: The possibility of vital status and outcome events follow up after informed consent withdrawal was added. Change 2: End of Trial was changed into End of |
| Description of change Rationale for change Section to be changed Description of change Rationale for change Section to be changed Description of change Rationale for change Rationale for change Section to be changed | Abbreviations LADA was added to the list. For clarification 3.1 Overall trial design and plan medication treatment permanently Typo correction 3.3.4.1 Removal of individual patients Change 1: The possibility of vital status and outcome events follow up after informed consent withdrawal was added. Change 2: |

| | Change 3:<br>(Follow up Visit) was added after V31 |
|---|---|
| | Change 4: Pancreatitis was added as a reason to stop the study medication. |
| | Change 5: "Permenantly" was added. |
| Rationale for change | Change 1: Obtain vital status and outcome events after withdrawal. |
| | Change 2: To be in line with the Flow chart |
| | Change 3: For clarification |
| | Change 4: Safety update |
| | Change 4: For clarification |
| Section to be changed | 4.2.1 Rescue medication, emergency procedures and additional treatment(s) |
| Description of change | For other than the protocol defined rescue medication it was specified that the study treatment should be discontinued when this rescue medication is contraindicated with the study treatment. |
| Rationale for change | For clarification |
| Section to be changed | 5.2.2.1 Definitions of adverse events |
| Description of change | Change 1: Reporting of non-serious AESIs according to the SAE procedure was added. |
| | Change 2: (with differentiation of bilirubin in direct and indirect <u>if total bilirubin is elevated</u> ) |


| | was added to the hepatic event bilirubin |
|-----------------------|----------------------------------------------|
| | testing. |
| Rationale for change | Change 1: |
| | Clarification of (S)AE and AESI reporting |
| | to be in line with Boehringer Ingelheim |
| | standard operating procedures. |
| | Change 2: |
| | For clarification |
| Section to be changed | 5.2.2.2 Adverse event and serious adverse |
| | event reporting |
| Description of change | Change 1: |
| | Introduction of the term follow-up period. |
| | Change 2: |
| | The following text was added: The |
| | investigator should report SAEs which |
| | occurred in a patient after the follow-up |
| | period, if the investigator becomes aware of |
| | them. |
| | Change 3: |
| | Paragraph regarding the immediate |
| | documentation of events was updated: The |
| | investigator must document immediately |
| | (within 24 hours of awareness or the next |
| | business day whichever is shorter) the |
| | following events on the SAE case page |
| | form in RDC: |
| | Change 4: |
| | Reporting of all AESIs according to the |
| | SAE procedure was added. |
| Rationale for change | Change 1: |
| <b></b> | To be in line with current Boehringer |
| | Ingelheim standard operating procedures. |
| | ingenienn standard operating procedures. |
| | Change 2: |
| | Clarification of (S)AE and AESI reporting |
| | to be in line with Boehringer Ingelheim |
| | standard operating procedures. |
| | Change 3: |

| | Clarification of (S)AE and AESI reporting to be in line with Boehringer Ingelheim standard operating procedures. Change 4: Clarification of (S)AE and AESI reporting to be in line with Boehringer Ingelheim standard operating procedures. |
|---|---|
| Dationals for shangs | |
| Rationale for change Section to be changed | 6.2.3 End of trial and Follow-up period |
| Description of change Rationale for change | Change 1: End of Trial was changed into End of Treatment Change 2: The possibility of vital status and outcome events follow up after informed consent withdrawal was added. Therefore the text about study end after ICF withdrawal was also removed. Change 1: To be in line with the Flow chart |
| | Change 2: Obtain vital status and outcome events after withdrawal. |
| Section to be changed | 7.1 Statistical Design – Model |
| Description of change | Change 1: Change 2: |

| Rationale for change | Changa 1: |
|-----------------------|------------------------------------|
| Rationale for change | Change 1: |
| | Measurements are only performed at |
| | <u>baseline.</u> |
| | Change 2: |
| | For clarification |
| Section to be changed | 7.3 Planned analyses |
| Description of change | Change 1: |
| | Change 2: |
| Rationale for change | Change 1: |
| | For clarification |
| | Change 2: |
| | Change 2. |

| Number of CTP modification | 5 |
|---|---|
| Date of CTP modification | 14 September 2015 |
| EudraCT number | 2009-013157-15 |
| BI Trial number | 1218.74 |
| BI Investigational Product(s) | Linagliptin |
| Title of protocol | A multicentre, international, randomised, parallel group, double blind study to evaluate Cardiovascular safety of linagliptin versus glimepiride in patients with type 2 diabetes mellitus at high cardiovascular risk. The CAROLINA Trial. |
| To be implemented only after approval of the | |

20 April 2016

Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19

**Protocol Revision 6** 


| IRB/IEC/Competent | |
|---|---|
| Authorities | |
| To be implemented | |
| immediately in order to | |
| eliminate hazard – | |
| IRB / IEC / Competent | |
| Authority to be notified of | |
| change with request for approval | |
| арргочаг | |
| Section to be changed | Title page |
| Description of change | Trial Clinical Monitor name and address |
| | details updated. |
| Rationale for change | New TCM assigned and address change. |
| Section to be changed | Flow chart |
| Description of change | Change 1: |
| | FU period changed from 7 to 30 days |
| | Change 2: |
| | Glomerular filtration rate and Fasting |
| | Plasma glucose samples to be taken at V31 |
| Rationale for change | Change 1: |
| | To be in line with the project FU period |
| | Change 2: |
| | To reflect actual testing done at V31 |
| Section to be changed | 3.1 Overall trial design and plan |
| Description of change | Text on Follow-up period was updated to |
| | reflect the 30d FU period |
| Rationale for change | For clarification |
| Section to be changed | 3.2 Discussion on trial design, including |
| D : ( C ) | the choice of control group |
| Description of change | Text on Follow-up period was updated to reflect the 30d FU period |
| Rationale for change | For clarification |
| Section to be changed | 3.3.4.1 Removal of individual patients |
| Description of change | Retention strategy language was updated + |
| | Follow-up period was updated to reflect the 30d FU period |
| Rationale for change | For clarification |
| Section to be changed | 4.2.1 Rescue medication, emergency |
| | procedures and additional treatment(s) |
| Description of change | 'Including during the FU period' was added |
| | <u> </u> |

| Rationale for change | Text on Follow-up period was updated to reflect the 30d FU period |
|---|---|
| Section to be changed | 5.2.2.1 Definitions of adverse events |
| Description of change | Change 1: AESI: alignment of text throughout the Lina project Change 2: addition of pancreatic cancer as AESI Change 3: throughout this section, text was updated to reflect current standard text |
| Rationale for change | Change 1: For clarification Change 1: Alignment within the Lina project Change 3: AE and SAE definitions were updated to reflect the latest standard text |
| Section to be changed | 5.2.2.2 Adverse event and serious adverse event reporting |
| Description of change | throughout this section, text was updated to reflect current standard text |
| Rationale for change | AE and SAE definitions were updated to reflect the latest standard text |
| Section to be changed | 5.2.2.3 Oncological adverse events |
| Description of change | Oncological assessment was added |
| Rationale for change | For clarification |
| Section to be changed | 5.2.3.4 Renal function impairment |
| Description of change | Formulas taken out and reference made to the Statistical Analysis Plan |
| Rationale for change | For clarification |
| Section to be changed | 6.2.3 End of trial and Follow-up period |
| Description of change | Text adapted to be in line with section 3.3.4.1 |
| Rationale for change | For clarification |
| Section to be changed | 7.1 Statistical design - model |
| Description of change | <u>Change 1</u> : |
| | <u>Change 2</u> : Secondary diabetic related endpoints |

20 April 2016

Boehringer Ingelheim BI Trial No.: 1218.74 Doc No.: c01618200-19

|------|-----|----|-----|

| | 'Urinary' added to albumin |
|----------------------|----------------------------|
| Rationale for change | Change 1: |
| | For clarification |
| | Change 2: |
| | For clarification |

| Number of CTP modification | 6 |
|---|---|
| Date of CTP modification | 20 April 2016 |
| EudraCT number | 2009-013157-15 |
| BI Trial number | 1218.74 |
| BI Investigational Product(s) | Linagliptin |
| Title of protocol | A multicentre, international, randomised, parallel group, double blind study to evaluate Cardiovascular safety of linagliptin versus glimepiride in patients with type 2 diabetes mellitus at high cardiovascular risk. The CAROLINA Trial. |
| To be implemented only after approval of the IRB/IEC/Competent Authorities | |
| To be implemented immediately in order to eliminate hazard — IRB / IEC / Competent Authority to be notified of change with request for approval | |
| Section to be changed | Title page |
| Description of change | <u>Change 1:</u> Trial Clinical Monitor name and address details updated. |
| Rationale for change | <u>Change 1:</u> Change in Trial Clinical Monitor |
| Section to be changed | Clinical Trial Protocol Synopsis |
| Description of change | Objectives: Change 1: Primary endpoint changed to time to the first occurrence of any of the following adjudicated components of the primary composite endpoint: CV death (including fatal stroke and fatal MI), nonfatal MI (excluding silent MI) or non-fatal stroke. |

| | <u>Change 3:</u> Estimated trial duration updated to 432 weeks. |
|---|---|
| | Cuitania fan afficacy: |
| | Criteria for efficacy: |
| | Change 4: Primary endpoint changed to time to the first occurrence of any of the following adjudicated components of the primary composite endpoint: CV death (including fatal stroke and fatal MI), nonfatal MI (excluding silent MI) or non-fatal stroke. |
| | Change 5: First key secondary endpoint changed to time to the first occurrence of any of the following adjudicated components of: CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI), non-fatal stroke or hospitalisation for unstable angina pectoris. |
| | Criteria for safety |
| | Change 6:silent myocardial infarction was changed into: and occurrence of and time to silent myocardial infarction. |
| Rationale for change | <u>Change 1, 4, 5:</u> |
| | Testing hierarchy revised following a unanimous request from the trial Academic Steering Committee. |
| | Change 2: For clarification. |
| | Change 3: Estimated trial duration increased due to change of primary endpoint. |


| | Change 6: Clarification added, that silent |
|---|---|
| | MI is not a by adjudication confirmed endpoint. |
| Section to be changed | Flowchart |
| Description of change | Change 1: Two additional visits added to |
| | the trial flow chart. |
| | Change 2: footnote 'n':at minimum a yearly telephone call and a telephone call at study end will be asked for, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit might be recorded. |
| | Was changed into: |
| | at minimum a yearly telephone call and a telephone call at study end (through the patient or alternative person designated by the patient) will be asked for, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit should be recorded. |
| Rationale for change | Change 1: Estimated trial duration increased due to change of primary endpoint. |
| | Change 2: for clarification. |
| Section to be changed | Abbreviations |
| Description of change | Abbreviations section updated. |
| Rationale for change | For clarification |
| Section to be changed | 1.2 Drug profile |
| <b>Description of change</b> | Drug profile section updated. |
| Rationale for change | For clarification per current version of the investigator brochure. |
| Section to be changed | 2.2 Trial objectives |
| Description of change | Change 1: Primary endpoint changed to time to the first occurrence of any of the following adjudicated components of the primary composite endpoint: CV death (including fatal stroke and fatal MI), nonfatal MI (excluding silent MI) or non-fatal stroke. |

|--|------|-----|----|-----|
|--|------|-----|----|-----|

| Rationale for change | Change 2: First key secondary endpoint changed to time to the first occurrence of any of the following adjudicated components of: CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI), non-fatal stroke or hospitalisation for unstable angina pectoris. Change 1, 2: Testing hierarchy revised following a unanimous request from the trial Academic Steering Committee. |
|---|---|
| Section to be changed | 3.1 Overall trial design and plan |
| Description of change | + + |
| Description of change | Change 1: Estimated treatment time updated to 432 weeks and duration of maintenance phase updated to an estimated 416 weeks. |
| | Change 2:at minimum a yearly telephone call and a telephone call at study end will be asked for, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit might be recorded. |
| | Was changed into:at minimum a yearly telephone call and a telephone call at study end (through the patient or alternative person designated by the patient) will be asked for, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit should be recorded. |
| | Change 3: Guidance revised on the timing of the EOT visit after study stop announcement after 631 endpoint events are reached. |
| Rationale for change | Change 1: Estimated trial duration increased due to change of primary endpoint. |
| | Change 2: For clarification. |

| |
|-----------------|
|-----------------|

| | <u>Change 3:</u> To clarify the respective actions |
|---|---|
| | to stop the trial when 631 endpoint events |
| | are reached. |
| Section to be changed | 3.2 Discussion of trial design, including the choice of control group |
| Description of change | Estimated trial duration updated to 432 weeks. |
| Rationale for change | Estimated trial duration increased due to change of primary endpoint. |
| Section to be changed | 3.3.1 administrative structure of the trial |
| Description of change | Clinical Event Committee was changed in Clinical Event Committees. |
| Rationale for change | Correction of typographical error |
| Section to be changed | 3.3.4.1 Removal of individual patients |
| Description of change | Change 1:at minimum a yearly telephone call and a telephone call at study end will be asked for, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit might be recorded. Was changed into:at minimum a yearly telephone call and a telephone call at study end (through the patient or alternative person designated by the patient) will be asked for, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit should be recorded. Change 2: See further details in section 4.2 was added following the last sentence of paragraph 5. Change 3Visit 31 (Follow-up) was alwayed into: Visit 32 (Follow-up) |
| Rationale for change | <i>changed into</i> : Visit 33 (Follow-up). Change 1+2: For clarification |
| National Ioi Change | <u>Change 1+2</u> . For clarification <u>Change 3:</u> Two additional Visits added as the estimated trial duration increased due to change of primary endpoint. |
| Section to be changed | 4.1.4 Drug assignment and |
| Description 6.1 | administration of doses for each patient |
| Description of change | IXRS will allocate medication kit numbers at each scheduled in-clinic visit (V2 – |

|------|-----|----|-----|
|------|-----|----|-----|

| | V20) A4i-i4- ( 204i4i11i |
|---|---|
| | V29)At visits 6-29 patients will receive one treatment box |
| | Was changed into:IXRS will allocate medication kit numbers at each scheduled in-clinic visit (V2 – V31)At visits 6-31 patients will receive one treatment box |
| Rationale for change | Two additional Visits added as the estimated trial duration increased due to change of primary endpoint. |
| Section to be changed | 5.1.1 Endpoint(s) off efficacy |
| Description of change | Change 1: Primary endpoint changed to time to the first occurrence of any of the following adjudicated components of the primary composite endpoint: CV death (including fatal stroke and fatal MI), nonfatal MI (excluding silent MI) or non-fatal stroke. |
| | Change 2: First key secondary endpoint changed to time to the first occurrence of any of the following adjudicated components of: CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI), non-fatal stroke or hospitalisation for unstable angina pectoris. |
| Rationale for change | Change 1, 2: Testing hierarchy revised following a unanimous request from the trial Academic Steering Committee. |
| Section to be changed | 5.2.2.1 Assessment of adverse events |
| Description of change | <b>AESI:</b> the following sentence was omitted Documentation should be done on the AESI |
| | and SAE form. |
| Rationale for change | |
| Rationale for change Section to be changed | and SAE form. Covered in section 5.2.2.2 adverse event |
| Ū | <ul> <li>and SAE form.</li> <li>Covered in section 5.2.2.2 adverse event and serious adverse event reporting.</li> <li>5.2.2.2 Adverse event and serious adverse</li> </ul> |
| Section to be changed | and SAE form. Covered in section 5.2.2.2 adverse event and serious adverse event reporting. 5.2.2.2 Adverse event and serious adverse event reporting Immediate documentations of events: On the SAE to the sponsor was changed into: |
| Section to be changed Description of change | and SAE form. Covered in section 5.2.2.2 adverse event and serious adverse event reporting. 5.2.2.2 Adverse event and serious adverse event reporting Immediate documentations of events: On the SAE to the sponsor was changed into: On the SAE form to the sponsor. |


| Rationale for change | Additional Visits added as the estimated trial duration increased due to change of primary endpoint. |
|---|---|
| Section to be changed | 6.2.2 Treatment phase |
| Description of change | Change 1:regularly scheduled randomization as specified was changed into: regularly scheduled Visits as specified |
| | Change 2: The following text was omitted either by clinic visits or by phone (refer to section 6.2.3) and the following text was added: If a patient who prematurely discontinued study drug is not willing to return at the pre-defined regular visit schedule, at minimum a yearly telephone call (preferably every 6 months) and a telephone call at study end (through the patient or alternative person designated by the patient) will be required, to document the occurrence of outcome events and vital status. If possible, also other AE's and concomitant therapy changes since last visit should be recorded. Every attempt will be made by the investigator to ensure patients continue participating in the study during study drug interruptions and after discontinuation of study drug. |
| | <u>Change 3</u> :even if the dose must be down titrated <i>was changed into</i> : even if the dose must be titrated |
| Rationale for change | <u>Change 1</u> : Correction of error. |
| | <u>Change 2</u> : For clarification and consistency with section 3. |
| | Change 3: For clarification. |
| Section to be changed | 6.2.3 End of trial and follow-up period |
| Description of change | Change 1: The following text was added: A patient has the right to withdraw informed consent for participation at any time for any reason. However, withdrawal of consent from study participation should be very rare and unusual. Because of this, the |

|--|------|-----|----|-----|
|--|------|-----|----|-----|

| | investigator must be involved in the discussions with the patient regarding a withdrawal of consent. Change 2: for end of treatment visit and visit 31 (follow-up) was changed into: or end of treatment visit and visit 33(follow-up). |
|---|---|
| | <u>Change 3:</u> Paragraph starting with patient who discontinueremoved |
| Rationale for change | <u>Change 1</u> : For clarification and consistency with section 3. |
| | <u>Change 2:</u> Two additional Visits added as the estimated trial duration increased due to change of primary endpoint. |
| | Change 3: Covered in section 6.2.2 and section 3. |
| Section to be changed | 7.1 STATISTICAL DESIGN - MODEL |
| Description of change | Change 1: Estimated trial duration updated to 432 weeks. Change 2: Primary endpoint changed to time to the first occurrence of any of the following adjudicated components of the primary composite endpoint: CV death (including fatal stroke and fatal MI), nonfatal MI (excluding silent MI) or non-fatal stroke. Change 3: First key secondary endpoint changed to time to the first occurrence of any of the following adjudicated components of: CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI), non-fatal stroke or hospitalisation for unstable angina pectoris. Change 4: List "time to silent MI" |
| | separately from adjudicated tertiary cardiovascular endpoints. |
| Rationale for change | Change 1: Estimated trial duration increased due to change of primary endpoint. |
| | <u>Change 2,3:</u> Testing hierarchy revised following an unanimous request from the trial Academic Steering Committee. |

| | Change 4: Clarification added, that silent |
|---|---|
| | MI is not a by adjudication confirmed |
| | endpoint. |
| Section to be changed | 7.2 NULL AND ALTERNATIVE |
| | HYPOTHESES |
| Description of change | First key secondary endpoint details removed. |
| Rationale for change | First key secondary endpoint was changed to time to the first occurrence of any of the following adjudicated components of: CV death (including fatal stroke and fatal MI), non-fatal MI (excluding silent MI), non-fatal stroke or hospitalisation for unstable angina pectoris. |
| Section to be changed | 7.3 PLANNED ANALYSES |
| Description of change | Change 1: Protocol violation is considered important if it can be expected to have a distorting influence on the assessment of the primary endpoint and/or first key secondary endpoint. The example of limited life expectancy (<5 |
| | years) due to various medical conditions) as important protocol violations was removed. Change 2: |
| Rationale for change | Change 1: Clarification that important protocol violations are defined in relation to adjudicated outcome events as part of primary and first key secondary endpoint. The trial Statistical Analysis Plan describes all important protocol violations in detail. Change 2: |
| Section to be changed | 7.3.1 Primary analyses |
| Description of change | A Bonferroni adjustment will be applied after the first DMC interim analysis for 4P-MACE and the following analyses based on 3P-MACE. The O'Brien & Fleming alphaspending function based on the new overall alpha (after Bonferroni adjustment) defines the overall significance level for the second DMC interim analysis and final analysis. Removed sentence, that the Steering |

Boehringer Ingelheim BI Trial No.: 1218.74

| | Committee will decide on the number of interim analyses. |
|---|---|
| Rationale for change | The change of the primary endpoint from time to first adjudicated event of the composite of 4P-MACE to the time to first adjudicated event of the composite of 3P-MACE requires adjustment of the alpha level which is addressed via a Bonferroni adjustment. |
| | The number of two interim analyses and the number of events required for each of the two interim analyses were defined by the Steering Committee to be based on approximately 190 and 411 primary endpoint events. This decision was documented in the SC minutes and the DMC Charter. |
| Section to be changed | 7.3.2 Secondary analyses |
| Description of change | Chi square test and logistic regression for CV endpoints removed. |
| Rationale for change | Cardiovascular events will be analysed by a Cox proportional hazards model and occurrence of events reported with frequency and incidence rates. Analyses that do not account for the time at risk are not required. |
| Section to be changed | 7.3.4 Interim analyses |
| Description of change | A Bonferroni adjustment will be applied after the first DMC interim analysis for 4P-MACE and the following analyses based on 3P-MACE. The O'Brien & Fleming alphaspending function based on the new overall alpha (after Bonferroni adjustment) defines the allocation of the overall significance level for the second interim analysis and final analysis. Removed sentence, that the Steering Committee will decide on the number of interim analyses. |
| Rationale for change | The change of the primary endpoint from time to first adjudicated event of the composite of 4P-MACE to the time to first adjudicated event of the composite of 3P-MACE requires adjustment of the alpha level which is addressed via a Bonferroni adjustment. |

Boehringer Ingelheim 20 April 2016

| | The number of two interim analyses and the number of events required for each of the two interim analyses were defined by the Steering Committee to be based on approximately 190 and 411 primary endpoint events. This decision was documented in the SC minutes and the DMC Charter. |
|---|---|
| Section to be changed | 7.6 DETERMINATION OF SAMPLE SIZE |
| Description of change | Change 1: A Bonferroni adjustment will be applied between the first DMC interim analysis for 4P-MACE and the following analyses regarding 3P-MACE. The O'Brien & Fleming alpha-spending function based on the new overall alpha (after Bonferroni adjustment) defines the allocation of the overall significance level for the second DMC interim analysis and final analysis. |
| | <u>Change 2:</u> Assumed annual event rates updated for changed primary endpoint. |
| Rationale for change | Change 1: The change of the primary endpoint from time to first adjudicated event of the composite of 4P-MACE to the time to first adjudicated event of the composite of 3P-MACE requires adjustment of the alpha level which is addressed via a Bonferroni adjustment. Change 2: Lower event rates assumed for |
| Section to be abanged | updated primary endpoint. |
| Section to be changed Description of change | 9.1 Published References Author of IB omitted and update of published references |
| Rationale for change | Change in authorship and reflected of published references used for the protocol revision. |
| Section to be changed | 10.5 SILENT MYOCARDIAL<br>INFARCTION |
| Description of change | Definition of silent MI requires no preceding clinical history of MI (including stent thrombosis and other coronary events) and investigator reporting of silent MI |

Boehringer Ingelheim
BI Trial No.: 1218.74
20 April 2016

| Rationale for change | Clarified that Silent MI is diagnosed on |
|----------------------|----------------------------------------------|
| | relevant ECG abnormalities, clinical history |
| | and investigator reporting. |